# **Cover Page for Statistical Analysis Plan**

| Sponsor name: | Novo Nordisk A/S |
|---|---|
| NCT number | NCT03989232 |
| Sponsor trial ID: | NN9535-4506 |
| Official title of study: | Efficacy and Safety of Semaglutide 2.0 mg s.c. Once-weekly Compared to Semaglutide 1.0 mg s.c. Once-weekly in Subjects With Type 2 Diabetes |
| Document date*: | 15 December 2020 |

<sup>\*</sup>Document date refers to the date on which the document was most recently updated.

Note: The date in the header from Page 2 is the date of compilation of the documents and not of an update to content.

Once-weekly Semaglutide
Trial ID: NN9535-4506
Clinical Trial Report
Appendix 16.1.9

Date: 15 December 2020 Version: 1.0
Status: Final

## 16.1.9 Documentation of statistical methods

## List of contents

| Statistical analysis plan | Link |
|-------------------------------------------|------|
| MedDRA searches for safety focus areas | Link |
| MedDRA searches – list of preferred terms | Link |

Redacted statistical analysis plan Includes redaction of personal identifiable information only. 
 Statistical analysis plan
 Date:
 11 September 2020
 Novo Nordisk

 Trial ID: NN9535-4506
 Version:
 1.0

 UTN: U1111-1224-5162
 Status:
 Final

 EudraCT No: 2018-004529-96
 Page:

# NN9535-4506

# Statistical analysis plan

Statistical analysis plan Trial ID: NN9535-4506 UTN: U1111-1224-5162 EudraCT No: 2018-004529-96

#### CONFIDENTIAL

Date: Version: Status: Page:

11 September 2020 | Novo Nordisk 1.0 Final


# **Table of contents**

| | | | | Page |
|---|---|---|---|---|
| Ta | able of | f content | S | 2 |
| Ta | able of | f tables | | 3 |
| V | ersion | history. | | 4 |
| 1 | Intro | duction | | 5 |
| • | 1.1 | | ves and endpoints | |
| | | 1.1.1 | Primary objective | |
| | | 1.1.2 | Secondary objective | |
| | | 1.1.3 | Primary endpoint | |
| | | 1.1.4 | Secondary endpoints | 5 |
| | | | 1.1.4.1 Confirmatory secondary endpoint | |
| | | | 1.1.4.2 Supportive secondary endpoints | |
| | 1.2 | Trial de | esign | 13 |
| 2 | Stati | stical hy | potheses | 13 |
| 3 | Sami | nle size d | letermination | 13 |
| 4 | | - | | |
| 5 | | stical an | alyses | 16 |
| | 5.1 | | l considerations | |
| | 5.2<br>5.3 | | disposition | |
| | 3.3 | 5.3.1 | / endpoint analysis | |
| | | 3.3.1 | 5.3.1.1 Primary hypothetical estimand | |
| | | | 5.3.1.2 Primary treatment policy estimand | |
| | | 5.3.2 | Sensitivity analyses | |
| | | | 5.3.2.1 Primary hypothetical estimand | |
| | | | 5.3.2.2 Primary treatment policy estimand | |
| | | 5.3.3 | Overview of statistical analyses and intercurrent events | |
| | 5.4 | | ary endpoint analysis | |
| | | 5.4.1 | Confirmatory secondary endpoints | |
| | | | 5.4.1.1 Main analytical approach | |
| | | 5.4.2 | 5.4.1.2 Sensitivity analyses | |
| | 5.5 | 5.4.2<br>Explore | Supportive secondary endpoints | |
| | 5.6 | | afety analyses | |
| | 5.7 | | nalyses | |
| | | 5.7.1 | Subgroup analyses | |
| | | | 5.7.1.1 Hypothetical strategy | |
| | | | 5.7.1.2 Treatment policy strategy | |
| | | 5.7.2 | Subpopulation analysis | |
| | | | 5.7.2.1 Hypothetical strategy | |
| | <b>.</b> 0 | <b>.</b> | 5.7.2.2 Treatment policy strategy | |
| | 5.8 | Interim | analyses | 25 |
| 6 | Supp | | ocumentation | |
| | 6.1 | Append | lix 1: List of abbreviations | 26 |
| | 6.2 | | lix 2: Changes to protocol-planned analyses | |
| | 6.3 | Append | lix 3: Definition and calculation of endpoints, assessments and derivations | 27 |
| 7 | Refe | rences | | 28 |

# **Table of tables**

| | | Page |
|---|---|---|
| Table 1 | Overview of estimands | 7 |
| Table 2 | Power for different scenarios | 14 |
| Table 3 | Statistical analyses of the confirmatory endpoints | 19 |
| Table 4 | Statistical handling of intercurrent events for the primary analyses of the confirmatory endpoints | 20 |
| Table 5 | Statistical analyses of the supportive secondary endpoints | 21 |
| Table 6 | Endpoints | 27 |

 Statistical analysis plan
 Date:
 11 September 2020
 Novo Nordisk

 Trial ID: NN9535-4506
 Version:
 1.0

 UTN: U1111-1224-5162
 Status:
 Final

 EudraCT No: 2018-004529-96
 Page:

# **Version history**

This Statistical Analysis Plan (SAP) for trial NN9535-4506 is based on the protocol version 4.0 dated 15JUN2020.

#### 1 Introduction

This SAP covers specification of statistical considerations and analyses for efficacy data and safety data available at time of partial data base lock performed after the date of last subject last treatment, where Novo Nordisk will become unblinded and complete efficacy data will be available and analysed, but where safety data will only be partial complete.

Only additional statistical analyses have been included, hence there are no changes to protocol specified statistical analyses.

#### 1.1 Objectives and endpoints

#### 1.1.1 Primary objective

To establish the superior effect of semaglutide s.c. 2.0 mg once-weekly versus semaglutide s.c. 1.0 mg once-weekly on glycaemic control in subjects with T2D, on a background of metformin with or without SU treatment.

#### 1.1.2 Secondary objective

To compare the effect of semaglutide s.c. 2.0 mg once-weekly versus semaglutide s.c. 1.0 mg once-weekly in subjects with T2D, on a background of metformin with or without SU treatment, on:

- Body weight
- Vital signs
- Hypoglycaemia
- General safety and tolerability

#### 1.1.3 Primary endpoint

• Change from baseline (week 0) to week 40 in HbA<sub>1c</sub> (%-point)

#### 1.1.4 Secondary endpoints

#### 1.1.4.1 Confirmatory secondary endpoint

• Change from baseline (week 0) to week 40 in body weight (kg)

#### 1.1.4.2 Supportive secondary endpoints

#### Supportive secondary effect endpoints

Change from baseline (week 0) to week 40 in:

- Fasting plasma glucose (FPG) (mmol/l)
- Body mass index (BMI) (kg/m<sup>2</sup>)
- Waist circumference (cm)

Statistical analysis plan UTN: U1111-1224-5162 Date: 11 September 2020 Status: Trial ID: NN9535-4506 EudraCT No: 2018-004529-96 Version: 1.0 Page:

- $HbA_{1c} < 7\%$  at week 40 (yes/no)
- $HbA_{1c} \le 6.5\%$  at week 40 (yes/no)
- Weight loss  $\geq 5\%$  at week 40 (yes/no)
- Weight loss  $\geq 10\%$  at week 40 (yes/no)

## Supportive secondary safety endpoints

- Number of treatment emergent severe or blood glucose confirmed symptomatic hypoglycaemic episodes from first dose to week 40
- Change from baseline (week 0) to week 40 in pulse rate (bpm)

Statistical analysis plan Trial ID: NN9535-4506

UTN: U1111-1224-5162 EudraCT No: 2018-004529-96

| Date: 11 September 2020 | Status: | Version: 1.0 | Page:

Final Novo Nordisk 7 of 28

# Table 1 Overview of estimands

| Objective | Estimand strategy | Estimand category | Estimand |
|---|---|---|---|
| Primary Objective: | Hypothetical | Primary (except US) | Treatment condition: 2.0 mg semaglutide s.c. once-weekly or 1.0 mg semaglutide s.c. once-weekly |
| To establish the superior effect | | | Variable/Endpoint: Change from baseline to week 40 in HbA <sub>1c</sub> |
| weekly versus semaglutide s.c. | | | Population of interest: All randomised |
| glycaemic control in subjects with T2D, on a background of metformin with or without SU treatment | | | <b>Intercurrent event strategy:</b> Initiation of rescue medication: "had rescue medication not been available" (hypothetical). Discontinuation of trial product before week 40: "had patients adhered to treatment" (hypothetical). Change in dose during and after dose escalation: "regardless of change in dose" (treatment policy). |
| | | | Population level summary measure: Mean difference |
| | | Secondary* | Treatment condition: 2.0 mg semaglutide s.c. once-weekly or 1.0 mg semaglutide s.c. once-weekly |
| | | | Variable/Endpoint: Change from baseline to week 40 in FPG |
| | | | Population of interest: All randomised |
| | | | Intercurrent event strategy: Initiation of rescue medication: "had rescue medication not been available" (hypothetical). Discontinuation of trial product before week 40: "had patients adhered to treatment" (hypothetical). Change in dose during and after dose escalation: "regardless of change in dose" (treatment policy). |
| | | | Population level summary measure: Mean difference |

| Final <b>Novo Nordisk</b><br>8 of 28 | | or 1.0 mg semaglutide s.c. once-weekly | | | "had rescue medication not been<br>re week 40: "had patients adhered to<br>e escalation: "regardless of change in | | or 1.0 mg semaglutide s.c. once-weekly | | | "had rescue medication not been<br>re week 40: "had patients adhered to<br>e escalation: "regardless of change in | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 11 September 2020 Status:<br>1.0 Page: | | Treatment condition: 2.0 mg semaglutide s.c. once-weekly or 1.0 mg semaglutide s.c. once-weekly | Variable/Endpoint: HbA <sub>1c</sub> < 7% at week 40 | Population of interest: All randomised | <b>Intercurrent event strategy:</b> Initiation of rescue medication: "had rescue medication not been available" (hypothetical). Discontinuation of trial product before week 40: "had patients adhered to treatment" (hypothetical). Change in dose during and after dose escalation: "regardless of change in dose" (treatment policy). | Population level summary measure: Odds ratio | Treatment condition: 2.0 mg semaglutide s.c. once-weekly or 1.0 mg semaglutide s.c. once-weekly | Variable/Endpoint: $HbA_{1c} \le 6.5\%$ at week 40 | Population of interest: All randomised | <b>Intercurrent event strategy:</b> Initiation of rescue medication: "had rescue medication not been available" (hypothetical). Discontinuation of trial product before week 40: "had patients adhered to treatment" (hypothetical). Change in dose during and after dose escalation: "regardless of change in dose" (treatment policy). | Population level summary measure: Odds ratio |
| Date:<br>Version: | Estimand | Treatment cond | Variable/Endpo | Population of in | Intercurrent event stra<br>available" (hypothetical)<br>treatment" (hypothetical,<br>dose" (treatment policy). | Population level | Treatment cond | Variable/Endpo | Population of in | Intercurrent event stra<br>available" (hypothetical)<br>treatment" (hypothetical<br>dose" (treatment policy) | Population leve |
| .24-5162<br>118-004529-96 | Estimand category | Secondary* | | | | | Secondary* | | | | |
| UTN: U1111-1224-5162<br>EudraCT No: 2018-004529-96 | Estimand strategy | | | | | | | | | | |
| Statistical analysis plan<br>Trial ID: NN9535-4506 | Objective | | | | | | | | | | |

| Treatment policy Primary (US) Hypothetical Secondary (except US) | UTN: U1111-1224-5162 Date: 11 September 2020 Status: EudraCT No: 2018-004529-96 Version: 1.0 Page: | ttus: Final $\left \begin{array}{c} \textit{Novo Nordisk} \\ \textit{9 of } 28 \end{array} \right $ |
|---|---|---|
| Treatment policy Primary (US) Hypothetical Secondary (except US) | Estimand category | |
| Hypothetical Secondary (except US) | Primary (US) | Treatment condition: 2.0 mg semaglutide s.c. once-weekly or 1.0 mg semaglutide s.c. once-weekly |
| Hypothetical Secondary (except US) | Variable/Endpoint: Change from baseline to week 40 in HbA <sub>1c</sub> | week 40 in HbA1c |
| Hypothetical Secondary (except US) | Population of interest: All randomised | |
| Hypothetical Secondary (except US) | Intercurrent event strategy: Initiation of rescue medication: "reg medication" (treatment policy). Discontinuation of trial product discontinuation due to adverse event" (treatment policy). dose escalation: "regardless of change in dose" (treatment policy). | Intercurrent event strategy: Initiation of rescue medication: "regardless of initiation of rescue medication" (treatment policy). Discontinuation of trial product due to adverse event: "regardless of trial product discontinuation due to adverse event" (treatment policy). Change in dose during and after dose escalation: "regardless of change in dose" (treatment policy). |
| Hypothetical Secondary (except US) | Population level summary measure: Mean difference | lifference |
| | Secondary (except | Treatment condition: 2.0 mg semaglutide s.c. once-weekly or 1.0 mg semaglutide s.c. once-weekly |
| | Variable/Endpoint: Change from baseline to week 40 in body weight | week 40 in body weight |
| | Population of interest: All randomised | |
| reatment" (hypothe sions hynoolycaemia general | Intercurrent event strategy: Initiation of rescavailable" (hypothetical). Discontinuation of tretreatment" (hypothetical). Change in dose duri | <b>Intercurrent event strategy:</b> Initiation of rescue medication: "had rescue medication not been available" (hypothetical). Discontinuation of trial product before week 40: "had patients adhered to treatment" (hypothetical). Change in dose during and after dose escalation: "regardless of change in dose" (treatment policy). |
| | Population level summary measure: Mean difference | lifference |

| | gory Estimand | Treatment condition: 2.0 mg semaglutide s.c. once-weekly or 1.0 mg semaglutide s.c. once-weekly | Variable/Endpoint: Change from baseline to week 40 in BMI | Population of interest: All randomised | Intercurrent event strategy: Initiation of rescue medication: "had rescue medication not been available" (hypothetical). Discontinuation of trial product before week 40: "had patients adhered to treatment" (hypothetical). Change in dose during and after dose escalation: "regardless of change in dose" (treatment policy). | Population level summary measure: Mean difference | Treatment condition: 2.0 mg semaglutide s.c. once-weekly or 1.0 mg semaglutide s.c. once-weekly | Variable/Endpoint: Change from baseline to week 40 in waist circumference | Population of interest: All randomised | Intercurrent event strategy: Initiation of rescue medication: "had rescue medication not been available." (hypothetical). Discontinuation of trial product before week 40: "had patients adhered to treatment" (hypothetical). Change in dose during and after dose escalation: "regardless of change in dose" (treatment policy). | Population level summary measure: Mean difference |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 224-5162<br>318-004529-96 | Estimand category | Secondary* | | | | | Secondary* | | | | |
| UTN: U1111-1224-5162<br>EudraCT No: 2018-004529-96 | Estimand strategy | | | | | | | | | | |
| Statistical analysis plan<br>Trial ID: NN9535-4506 | | | | | | | | | | | |

| Statistical analysis plan<br>Trial ID: NN9535-4506 | UTN: U1111-1224-5162<br>EudraCT No: 2018-004529-96 | 224-5162<br>318-004529-96 | Date:<br>Version: | 11 September 2020 Status:<br>1.0 Page: | Final Novo Nordisk |
|---|---|---|---|---|---|
| Objective | Estimand strategy | Estimand category | Estimand | | |
| | | Secondary* | Treatment condition | Treatment condition: 2.0 mg semaglutide s.c. once-weekly or 1.0 mg semaglutide s.c. once-weekly | semaglutide s.c. once-weekly |
| | | | Variable/Endpoint: | Variable/Endpoint: Body weight loss $\geq 5\%$ at week 40 | |
| | | | Population of interest: All randomised | st: All randomised | |
| | | | Intercurrent event strat<br>available" (hypothetical)<br>treatment" (hypothetical)<br>dose" (treatment policy). | Intercurrent event strategy: Initiation of rescue medication: "had rescue medication not been available" (hypothetical). Discontinuation of trial product before week 40: "had patients adhered to treatment" (hypothetical). Change in dose during and after dose escalation: "regardless of change in dose" (treatment policy). | cue medication not been<br>40: "had patients adhered to<br>ion: "regardless of change in |
| | | | Population level sun | Population level summary measure: Odds ratio | |
| | | Secondary* | Treatment condition | Treatment condition: 2.0 mg semaglutide s.c. once-weekly or 1.0 mg semaglutide s.c. once-weekly | semaglutide s.c. once-weekly |
| | | | Variable/Endpoint: | Variable/Endpoint: Body weight loss ≥ 10% at week 40 | |
| | | | Population of interest: All randomised | st: All randomised | |
| | | | Intercurrent event stra<br>available" (hypothetical)<br>treatment" (hypothetical<br>dose" (treatment policy) | Intercurrent event strategy: Initiation of rescue medication: "had rescue medication not been available" (hypothetical). Discontinuation of trial product before week 40: "had patients adhered to treatment" (hypothetical). Change in dose during and after dose escalation: "regardless of change in dose" (treatment policy). | cue medication not been<br>40: "had patients adhered to<br>ion: "regardless of change in |
| | | | Population level sun | Population level summary measure: Odds ratio | |

| Statistical analysis plan Trial ID: NN9535-4506 | UTN: U1111-1224-5162<br>EudraCT No: 2018-004529-96 | 224-5162<br>318-004529-96 | Date: Version: | 11 September 2020 Status:<br>1.0 Page: | Final<br>12 of 28 | Novo Nordisk |
|---|---|---|---|---|---|---|
| | Estimand strategy | Estimand category | Estimand | | | |
| L | Freatment policy | Secondary (US) | Treatment conditio | <b>Treatment condition:</b> 2.0 mg semaglutide s.c. once-weekly or 1.0 mg semaglutide s.c. once-weekly | semaglutide | s.c. once-weekly |
| | | | Variable/Endpoint: | Variable/Endpoint: Change from baseline to week 40 in body weight | | |
| | | | Population of interest: All randomised | sst: All randomised | | |
| | | | Intercurrent event medication" (treatmential product disconti | Intercurrent event strategy: Initiation of rescue medication: "regardless of initiation of rescue medication" (treatment policy). Discontinuation of trial product due to adverse event: "regardless of trial product discontinuation due to adverse event" (treatment policy). Change in dose during and after | ss of initiatic<br>adverse even<br>Thange in dog | on of rescue<br>t: "regardless of<br>se during and after |
| | | | dose escalation: "reg | dose escalation: 'regardless of change in dose'' (treatment policy). | a<br>a | ٥ |
| | | | Population level su | Population level summary measure: Mean difference | | |

The hypothetical estimand will be considered the primary estimand except in the US, where FDA specifically has requested the treatment policy estimand to be the primary.

<sup>\*</sup>Not related to any confirmatory hypothesis

Statistical analysis plan Trial ID: NN9535-4506 UTN: U1111-1224-5162 EudraCT No: 2018-004529-96


Date: Version: Status: Page:

11 September 2020 | Novo Nordisk Final


#### 1.2 Trial design

See protocol section 5.

#### 2 **Statistical hypotheses**

The statistical testing strategy will be performed for the primary analysis of each of the two estimand strategies separately. I.e. statistical testing will be performed separately for the hypothetical strategy and the treatment policy strategy. In order to preserve the overall type-I error in the strong sense at a 5% significance level (two-sided) within each estimand strategy, the conclusion of superiority of semaglutide 2.0 mg versus semaglutide 1.0 mg will be evaluated hierarchically according to the sequence below. The treatment difference is defined as  $\mu =$ (semaglutide 2.0 mg minus semaglutide 1.0 mg).

- 1. Superiority of semaglutide 2.0 mg versus semaglutide 1.0 mg on change from baseline to week 40 in HbA<sub>1c</sub>
  - $H_0$ :  $\mu \ge 0.0$  %-point against  $H_a$ :  $\mu < 0.0$  %-point
- 2. Superiority of semaglutide 2.0 mg vs. semaglutide 1.0 mg on change from baseline to week 40 in body weight
  - $H_0$ :  $\mu \ge 0.0$  kg against  $H_a$ :  $\mu < 0.0$  kg

#### Sample size determination 3

The primary endpoint is change from baseline (week 0) to week 40 in HbA<sub>1c</sub> (%-point) and the confirmatory secondary endpoint is change from baseline (week 0) to week 40 in body weight (kg). Both endpoints will be tested for superiority. The type-I error rate will be controlled in the strong sense across the primary and the confirmatory secondary hypotheses, separately for each estimand, at an overall alpha level (two-sided) of 0.05. Multiplicity control and criteria for confirming the hypotheses is described in section 2.

The sample size calculation is performed to ensure sufficient power for confirming superiority of semaglutide 2.0 mg vs. semaglutide 1.0 mg on change from baseline to week 40 in HbA<sub>1c</sub> (%-point) based on each estimand separately.

#### **Primary endpoint**

An on-treatment HbA<sub>1c</sub> treatment effect of -0.26%-point was predicted based on exposure-response modelling.

To accommodate the treatment policy estimand, the on-treatment effect is adjusted by 15% based on results from the SUSTAIN phase 3a programme, where a lower effect was observed for the treatment policy estimand as compared to the on-treatment effect. With the adjusted HbA<sub>1c</sub> treatment effect of -0.22%-point and a standard deviation of 1.1%-point, 964 subjects will be randomised in order to obtain 87% power for confirming superiority for the primary endpoint based on the treatment policy estimand and at least 87% power for confirming superiority for the primary

| Statistical analysis plan | | Date: | 11 September 2020 | Novo Nordisk |
|---|---|---|---|---|
| UTN: U1111-1224-5162 | CONTIDENTIAL | Status: | Final | |
| EudraCT No: 2018-004529-96 | | Page: | 14 of 28 | |

endpoint based on the hypothetical estimand. This is based on a 1:1 randomisation, a two-sided significance level of 0.05, and a t-test. The assumed standard deviation is based on the SUSTAIN programme.

## **Confirmatory secondary endpoint**

With 964 subjects randomised to ensure sufficient power (87%) for confirming superiority for the primary endpoint based on the treatment policy estimand, a marginal power of 90% for confirming that semaglutide 2.0 mg is superior to semaglutide 1.0 mg on change from baseline to week 40 in body weight (based on each estimand) is obtained if the true treatment difference is as low as - 0.84 kg. This is based on a 1:1 randomisation, a two-sided significance level of 0.05, a t-test, and a standard deviation of 4.0 kg. The assumed standard deviation is based on the SUSTAIN programme.

#### Sensitivity analyses for the sample size calculation

The sensitivity of power for confirming superiority for the primary endpoint based on the treatment policy estimand for a fixed sample size of 964 subjects is presented in <u>Table 2</u>.

 Table 2
 Power for different scenarios

| Scenario | On-treatment | Adjusted for the | Adjusted | Randomised | Power |
|---|---|---|---|---|---|
| | effect | treatment policy | treatment effect | subjects | |
| | | estimand | | | |
| Scenario 1 | -0.25 %-point | 15 % | -0.21 | 964 | 84 % |
| Scenario 2 | -0.25 %-point | 20 % | -0.20 | 964 | 81 % |
| Scenario 3 | -0.27 %-point | 15 % | -0.23 | 964 | 90 % |
| Scenario 4 | -0.27 %-point | 20 % | -0.22 | 964 | 87% |
| Scenario 5 | -0.29 %-point | 15 % | -0.25 | 964 | 94 % |
| Scenario 6 | -0.29 %-point | 20 % | -0.23 | 964 | 90 % |

## 4 Analysis sets

Data selection for statistical analyses will be a two-step process, first selecting subjects based on the analysis population and subsequently events/data for those subjects based on the observation period.

Full analysis set (FAS): All randomised subjects. Subjects will be analysed according to the treatment to which they were assigned at randomisation.

Safety analysis set (SAS): All subjects exposed to at least one dose of trial product. Subjects will be analysed according to the trial product received for the majority of the period they were on treatment.

'In-trial' observation period: This observation period is defined as the period from the date of randomisation to the first of the following dates, both inclusive:

- The follow-up visit (P11)
- Date of death
- Date when subject withdrew informed consent
- Date of last contact for subjects lost to follow-up

'On-treatment' observation period: This observation period is a sub-set of the 'in-trial' observation period and represents the time period where subjects are considered exposed to trial product. The observation period starts at the date of first dose of trial product and ends at an endpoint-specific end-date. For adverse events including hypoglycaemic events, the observation period ends at the first date of any of the following:

- The follow-up visit (P11)
- The treatment discontinuation follow-up visit (P11A)
- The date of last dose of trial product +49 days
- The end-date for the 'in-trial' observation period

The follow-up visit is scheduled to take place 7 weeks after the last date on trial product, i.e., 49 days.

For efficacy and other safety assessments (laboratory assessments, body measurements, and vital signs) the 'on-treatment' observation period ends at the last date on trial product with a visit window of +14 days. Hence, for these assessments, the 'on-treatment' observation period reflects the period in which subjects are treated.

'On-treatment without rescue medication' observation period: This observation period is a sub-set of the 'on-treatment' observation period and represents the time period where subjects are considered treated with trial product but have not initiated any rescue medications. The observation period starts at the date of first dose of trial product and ends at the first date of any of the following:

| Statistical analysis plan | Date: | 11 September 2020 | Novo Nordisk |
|---|---|---|---|
| EudraCT No: 2018-004529-96 | Page: | 16 of 28 | |

- Initiation of rescue medication
- The date of last dose of trial product +14 days

Data points collected outside an observation period will be treated as missing in the analysis. Baseline data will always be included in an observation period.

Rescue medication is defined as any new anti-diabetic medication and/or intensification of anti-diabetic medication initiated at or after date of randomisation and before last date on trial product.

The following rules will be applied based on the concomitant medication data reported by the investigator, to determine whether or not the recorded anti-diabetic medication is 1. *New anti-diabetic medication* or 2. *Intensification of anti-diabetic medication* 

*New anti-diabetic medication:* Anti-diabetic medication (4th-level ATC code) that is initiated after randomisation and is new compared to the anti-diabetic background medication at randomisation and with a dosing duration of more than 21 days.

*Intensification of anti-diabetic medication:* A more than 20% increase in the dose of anti-diabetic medication after randomisation as compared to the anti-diabetic medication dose at randomisation (5th-level ATC code not changed) and with a dosing duration of more than 21 days.

Before data are locked for statistical analysis, a review of all data will take place. In general subjects should not be excluded from an analysis set and observations should not be excluded from an observation period, if they fulfil the criteria. If subjects or observations are excluded, the reasons for their exclusion must be documented before database lock and described in the clinical trial report. Any decision to exclude either a subject or single observation from the statistical analysis is the joint responsibility of the members of the Novo Nordisk study group.

## 5 Statistical analyses

#### 5.1 General considerations

The comparison presented from a statistical analysis will be semaglutide 2.0 mg versus semaglutide 1.0 mg and results will be presented by the estimated treatment contrast with associated two-sided 95% confidence intervals and *p*-values corresponding to two-sided tests of no difference if not otherwise specified.

Data from all sites will be analysed and reported together.

If no statistical analysis is specified, data will be presented using relevant summary statistics. Accordingly, adverse events will be summarised descriptively. Data collected before randomisation (V2) will only be summarised descriptively.

| Statistical analysis plan | Date: | 11 September 2020 | Novo Nordisk |
|---|---|---|---|
| EudraCT No: 2018-004529-96 | Page: | 17 of 28 | |

A partial database lock will be performed at the end of the treatment period for all subjects, i.e. after the date of the last patient last treatment (LPLT) visit. The database will be updated after the partial database lock to include remaining PK data and any additional safety information. The full database lock will be performed after the date of the last patient last visit (LPLV).

Novo Nordisk will become unblinded at the time of the partial database lock, whereas subjects and investigators will remain blinded until after last patient last visit (LPLV). The analysis of the primary endpoint and all other efficacy endpoints will be performed based on the data from the partial database lock. Analysis of safety and PK data will be performed after the full database lock. This approach is implemented to allow earlier availability of semaglutide 2 mg to the patient population expected to benefit from a higher dose and to support further development activities with semaglutide s.c. A detailed plan for data handling and operational aspects of the partial database lock and the database update will be finalised before the partial database lock.

#### 5.2 Subject disposition

See mock TFLs.

#### 5.3 Primary endpoint analysis

#### 5.3.1 Main analytical approach

#### 5.3.1.1 Primary hypothetical estimand

The primary (except US) hypothetical estimand, see <u>Table 1</u>, will be estimated based on FAS using post-baseline data collected up to and including week 40 from the 'on-treatment without rescue medication' observation period.

Imputation of missing data will be handled by multiple imputation (MI) assuming that missing data are missing at random (MAR). The imputation will be performed separately within each treatment group defined by randomised treatment. First, intermittent missing values are imputed using a Markov Chain Monte Carlo (MCMC) method, to obtain a monotone missing data pattern, generating 500 complete data sets. Secondly, a sequential conditional linear regression approach for imputing monotone missing values will be implemented starting with the first visit after baseline and sequentially continuing to the last planned visit at week 40. The model used for imputation will include the baseline and post-baseline HbA<sub>1c</sub> values observed prior to the visit in question as covariates.

The 500 complete datasets will be analysed using an analysis of covariance (ANCOVA) with treatment and stratification as fixed factors and the baseline  $HbA_{1c}$  as covariate. Rubin's rule<sup>1</sup> will be applied to obtain inference.

#### 5.3.1.2 Primary treatment policy estimand

The primary (US) treatment policy estimand, see <u>Table 1</u>, will be estimated based on the FAS using week 40 data from the 'in-trial' observation period.

Imputation of missing data will be handled by MI assuming that missing data are missing at random. The imputation will be performed by imputing missing week 40 data separately within groups defined by randomised treatment and treatment status at week 40 (retrieved drop-out), in total, four groups as follows; (i) semaglutide 1.0 mg and on-treatment at week 40, (ii) semaglutide 1.0 mg and off-treatment at week 40, (iii) semaglutide 2.0 mg and on-treatment at week 40, (iv) semaglutide 2.0 mg and off-treatment at week 40.

For each of the four groups an ANCOVA with baseline  $HbA_{1c}$  as covariate will be fitted to observed values of the change from baseline in  $HbA_{1c}$  at week 40. The estimated parameters for location and dispersion will then be used to impute 500 values for each subject with missing week 40 data based on only baseline  $HbA_{1c}$ .

The 500 complete datasets will be analysed using an analysis of covariance (ANCOVA) with treatment and stratification as fixed factors and the baseline  $HbA_{1c}$  as covariate. Rubin's rule<sup>1</sup> will be applied to obtain inference.

#### 5.3.2 Sensitivity analyses

#### 5.3.2.1 Primary hypothetical estimand

A tipping point sensitivity analysis will be performed for the primary (except US) hypothetical estimand, by repeating the ANCOVA described in section 5.3.1.1, however, prior to analysis subjects from the semaglutide 2.0 mg group with missing observations at week 40 will be given a penalty, i.e., it is assumed that subjects with missing observations who are randomised to semaglutide 2.0 mg will receive a treatment that is less beneficial than subjects with observed values who are randomised to semaglutide 2.0 mg. The addition of the penalty values and subsequent analysis steps should be repeated with increasing penalty values until a significant result in the corresponding superiority analysis is no longer significant. This analysis will only be performed if superiority is confirmed based on the primary analysis.

#### 5.3.2.2 Primary treatment policy estimand

A tipping point sensitivity analysis for the primary (US) treatment policy estimand will be performed by repeating the ANCOVA described in section 5.3.1.2, however, prior to analysis subjects from the semaglutide 2.0 mg group with missing observations at week 40 will be given a penalty. The addition of the penalty values and subsequent analysis steps should be repeated with increasing penalty values until a significant result in the corresponding superiority analysis is no longer significant. This analysis will only be performed if superiority is confirmed based on the primary analysis.

| Statistical analysis plan | Date: | 11 September 2020 | Novo Nordisk |
|---|---|---|---|
| EudraCT No: 2018-004529-96 | Page: | 19 of 28 | |

In addition, a two-way tipping point sensitivity analysis will be conducted as this may be a more reflective of a real-world situation for missing data from both treatment arms. The ANCOVA described in section 5.3.1.2 is repeated, however prior to analysis penalties of opposite sign are added to the imputed values at week 40 in both treatment arms simultaneously. The approach is to explore a range of penalties for both treatment groups, and the impact these would have on the study conclusions. This sensitivity analysis evaluates the robustness of the superiority conclusions to departures from the imputed change in HbA<sub>1c</sub> in both treatment groups. The analysis will only be performed if superiority is confirmed based on the primary analysis.

Let  $(\Delta_{2.0 mg}, \Delta_{1.0 mg})$  denote a pair of penalties to (semaglutide 2.0 mg, semaglutide 1.0 mg). Then, for a given superiority hypothesis that is confirmed, denote the corresponding 'one-way' tipping points with  $(\Delta_{2.0 mg}^1, 0)$  for semaglutide 2.0 mg and  $(0, \Delta_{1.0 mg}^1)$  for semaglutide 1.0 mg. It follows that the domain of penalties in a 'two-way' tipping point analysis should include a grid over (0,0) to  $(\Delta_{2.0 mg}^1, \Delta_{1.0 mg}^1)$ .

The analyses are presented as contour plots for the test probability (p-value) of superiority as a function of the penalties ( $\Delta_{2.0 mg}$ ,  $\Delta_{1.0 mg}$ ). In this representation the contour line corresponding to 0.05 will partition the grid of penalties into two regions: a region where superiority of semaglutide 2.0 mg is confirmed at a 5% significance level and a region where superiority is no longer confirmed.

#### 5.3.3 Overview of statistical analyses and intercurrent events

An overview of all analyses addressing the two primary estimands for the confirmatory endpoints is provided in Table 3.

Table 3 Statistical analyses of the confirmatory endpoints

| | | Analysis | Observation | Statistical | | Sensitivity |
|---|---|---|---|---|---|---|
| Endpoint | Estimand | set | period | model | Imputation approach | analysis |
| Primary endpoin | t | | | | | |
| | Hypothetical | FAS | On- | ANCOVA | MAR within randomised | Tipping |
| | | | treatment | | treatment group | point |
| Change in | | | w/o rescue | | | analysis |
| HbA <sub>1c</sub> (%-point) | Treatment | FAS | In-trial | ANCOVA | MAR within group | One-way and |
| TIDAIc (70-point) | policy | | | | defined by randomised | two-way |
| | | | | | treatment and treatment | tipping point |
| | | | | | status at week 40 | analyses |
| Confirmatory sec | ondary endpoi | int | | | | |
| | Hypothetical | FAS | On- | ANCOVA | MAR within randomised | Tipping |
| | | | treatment | | treatment group | point |
| Change in body | | | w/o rescue | | | analysis |
| weight (kg) | Treatment | FAS | In-trial | ANCOVA | MAR within group | One-way and |
| weight (kg) | policy | | | | defined by randomised | two-way |
| | | | | | treatment and treatment | tipping point |
| | | | | | status at week 40 | analyses |

Abbreviations: ANCOVA; analysis of covariance; FAS: full analysis set; MAR: missing at random.

| Statistical analysis plan | Date: | 11 September 2020 | Novo Nordisk |
|---|---|---|---|
| EudraCT No: 2018-004529-96 | Page: | 20 of 28 | |

The following <u>Table 4</u> describes how anticipated intercurrent events during the trial are handled for confirmatory endpoints. The different intercurrent events will be handled in the same manner for both confirmatory endpoints.

Table 4 Statistical handling of intercurrent events for the primary analyses of the confirmatory endpoints

| | | Handling | | |
|---|---|---|---|---|
| | Hypothetical estimand | | Treati | nent policy estimand |
| Intercurrent event | Strategy | Data | Strategy | Data |
| Change in dose<br>during and after the<br>dose escalation<br>period | Treatment policy | Assessments will be performed and collected at scheduled visits after the intercurrent event and used in the analysis | Treatment policy | Assessments will be performed and collected at scheduled visits after the intercurrent event and used in the analysis |
| <ul> <li>Treatment<br/>discontinuation due<br/>to AEs</li> <li>Initiation of rescue<br/>(anti-diabetic)<br/>medication</li> </ul> | Hypothetical | Assessments for scheduled visits after the time of the intercurrent event are considered missing and will be imputed assuming MAR as described in the analysis | Treatment policy | Assessments will be performed and collected at scheduled visits after the intercurrent event and used in the analysis |

## 5.4 Secondary endpoint analysis

#### **5.4.1** Confirmatory secondary endpoints

The confirmatory secondary endpoint is change from baseline (week 0) to week 40 in body weight (kg).

#### 5.4.1.1 Main analytical approach

## Secondary hypothetical estimand

Similar analyses as described in section 5.3.1.1 with body weight values instead of HbA<sub>1c</sub> values will be performed.

#### Secondary treatment policy estimand

Similar analyses as described in section 5.3.1.2 with body weight values instead of HbA<sub>1c</sub> values will be performed.

Statistical analysis plan Trial ID: NN9535-4506 UTN: U1111-1224-5162 EudraCT No: 2018-004529-96


Date: Version: Status: Page:

11 September 2020 | Novo Nordisk Final 21 of 28

#### 5.4.1.2 Sensitivity analyses

#### Secondary hypothetical estimand

One-way tipping point sensitivity analysis as described in section 5.3.2.1 with body weight values instead of HbA<sub>1c</sub> values will be performed.

#### Secondary treatment policy estimand

Both one-way and two-way tipping point analyses as those described in section 5.3.2.2 with body weight values instead of HbA<sub>1c</sub> values will be performed.

#### 5.4.2 Supportive secondary endpoints

The supportive secondary endpoints are listed in Table 6 and all relevant estimands are described in Table 1. A hypothetical estimand strategy will be applied for all supportive secondary endpoints.

#### **Continuous endpoints**

Analyses of change in FPG, BMI and waist circumference will be performed as described in section 5.3.1.1 with values for the given parameter instead of  $HbA_{1c}$  values based on FAS using data from the 'on-treatment without rescue medication' observation period. The analysis of change from baseline to week 40 in pulse rate will be based on SAS using data from the 'on-treatment' observation period, but otherwise using the same approach as described in section 5.3.1.1.

#### Responder endpoints

To account for missing data, the binary endpoints will be derived from the 500 imputed datasets described in section 5.3.1.1. Each of the complete data sets will be analysed using a logistic regression (LR) model with treatment and stratification as fixed effects and associated baseline response as covariate. Estimated odds ratios will be log-transformed and inference will be drawn using Rubin's rule<sup>1</sup>. The results will be back-transformed and described by the odds ratio between treatments and the associated 95% CI and p-value for no treatment difference.

#### Overview of statistical analyses

An overview of all analyses of the supportive secondary endpoints is provided in Table 5.

Table 5 Statistical analyses of the supportive secondary endpoints

| | | Analysis | Observation | Statistical | |
|---|---|---|---|---|---|
| Endpoint | Estimand | set | period | model | Imputation approach |
| Supportive secondary endpoints (effect related) | | | | | |
| Change in FPG | Hypothetical | FAS | On-treatment | ANCOVA | MAR within randomised |
| (mmol/) | | | w/o rescue | | treatment group |
| Change in BMI | Hypothetical | FAS | On-treatment | ANCOVA | MAR within randomised |
| (kg/m <sup>2</sup> ) | | | w/o rescue | | treatment group |

| | | Analysis | Observation | Statistical | |
|---|---|---|---|---|---|
| Endpoint | Estimand | set | period | model | Imputation approach |
| Change in waist | Hypothetical | FAS | On-treatment | ANCOVA | MAR within randomised |
| circumference (cm) | | | w/o rescue | | treatment group |
| $HbA_{1c} < 7\% \text{ (yes/no)}$ | Hypothetical | FAS | On-treatment | LR | MAR within randomised |
| | | | w/o rescue | | treatment group |
| $HbA_{1c} \le 6.5\%$ | Hypothetical | FAS | On-treatment | LR | MAR within randomised |
| (yes/no) | | | w/o rescue | | treatment group |
| Weight loss ≥ 5% | Hypothetical | FAS | On-treatment | LR | MAR within randomised |
| (yes/no) | | | w/o rescue | | treatment group |
| Weight loss ≥ 10% | Hypothetical | FAS | On-treatment | LR | MAR within randomised |
| (yes/no) | | | w/o rescue | | treatment group |
| Supportive secondary | endpoints (sat | fety related) | ) | | |
| Change in pulse | - | SAS | On-treatment | ANCOVA | MAR within randomised |
| (bpm) | | | | | treatment group |
| Number of | - | SAS | On-treatment | NBR | - |
| hypoglycaemic | | | | | |
| episodes | | | | | |

**Abbreviations:** ANCOVA; analysis of covariance; FAS: full analysis set; LR: logistic regression; MAR: missing at random; NBR: negative binomial regression; SAS: safety analysis set

#### 5.5 Exploratory endpoint analysis

Not applicable.

#### 5.6 Other safety analyses

Number of treatment emergent severe or blood glucose confirmed symptomatic hypoglycaemic episodes at week 40 will be analysed using a negative binomial regression (NBR) model with a log-link function and the logarithm of the time period covered by the subject's 'on-treatment' observation period as offset. The model will include treatment and stratification as fixed factors and baseline HbA<sub>1c</sub> as a covariate. This analysis will be based on the SAS using the 'on-treatment' observation period. The results will be described by the rate ratio between treatments and the associated 95% CI and *p*-value for no treatment difference.

The binary assessment indicating whether a subject has had no treatment emergent severe or blood glucose confirmed symptomatic hypoglycaemic episodes at week 40 or at least one will be analysed using a logistic regression model. The model will include treatment and stratification as fixed effects and baseline  $HbA_{1c}$  as covariate, and the analysis will be based on SAS using data from the 'on-treatment' observation period. The results will be described by the odds ratio between treatments and the associated 95% confidence interval and p-value for no treatment difference.

| Statistical analysis plan | Date: | 11 September 2020 | Novo Nordisk |
|---|---|---|---|
| EudraCT No: 2018-004529-96 | Page: | 23 of 28 | |

#### 5.7 Other analyses

Population PK modelling and exposure-response analyses may be included to support dose selection and to explore the benefits of high versus lower doses of semaglutide in subjects with T2D.

The modelling will include data from all randomised subjects that were exposed to semaglutide in this trial and might be performed as a meta-analysis including data from historical trials. Actual dose and date of administration of last dose before PK sampling will be registered in the CRF and used in the analysis, together with actual time point for PK sampling. The analysis will be further specified in a modelling analysis plan that is to be prepared before database lock.

The modelling analyses will be performed by Quantitative Clinical Pharmacology at Novo Nordisk A/S and will be reported separately from the CTR.

## 5.7.1 Subgroup analyses

Change from baseline to week 40 in HbA<sub>1c</sub> will be analysed according to the following three subgroup splits:

- $HbA_{1c} < 9\%$  and  $HbA_{1c} \ge 9\%$  at baseline
- BMI < 30 and BMI  $\ge 30$  at baseline
- BMI < 35 and BMI  $\ge 35$  at baseline

The rationale for conducting these subgroup analyses is to generate evidence to support potential individualised treatment in clinically relevant subpopulations with high  $HbA_{1c}$  or BMI, where subjects may experience even further improvement of glycaemic control from advancing to a higher dose of semaglutide.

From each analysis the estimated treatment differences in change from baseline to week 40 in HbA<sub>1c</sub> across subgroups with 95% confidence intervals will be presented.

#### 5.7.1.1 Hypothetical strategy

The effect of randomised treatment on change from baseline to week 40 in  $HbA_{1c}$  across subgroups will be analysed based on a hypothetical estimand strategy by using the same 500 imputed and complete data sets as described in section 5.3.1.1. On these 500 complete data sets an ANCOVA having baseline  $HbA_{1c}$  level as covariate, treatment and stratification as well as the interaction between the relevant subgroup and treatment as fixed factors, will be applied. Rubin's rule will be applied to obtain inference.

#### 5.7.1.2 Treatment policy strategy

Addressing the effect of randomised treatment on change from baseline to week 40 in  $HbA_{1c}$  across subgroups by a treatment policy strategy the 500 imputed data described in section 5.3.1.2, will also

| Statistical analysis plan | Date: | 11 September 2020 | Novo Nordisk |
|---|---|---|---|
| EudraCT No: 2018-004529-96 | Page: | 24 of 28 | |

be analysed by an ANCOVA having baseline HbA<sub>1c</sub> level as covariate, treatment and stratification as well as the interaction between the relevant subgroup and treatment as fixed factors, will be applied. Rubin's rule<sup>1</sup> will be applied to obtain inference.

## 5.7.2 Subpopulation analysis

To further support individualised treatment, an analysis of change in HbA<sub>1c</sub> from week 12 to week 40 will be performed in the subpopulation of all randomised subjects that are on-treatment, have not initiated rescue medication and are adherent to semaglutide 1.0 mg at week 12, having a week 12 HbA<sub>1c</sub>  $\geq$  7%.

This represents a clinically meaningful and important subpopulation of patients that are expected to particularly benefit from advancing to a higher dose of semaglutide.

Due to the trial design, where both treatment arms receive semaglutide unblinded for the first 12 weeks, subpopulation membership is arguably unrelated to treatment assignment. Accordingly, an analysis of change from week 12 to week 40 in  $HbA_{1c}$  in this subpopulation will still have the benefit of randomisation.

#### 5.7.2.1 Hypothetical strategy

The endpoint change from week 12 to week 40 in HbA<sub>1c</sub> in the subpopulation will be analysed with the hypothetical estimand strategy, see <u>Table 1</u> for definition of intercurrent events.

Imputation of missing data will be handled by MI assuming that missing data pattern is MAR. The imputation will be performed separately within each treatment group defined by randomised treatment. First, intermittent missing values are imputed using a Markov Chain Monte Carlo (MCMC) method, to obtain a monotone missing data pattern, generating 500 complete data sets. Secondly, a sequential conditional linear regression approach for imputing monotone missing values will be implemented starting with the first visit after week 12 and sequentially continuing to the last planned visit at week 40. The model used for imputation will include the HbA<sub>1c</sub> at week 12 and post-baseline HbA<sub>1c</sub> values observed prior to the visit in question as covariates.

The 500 complete datasets will be analysed using an analysis of covariance (ANCOVA) with treatment and stratification as fixed factors and HbA<sub>1c</sub> at week 12 as covariate. Rubin's rule<sup>1</sup> will be applied to obtain inference.

## 5.7.2.2 Treatment policy strategy

The endpoint change from week 12 to week 40 in  $HbA_{1c}$  in the subpopulation will be analysed with the treatment policy estimand strategy, see Table 1 for definition of intercurrent events.

Imputation of missing data will be handled by MI assuming that missing data pattern is MAR. The imputation will be performed by imputing missing week 40 data separately within groups defined

| Statistical analysis plan | Date: | 11 September 2020 | Novo Nordisk |
|---|---|---|---|
| EudraCT No: 2018-004529-96 | Page: | 25 of 28 | l |

by randomised treatment and treatment status at week 40 (retrieved drop-out), in total, four groups as follows; (i) semaglutide 1.0 mg and on-treatment at week 40, (ii) semaglutide 1.0 mg and off-treatment at week 40, (iii) semaglutide 2.0 mg and on-treatment at week 40, (iv) semaglutide 2.0 mg and off-treatment at week 40.

For each of the four groups an ANCOVA with HbA<sub>1c</sub> at week 12 as covariate will be fitted to observed values of the change from week 12 to week 40 in HbA<sub>1c</sub>. The estimated parameters for location and dispersion will then be used to impute 500 values for each subject with missing week 40 data based on only HbA<sub>1c</sub> at week 12.

The 500 complete datasets will be analysed using an analysis of covariance (ANCOVA) with treatment and stratification as fixed factors and HbA<sub>1c</sub> at week 12 as covariate. Rubin's rule<sup>1</sup> will be applied to obtain inference.

#### 5.8 Interim analyses

Not applicable.

Statistical analysis plan Trial ID: NN9535-4506 UTN: U1111-1224-5162 EudraCT No: 2018-004529-96


Date: Version: Status: Page:

11 September 2020 | Novo Nordisk

Final


#### **Supporting documentation** 6

#### 6.1 **Appendix 1: List of abbreviations**

ΑE adverse event

**ANCOVA** analysis of covariance

**ATC** Anatomical Therapeutic Chemical

BMI body mass index

bpm beats per minute

CI confidence interval

**CRF** case report form

**CTR** clinical trial report

**EMA** European Medicines Agency

**FAS** full analysis set

**FDA** US Food and Drug Administration

**FPG** fasting plasma glucose

ICH International Council on Harmonization

LR logistic regression

**LPLT** last patient last treatment

**LPLV** last patient last visit

MAR missing at random

**MCMC** Markov Chain Monte Carlo

MImultiple imputation

**NBR** negative binomial regression

PK pharmacokinetics

SAS safety analysis set

s.c. subcutaneous Statistical analysis plan Date: 11 September 2020 | Novo Nordisk Trial ID: NN9535-4506

UTN: U1111-1224-5162 EudraCT No: 2018-004529-96


Version: Status: Page:

1.0 Final


SU sulfonylureas

T2D Type 2 diabetes

TFL Tables, figures and listings

w/owithout

#### **6.2 Appendix 2: Changes to protocol-planned analyses**

Corrected the end of the in-trial observation period, from end-of-treatment visit (V10) to the followup visit (P11).

A schematic overview of the estimands has been provided, see <u>Table 1</u>.

Clarification in section 2 that statistical testing is performed for each estimand strategy separately.

A clarification of rescue medication has been included, see section 4.

A two-way tipping point sensitivity analysis has been added based on feedback from FDA, see sections <u>5.3.2.2</u> and <u>5.4.1.2</u>.

Subgroup analyses have been included, see section 5.7.1, as well as a subpopulation analysis, see section 5.7.2.

#### 6.3 Appendix 3: Definition and calculation of endpoints, assessments and derivations

Table 6 **Endpoints** 

| Type | Title | Time frame | Unit |
|---|---|---|---|
| Primary endpoint | Change from baseline (week 0) to week 40 in glycosylated haemoglobin (HbA <sub>1c</sub> ) | From baseline (week 0) to week 40 | % |
| Confirmatory secondary endpoint | Change from baseline (week 0) to week 40 in body weight | From baseline (week 0) to week 40 | kg |
| Supportive secondary endpoint | Change from baseline (week 0) to week 40 in fasting plasma glucose | Week 40 | mmol/L |
| Supportive secondary endpoint | Change from baseline (week 0) to week 40 in BMI | Week 40 | kg/m <sup>2</sup> |
| Supportive secondary endpoint | Change from baseline (week 0) to week 40 in waist circumference | Week 40 | cm |
| Supportive secondary endpoint | HbA <sub>1c</sub> < 7.0% (53 mmol/mol) | Week 40 | Yes/no |
| Supportive secondary endpoint | $HbA_{1c} \le 6.5\%$ (48 mmol/mol) | Week 40 | Yes/no |
| Supportive secondary endpoint | Weight loss ≥ 5 kg | Week 40 | Yes/no |

 Statistical analysis plan
 Date:
 11 September 2020
 Novo Nordisk

 Trial ID: NN9535-4506
 Version:
 1.0

 UTN: U1111-1224-5162
 Status:
 Final

 EudraCT No: 2018-004529-96
 Page:

| Type | Title | Time frame | Unit |
|---|---|---|---|
| Supportive secondary endpoint | Weight loss ≥ 10 kg | Week 40 | Yes/no |
| Supportive secondary endpoint | Number of treatment emergent severe or blood glucose confirmed symptomatic hypoglycaemic episodes from baseline (week 0) to week 40 | From week 0 to week 40 | Count |
| Supportive secondary endpoint | Change from baseline (week 0) to week 40 in pulse | From week 0 to week 40 | bpm |

# 7 References

1. Little RJA, Rubin DB. Statistical analysis with missing data. New York: Wiley. 1987. xiv, 278 p. p.



# Memo

From:

To:

Whom it may concern

Date: 28-Aug .2020

Ref.:

# Identification and presentation of Areas of Special Interest for NN9535-4506 – Memo version [2.0] – Task 088

This document aims to provide an overview of MedDRA queries (SMQs and NNMQs) in relation to CTR for the above trial

Areas of special interest are identified as outlined in the table below in MedDRA version [23.0]. Please make sure that no duplicate Preferred Terms are included in any of the separate searches.

If the Safety area of special interest is covered by a custom query (e.g. NNMQ) the text included in the table under 'Safety Area of Special Interest' should be included as the **CQNAM** in the SAS data set (left blank if SMQ).

If the Safety area of special interest is covered by a SMQ, the title of the SMQ should be included as the **SMQNAM** in the SAS data.

| N | Safety Area of Special<br>Interest (if defined by<br>an NNMQ, CQNAM in<br>SAS dataset) | Search criteria by NNMQ, SMQ, SOC<br>and/or specific Preferred Terms (if<br>defined by SMQ, SMQNAM in SAS<br>dataset) | Scope / Filter - include scope for each component (tick one per area) |
|---|---|---|---|
| 1 | Gastrointestinal adverse events | NNMQ GI SOC | <ul><li>☑ Primary terms only</li><li>☐ Both primary and secondary term</li></ul> |
| 2 | Cardiovascular disorders | NNMQ Cardiovascular disorders | <ul><li>☑ All terms</li><li>☐ Narrow term only</li></ul> |
| 3 | Acute gallstone disease | NNMQ Gallbladder related disorders | <ul><li>☐ All terms</li><li>☒ Narrow term only</li></ul> |
| 4 | Pancreatitis | NNMQ Pancreatitis | ☐ All terms ☐ Narrow term only |
| 5 | Acute renal failure | SMQ Acute renal failure | <ul><li>☐ All terms</li><li>☒ Narrow term only</li></ul> |
| 6 | Diabetic retinopathy adverse events | NNMQ Retinopathy phase 3a<br>- single PTs | ⊠All terms □ Narrow term only |
| 7 | Hepatic disorders | SMQ Drug related hepatic disorders | Comprehensive search |
| 8 | Allergic reactions | NNMQ Allergic reactions | ☐ All terms |

| | | | ☑ Narrow term only |
|---|---|---|---|
| 9 | Medication<br>error/overdose | SMQ Medication error,<br>NNMQ Abuse/Misuse,<br>NNMQ Overdose | <ul><li>☑ All terms</li><li>☐ Narrow term only</li></ul> |
| | | | Duplicate terms should be included only once |
| 10 | Rare events | NNMQ Rare | ☑ All terms |
| | | | ☐ Narrow term only |
| | | | Excluding terms caught in other searches |
| 11 | Neoplasms | NNMQ Neoplasms | ☑ All terms |
| | | | ☐ Narrow term only |
| 12 | Malignant neoplasms | SMQ Malignant tumours | ☐ All terms |
| | | | ☑ Narrow term only |
| 13 | Injection site reaction | NNMQ Injection site reaction | ☑ All terms |
| | | | □ Narrow term only |
| 14 | Suspected transmission | NNMQ Transmission | ☑ Primary terms only |
| | of an infectious agent | | ☐ Both primary and secondary term |

| Memo<br>version | MedDRA version | Description of change |
|---|---|---|
| 1.0 | 23.0 | This is the first version of memo. |
| | | To be used for task 088 |
| 2.0 | 23.0 | Memo has been updated to include the diabetic retinopathy phase 3a search instead of retinal disorders which is in agreement with a safety committee decision taking 2017-09-08. The phase 3a search is using MedRA v. 13.1 and it is recognised that PT terms may have been demoted or other changes when used in data coded in the current version of MedDRA is affecting the output. |

| NN9535 | | Date: | 04 December 2020 | Novo Nordisk |
|---|---|---|---|---|
| NN9535-4506 | CONFIDENTIAL | Version: | 1.0 | |
| Clinical Trial Report | | Status: | Final | |
| - | | Page: | 1 of 229 | |

# **Table of contents**

| | Page |
|---------------------------------------------------------|------|
| 1. Pre-defined MedDR A search - list of preferred terms | 2 |

| Novo Nordisk | |
|-----------------------|-------------|
| Final | 2 of 229 |
| Status: | Page: |
| 04 December 2020 | 1.0 |
| Date: | Version: |
| Clinical Trial Report | - |
| NN9535 | NN9535-4506 |

| 1: Pre-defined MedDRA search - list of preferred terms | eferred terms |
|--------------------------------------------------------|----------------|
| Pre-defined MedDRA search | Preferred term |

Acute gallstone disease

```
AIDS cholangiopathy
Ampulla of Vater stenosis
Autoimmune cholangitis
Bile culture positive
Bile culture positive
Bile duct pressure increased
Bile duct pressure increased
Bile duct stenosis traumatic
Bile duct stenosis traumatic
Bile duct stenosis traumatic
Bile duct stenosis traumatic
Bile duct stenosis complication
Bile duct stenosis complication
Bile output decreased
Bile output abnormal
Bile output increased
Bile output increased
Bile output increased
Bile output increased
Bile output decreased
Bile output increased
Bi
```

| Novo Nordisk | | 1 |
|---|---|---|
| Final | 3 of 229 | |
| Status: | Page: | |
| 04 December 2020 | 1.0 | |
| Clinical Trial Report | 1 | f preferred terms |
| NN9535 | NN9535-4506 | Pre-defined MedDRA search - list of preferred |

Preferred term

Acute gallstone disease

Pre-defined MedDRA search

Biloma
Biloma rupture
Biloma rupture
Biloma rupture
Bilopsy pallbladder abnormal
Blopsy gallbladder abnormal
Blood bilirubin abnormal
Blood bilirubin increased
Cholangiectasis acquired
Cholangicis increased
Cholangitis chronic
Cholangitis chronic
Cholangitis infective
Cholangitis infective
Cholangitis infective
Cholangitis infective
Cholangitis infective
Cholangitis infective
Cholangitis infective
Cholacystitis chronic
Cholacystitis infective
Cholacystitis infective
Cholacystitis infective
Cholacystitis infective
Cholacystopram oral abnormal
Cholacystopram intravenous abnormal
Cholacystopram intravenous
Cholacystopram intravenous
Cholacystopram intravenous
Cholacystopram intravenous
Cholacochoctomy
Cholacochoctomy
Cholacochoctomy
Cholacochoctomy
Cholacochoctomy
Cholacochoctomy
Cholacochoctomy
Cholacochoctomy
Cholacitais migration
Cholalithiasis obstructive
Cholalithiasis obstructive
Cholactasis of pregnancy
Cholactasis of pregnancy
Cholactasis
Cholactasis of pregnancy
Cholactasis of pregnancy
Cholactasis
Cholac
| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 4 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I I |

Acute gallstone disease

Gallbladder cholesterolosis
Gallbladder disorder
Gallbladder enlargement
Gallbladder enlargement
Gallbladder fistula
Gallbladder fistula repair
Gallbladder fistula repair
Gallbladder hyperfunction
Gallbladder injury
Gallbladder motocole
Gallbladder operation
Gallbladder operation
Gallbladder operation
Gallbladder operation
Gallbladder operation
Gallbladder vorices
Gallbladder varices
Gallbladder varices
Gallbladder varices
Gallbladder varices
Gallbladder fistula
Gallbladder fistula
Gallbladder fistula
Gallbladder operation
Gallbladder operation
Gallbladder fisture
Hepatobilary infection
Hepatobilary infection
Hepatobilary infection
Hyperplastic cholecystitis
Ischaemic cholestatic
Jaundice extrahepatic obstruction
Immune-mediated cholanitis
Ischaemic cholestatic
Jaundice extrahepatic obstruction
Fanceatobilary sphincterotomy
Parenteral nutrition associated liver disease
Ferforation bile duct
Forcelain gallbladder
Forcelain gallbladder
Forcelain gallbladder
Forcelain gallbladder
Forcelain fist bile fielek

| NN9535<br>NN9535-4506 | Clinical Trial Report<br>- | Date: | 04 December 2020 Status:<br>1.0 Page: | Final 5 of 229 | Final Novo Nordisk<br>f 229 |
|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | |
| Acute gallstone disease | Primary biliary cholangitis Pseudocholelithiasis Recurrent pyogenic cholangitis Reynold's syndrome Sphincter of Oddi dysfunction Ultrasound biliary tract abnormal Vanishing bile duct syndrome X-ray hepatobiliary abnormal | langitis<br>s<br>cholangitis<br>ysfunction<br>tract abnormal<br>syndrome<br>abnormal | | | |

Acquired C1 inhibitor deficiency Azotaemia
Azotaemia
Continuous haemodiafiltration
Dialysis
Foetal renal impairment
Haemodialysis
Haemofiltration
Neonatal anuria
Nephropathy toxic
Oliguria
Peritoneal dialysis
Frerenal failure
Renal failure
Renal failure
Renal failure
Renal impairment
Renal impairment
Renal impairment
Renal impairment subacute kidney injury Acute kidney injury Acute phosphate nephropathy Anuria Allergic reactions

Acute renal failure

Acute generalised examblemations Administration related reaction Administration site dermatitis Administration site dermatitis
Administration site hypersensitivity
Administration site reach
Administration site recall reaction
Administration site recall reaction
Administration site vasculitis
Allergic bronchitis
Allergic cough
Allergic cough
Allergic cough
Allergic cough
Allergic cough
Allergic cough

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 6 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Allergic gastroenteritis
Allergic gastroenteritis
Allergic keratitis
Allergic ceratitis
Allergic octitis externa
Allergic ottiss media
Allergic ottiss media
Allergic ottiss media
Allergic traction to excipient
Allergic respiratory disease
Allergic respiratory disease
Allergic respiratory symptom
Allergic respiratory symptom
Allergic respiratory symptom
Allergic sinusitis
Allergic respiratory symptom
Allergy alert test positive
Allergy to immunoglobulin therapy
Allergy to surgical sutures
Allergy to vaccine
Analyblactic reaction
Anaphylactic reaction
Anaphylactic reaction
Anaphylactic treatment
Anaphylactic treatment
Anaphylactic shock
Anaphylactic shock
Anaphylactic shock
Anaphylactic shock
Anaphylactic shock
Anaphylactic shock
Anaphylactic treatment
Anaphylactic treatment
Anaphylactic shock
Anaphylactic shock
Anaphylactic treatment
Anaphylactic treatment
Antiallergic therapy
Antiallergic therapy
Antiallergic therapy
Antiallergic therapy
Antiallergic therapy
Antiallergic site askersensitivity
Application site tash
Application site vasculitis
Application site uraciaria
Application site uraciaria
Application site uraciaria
Application site vasculitis
Archiris allergic
Actoric cough
Actoric
Actoric Actoric Actoric
Actoric Actoric Actoric
Actoric Actoric Cough
Actoric Cough

| NN9535-4506 - Version: | Date: 04 December 2020 Version: 1.0 | 720 Status:<br>1.0 Page: 7 | Final <b>Novo N</b> 7 of 229 |
|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | - | - | _ |

Nordisk

Allergic reactions

Pre-defined MedDRA search

Blood immunoglobulin E abnormal
Blood immunoglobulin E increased
Bromoderma
Bromoderma
Bullous haemorrhagic dermatosis
Catheter site dezema
Catheter site eczema
Catheter site nash
Catheter site wypersensitivity
Catheter site utticaria
Catheter site utticaria
Catheter site vasculitis
Catheter site vasculitis
Catheter site utticaria
Catheter site utticaria
Catheter site utticaria
Catheter site utticaria
Catheter site utticaria
Catheter site utticaria
Catheter site utticaria
Catheter site organia
Catheter site utticaria
Catheter site organia
Catheter site ocommities
Chronic hyperplastic cosinophilic sinusitis
Chromoral codema
Circumoral codema
Confunctival codema
Contrast media reaction
Contrast media reaction
Contrast media reaction
Contrast media reaction
Contrast media reaction
Contrast media reaction
Contrast sconfact
Contrastiis aconfact
Dermatitis acopic
Dermatitis sexfoliative
Dermatitis herpetiformis
Dermatitis herpetiformis
Dermatitis herpetiformis
Dermatitis infected
Dermatitis infected
Dermatitis procriasiform
Device allergy
Dialysis membrane reaction
Distributive shock
Documented hypersensitivity to administered

product
Drug eruption
Drug hypersensitivity
Drug provocation test

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 8 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ı |

Drug reaction with eosinophilia and systemic symptoms
Eczema infantile
Eczema infantile
Eczema nummular
Eczema vecinatum
Eczema weeping
Encephalitis allergic
Encephalitis allergic
Encephalitis allergic
Encephalitis bullosa
Epidermal necrosis
Explication ocelema
Erythema moultiforme
Erythema moultiforme
Erythema moulting
Explication ocelema
Erythema necema
Explication ocelema
Experimation ocelema
Face ocelema
Fixed eruption
Gingival ocelema
Gingival ocelema
Gingival ocelema
Gingival ocelema
Gingival sepullang
Gleich's syndrome
Haemorrhagic urticaria
Hand dermatitis
Henoch-Schonlein purpura
Hereditary anglocedema with Cl esterase inhibitor
Geficiency
Hypersensitivity myocarditis
Hypersensitivity wasculitis
Hypersensitivity wasculitis
Hypersensitivity wasculitis
Idiopathic urticaria

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final Novo |
|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 9 of 229 |
| Pre-defined MedDRA search - list of preferred | f preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | |

Immune Voice and continue induments to the analysis of the area in implant site hypersensitivity implant site hypersensitivity implant site rash implant site are not a reach incision site dermatitis incision site and hypersensitivity reaction infusion related reaction infusion site dermatitis infusion site eczema infusion site eczema infusion site rash infusion site rash infusion site racall reaction infusion site urticaria infusion site dermatitis injection site dermatitis injection site eczema injection site recall reaction injection site recall reaction injection site recall reaction injection site urticaria injection site vasculitis injection site vasculitis injection site vasculitis instillation site vasculitis instillation site vasculitis instillation site rash instillation site rash instillation site rash instillation site rash intestinal angioedema Immediate post-injection reaction Immune thrombocytopenia Immune tolerance induction Iodine allergy
Kaposi's varicelliform eruption
Kounis syndrome
Laryngeal oedema
Laryngitis allergic Laryngotracheal oedema Limbal swelling Laryngospasm

Lip oedema Lip swelling Mast cell degranulation present Medical device site dermatitis

vo Nordisk

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | 1.0 Page: | 10 of 229 |
| Pre-defined MedDRA search - list of preferred | f preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | |

Nutritional rash
Nutritional supplement allergy
Oculomecocutaneous syndrome
Oculorespiratory syndrome
Oculorespiratory syndrome
Oculorespiratory syndrome
Oral allergy syndrome
Oropharyngeal blistering
Oropharyngeal swelling
Palatal ocdema
Oropharyngeal swelling
Palatal ocema
Palatal welling
Palsaded neutrophilic granulomatous dermatitis
Palpable purpura
Palsaded neutrophilic granulomatous dermatitis
Palpable purpura
Palsaded swelling
Palsaded swelling
Palsaded swelling
Parioral dermatitis
Periorbital swelling
Procedural swelling
Procedural Medical device site eczema
Medical device site hypersensitivity
Medical device site rash
Medical device site recall reaction
Medical device site recall reaction
Mouth swelling Muccoutaneous rash Multiple allergies Nephritis allergic Nikolsky's sign Nodular rash

| NN9535<br>NN9535-4506 | Clinical Trial Report<br> - | Date: 0 Version: | 1.0 December 2020 | Status:<br>Page: | Final<br>11 of 229 | Final <b>Novo Nordisk</b><br>if 229 |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | st of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Rash pustular
Rash rubelliform
Rash vacialiform
Rash vesicular
Reaction to colouring
Reaction to excipient
Reaction to preservatives
Reaction to preservative
Soleritis allergic
Scrotal dermatitis
Scleritis allergic
Scrotal odematitis
Skin necrosis
Skin necrosis
Skin reaction
Skin reaction
Skin reaction
Skin reaction
Skin test positive
Solvent sensitivity
Stoma site rash
Scoma site rash
Scoma site rash
Swelling of eyelid

Jourge occasion of the control of th

| NN9535<br>NN9535-4506<br>Pre-defined MedDRA search - list of | Clinical Trial Report | Date: | 04 December 2020 Status:<br>1.0 Page: | Final No. 12 of 229 | Novo Nordisk |
|---|---|---|---|---|---|
| )<br>1<br>1 | Preferred term | | | | |
| Allergic reactions | Urticaria cholinergic Urticaria chronic Urticaria contact Urticaria papular Urticaria pigmentosa Urticaria pigmentosa Urticaria pigmentosa Urticarial dermatitis Urticarial dermatitis Urticarial dermatitis Urticarial dermatitis Vaccination site eczema Vaccination site ercena Vaccination site rash Vaccination site rash Vaccination site rash Vaccination site rash Vaccination site vasculitis Vaccination site vasculitis Vaccination site vascules Vaccination site vascules Vaccination site vascules Vaccination site vascules Vaccination site vascules Vasculitic rash Versal puncture site rash Vessel puncture site rash Vessel puncture site rash Vulval ulceration Vulval ulceration Vulvovaginal ulceration Vulvovaginal ulceration | olinergic nronic nntact pular yysical gmentosa ssiculosa lermatitis saculitis site eczema site eczema site exfoliation site reash site reash site recall reaction site urticaria site vesicles site vesicles ration ash ure site rash | | | |
| Cardiovascular disorders | Acute kidney injury Anuria Neonatal anuria Prerenal failure Renal failure Renal failure Renal failure Renal failure Administration site vasculitis Anaphylactic reaction Anaphylactic transfusion reaction Anaphylactic transfusion reaction Anaphylactid shock Anaphylactid shock Anaphylactid shock | y atal ijury e vasculitis ion fusion reaction ttion | | | |

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 13 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | t of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Anti-neutrophil cytoplasmic antibody positive vasculitis
Application site vasculitis
Circulatory collapse
Cutaneous vasculitis
Distributive shock
Eosinophilic granulomatosis with polyangiltis
Henoch-Schonlein purpura nephritis
Henoch-Schonlein purpura nephritis
Henoch-Schonlein purpura nephritis
Heparin-induced thrombocytopenia
Hypersensitivity myocarditis
Infusion site vasculitis
Infusion site vasculitis
Infusion site vasculitis
Infusion site vasculitis
Infusion site vasculitis
Vounis syndrome
Palpable purpura
Procedural shock
Shock

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 14 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | 1 1 |

Amyloid related imaging abnormalities
Amyloid related imaging
abnormality-microhaemorrhages and haemosiderin
deposits
Amyloid related imaging
abnormality-oedema/effusion
Andersen-Tawii syndrome
Angina unstable
Angina unstable
Angina unstable
Angina unstable
Angina unstable
Angina unstable
Angina unstable
Angiogram abnormal
Angiogram peripheral abnormal
Angiogram peripheral abnormal
Angiogram peripheral abnormal
Anti-glomerular basement membrane disease
Anti-glomerular basement membrane disease
Anti-glomerular basement membrane disease
Anti-glomerular basement membrane disease
Anti-glomerular basement membrane disease
Antibody test positive
Arrhythmia neonatal
Arrhythmia neonatal
Arrhythmia supraventricular
Arrhythmia supraventricular
Arrhythmia supraventricular
Arrhythmia supravention
Arterial bypass occlusion
Arterial bypass occlusion
Arterial bypass socclusion
Arterial bypass socclusion
Arterial careft
Arterial stent insertion
Arterial stent insertion
Arterial stent insertion
Arterial therapeutic procedure

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Novo |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | 1.0 Page: | 15 of 229 | |
| Pre-defined MedDRA search - list of preferred | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Atrioventricular block
Atrioventricular block
Atrioventricular block complete
Atrioventricular block first degree
Atrioventricular block second degree
Atrioventricular conduction time shortened
Atrioventricular dissociation
Atrioventricular node dispersion
Atrioventricular node dispersion
Atrioventricular node dispersion
Atrioventricular node dispersion
Atrioventricular node Balinction
Autoimmune myocarditis
Axillary vein thrombosis
BRASH syndrome
Balint's syndrome Atrial appendage cloure
Atrial appendage resection
Atrial appendage resection
Atrial enlargement
Atrial fibrillation
Atrial flutter
Atrial hypertrophy
Atrial natriuretic peptide abnormal
Atrial parasystole
Atrial persone increased
Atrial persone increased
Atrial septal defect acquired
Atrial thombosis Arteritis
Arteritis coronary
Artificial blood vessel occlusion
Artificial heart implant
Ascites Arterial thrombosis
Arteriogram abnormal
Arteriogram carotid abnormal
Arteriogram coronary abnormal
Arteriosclerosis coronary artery Arteriotomy
Arteriovenous fistula occlusion
Arteriovenous fistula thrombosis
Arteriovenous graft thrombosis Atherosclerotic plaque rupture Arteriospasm coronary Atherectomy

o Nordisk

| Novo Nordisk | | 1 |
|---|---|---|
| Final | 16 of 229 | |
| Status: | Page: | |
| 04 December 2020 | 1.0 | |
| Clinical Trial Report | 1 | f preferred terms |
| N9535 | N9535-4506 | Pre-defined MedDRA search - list of preferred terms |

Cardiovascular disorders

Pre-defined MedDRA search

Basal ganglia haematoma
Basal ganglia haemcrhage
Basal ganglia infarction
Basal ganglia infarction
Basal ganglia infarction
Basal ganglia infarction
Basal ganglia infarction
Basilar artery aneurysm
Basilar artery perforation
Blood brain barrier defect
Blood creatine phosphokinase MB increased
Blood creatine phosphokinase increased
Blood creatine phosphokinase increased
Blood creatine phosphokinase increased
Blood creatine phosphokinase increased
Blood pressure diastolic decreased
Blood pressure fluctuation
Blood pressure systolic abnormal
Blood pressure systolic increased
B

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| IN9535-4506 | | Version: | 1.0 | Page: | 17 of 229 | |
| Pre-defined MedDRA search - list of preferred | preferred terms | | | | | |

Pre-defined MedDRA search

Brain natriuretic peptide abnormal
Brain stem embolism
Brain stem natatoma
Brain stem haematoma
Brain stem haematoma
Brain stem infarction
Brain stem infarction
Brain stem microhaemia
Brain stem microhaemorrhage
Brain stem microhaemorrhage
Brain stem fironaemorrhage
Brain stem fironaemorrhage
Brain stem fironaemorrhage
Brain stem broke
Brain stem broke
Brain stem broke
Brain stem broke
Brain stem broke
Brain stem fironaemorrhage
Brain stem fironaemorphore
Bundle branch block
Bundle branch block bilateral
Bundle branch block left
Bundle branch block right

Preferred term

CARASIL syndrome
CSF bilirubin positive
CSF red blood cell count positive
CT hypotension complex
Capillaritis
Capsular warning syndrome
Cardiac amyloidosis

Cardiac amyllucats
Cardiac arrest neonatal
Cardiac arrest neonatal
Cardiac arrest neonatal
Cardiac carhosis
Cardiac cirrhosis
Cardiac death
Cardiac device reprogramming
Cardiac device reprogramming
Cardiac dystunction
Cardiac factorophysiologic study abnormal
Cardiac fallure
Cardiac fallure chronic
Cardiac fallure chronic
Cardiac fallure high output
Cardiac fallure high output
Cardiac filutter

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 18 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | : preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

cardiac hypertrophy

Cardiac imaging procedure abnormal

Cardiac index abnormal

Cardiac index abnormal

Cardiac index increased

Cardiac monitoring abnormal

Cardiac monitoring abnormal

Cardiac output decreased

Cardiac output decreased

Cardiac output decreased

Cardiac perfusion defect

Cardiac septal hypertrophy

Cardiac septal hypertrophy

Cardiac septal hypertrophy

Cardiac sets test abnormal

Cardiac ventricular scarring

Cardiac ventricular scarring

Cardiac ventricular scarring

Cardiac ventricular strest

Cardiac ventriculogram left abnormal

Cardiac ventriculogram strest

Cardiac ventriculogram strest

Cardiac ventriculogram left abnormal

Cardiac ventriculogram strest

Cardiac ventriculogram strest

Cardiac ventriculogram left abnormal

Cardiocrespiratory arrest neonatal

Cardiomopathy acute

Cardiomyopathy alcoholic

Cardiothoracic ratio increased

Cardiothoracic ratio increased

Cardiovascular disorder

Cardiovascular function test abnormal

Cardiovascular insufficiency

Cardiovascular insufficiency

Carctid aneurysm rupture

Carctid aneurysm rupture

Carctid aneurysm rupture

Carctid arterial embolus

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 Page: | age: | 19 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Carotid arteriosclerosis
Carotid artery aneurysm
Carotid artery bypass
Carotid artery dissection
Carotid artery dissection
Carotid artery dolichoectasia
Carotid artery perforation
Carotid artery perforation
Carotid artery perforation
Carotid artery sestenosis
Carotid artery thrombosis
Central bradycarda
Central bradycarda
Central artery thrombosis
Central artery thrombosis
Cerebellar artery thrombosis
Cerebellar macrothage
Cerebellar haemarchage
Cerebellar ischaemia
Cerebellar ischaemia
Cerebellar incroheemorrhage
Cerebral aneurysm ruptured syphilitic
Cerebral arterioxenous malformation haemorrhagic
Cerebral arterioxelerosis

| NN9535<br>NN9535-4506 | Clinical Trial Report<br> - | Date: ( | 04 December 2020 Status:<br>1.0 Page: | Status:<br>Page: | Final<br>20 of 229 | Final <b>Novo Nordisk</b> of 229 |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | t of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ı |

Cerebral artery restenosis
Cerebral artery stenosis
Cerebral artery stenosis
Cerebral artery stenosis
Cerebral capillary telangiectasia
Cerebral capillary telangiectasia
Cerebral cavernous malformation
Cerebral congestion
Cerebral endovascular aneurysm repair
Cerebral das embolism
Cerebral haemorrhage neonatal
Cerebral haemorrhage foetal
Cerebral haemorrhage neonatal
Cerebral haemorrhage neonatal
Cerebral haemorrhage neonatal
Cerebral infarction
Cerebral infarction
Cerebral infarction
Cerebral infarction
Cerebral microampolism
Cerebral microampolism
Cerebral microampolism
Cerebral microampolism
Cerebral microampolism
Cerebral microampolism
Cerebral septic infarct
Cerebral septic infarct
Cerebral trombosis
Cerebral venous thrombosis
Cerebral venous thrombosis
Cerebral venous thrombosis
Cerebral venous thrombosis
Cerebral venous thrombosis
Cerebral venous thrombosis
Cerebral venous thrombosis
Cerebral venous malformation
Cerebrovascular accident prophylaxis
Cerebrovascular accident prophylaxis
Cerebrovascular accident prophylaxis
Cerebrovascular insufficiency
Cerebrovascular insufficiency
Cerebrovascular spendanencysm
Cerebrovascular spendianencysm
Cerebrovascul

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 21 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I I |

Chagas' cardiomyopathy
Charcot-Bouchard microaneurysms
Chest X-ray abnormal
Choroidal infarction
Choroidal infarction
Chronic cerebrospinal venciular failure
Chronic cerebrospinal venciular
Chronic pigmented purpura
Chronic pigmented purpura
Chronic pigmented purpura
Chronic pigmented purpura
Chronic pigmented purpura
Chronic pigmented purpura
Chronic ratery occlusion
Compan's syndrome
Collateral circulation
Computerised tomogram coronary artery abnormal
Computerised tomogram thorax abnormal
Computerised tomogram thorax abnormal
Congenital cerebrovascular anomaly
Congenital supraventricular tachycardia
Congenital supraventricular tachycardia
Congestive cardiomyopathy
Congestive cardiomyopathy
Congestive hepatopathy
Cor pulmonale acute
Cor pulmonale chronic
Coronary artery compression
Coronary artery disease
Coronary artery disease
Coronary artery embolism
Coronary artery restenosis
Coronary artery restenosis
Coronary artery thrombosis
Coronary artery thrombosis
Coronary artery thrombosis
Coronary artery thrombosis
Coronary artery thrombosis
Coronary artery thrombosis
Coronary bypass thrombosis
Coronary bypass thrombosis
Coronary bypass thrombosis

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 22 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | : preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ı |

Coronary no-reflow phenomenon
Coronary ostial stenosis
Coronary schascular stenosis
Coronary steal stenosis
Coronary steal syndrome
Coronary steal syndrome
Coronary vascular graft occlusion
Coronary vascular graft occlusion
Coronary vascular graft stenosis
Coxsackie carditis
Coxsackie myocarditis
Coxsackie myocarditis
Cryoglobulins present
Decreased ventricular
Decreased uschaemin extention
Device embolisation
Device embolisation
Device embolisation
Device embolisation
Device eralated thrombosis
Diabetic coronary microangiopathy
Diabetic coronary microangiopathy
Diabetic coronary microangiopathy
Diabetic orconary microangiopathy
Diabetic arteritis
Diatetion atcilits
Diatetion atcilits
Diatetion atcilits
Diatetion atcilits
Disseminated intravascular coagulation
Disseminated intravascular coagulation
Disseminated intravascular scale
Disseminated intravascular coagulation
Disseminated intravascular coagulation
Disseminated intravascular coagulation
Disseminated intravascular accompanient
Disseminated intravascular coagulation
Disseminated intravascular coagulation
Disseminated intravascular coagulation
Disseminated intravas

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 23 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | E preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Electrocardiogram P wave abnormal Electrocardiogram P wave abnormal Electrocardiogram P R prolongation Electrocardiogram PR segment depression Electrocardiogram PR shortened Electrocardiogram Q wave abnormal Electrocardiogram QT prolonged Electrocardiogram ST segment abnormal Electrocardiogram ST segment depression Electrocardiogram ST-T segment depression Electrocardiogram ST-T segment debression Electrocardiogram T wave inversion Electrocardiogram T wave inversion Electrocardiogram U wave inversion Electrocardiogram U wave bnormal Electrocardiogram U wave bnormal Electrocardiogram U wave shormal Electrocardiogram du-wave abnormal Electrocardiogram delta waves abnormal Electrocardiogram abnormal Electrocardiogram delta waves abnormal Electrocardiogram delta waves abnormal Electrocardiogram delta waves bnormal Electrocardiogram repolarisation abnormal Embolism arterial Endocardial fibrocardiis Endocardial Endocardiis Endocardiis Endocardiis Exercise electrocardiogram abnormal Exercise electrocardiogram abnormal Exercise electrocardiogram abnormal

| NN9535<br>NN9535-4506 | Clinical Trial Report<br> - | Date:<br>Version: | 04 December 2020 Status: 1.0 Page: | Status: Page: | Final <b>Novc</b> 24 of 229 |
|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred | f preferred terms | | | | |
| The Adriant Manitan | 0 + 1 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | | | | |

Eye infarction
Femoral artery embolism
Fluorescence angiogram abnormal
Fluorescence angiogram abnormal
Foetal arrhythmia
Foetal heart rate acceleration abnormality
Foetal heart rate deceleration abnormality
Foetal heart rate disorder
Foetal achyarrhythmia
Footil expudrome
Frederick's syndrome Haemorrhage coronary artery
Haemorrhage intracranial
Haemorrhagic adrenal infarction
Haemorrhagic cerebral infarction
Haemorrhagic infarction
Haemorrhagic stroke
Haemorrhagic stroke
Haemorrhagic transformation stroke
Haemorrhagic vasculitis
Haemorrhagic vasculitis
Haemorrhagic vasculitis
Haert alternation
Heart alternation
Heart rate abnormal
Heart rate decreased
Heart rate increased
Heart rate increased
Heart rate increased
Heart rate increased
Heart rate increased
Heart rate increased
Heart rate increased
Heart rate increased
Heart transplant
Heart transplant
Heart transplant
Heart transplant
Heart transplant
Hemianesthesia Giant cell myocarditis
Gonococcal heart disease
Goodpasture's syndrome
Graft thrombosis
Granulomatosis with polyangiitis
Granulomatosis with polyangiitis
HIV cardiomyopathy Extraischaemic cerebral haematoma External counterpulsation
Extra-axial haemorrhage
Extradural haematoma
Extradural haematoma evacuation Extrasystoles

Hemiasomatognosia

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final Novo A | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 25 of 229 | |
| Pre-defined MedDRA search - list of preferred | preferred terms | | | | | |

Cardiovascular disorders

Pre-defined MedDRA search

Hemiataxia
Hemidysaesthesia
Hemidysaesthesia
Hemidyperaesthesia
Hemidyperaesthesia
Hemidyperaesthesia
Hemidyperaesthesia
Hemidylegia
Hepatic artery embolism
Hepatic artery thrombosis
Hepatic infarction
Hepatic vein embolism
Hepatic vein embolism
Hepatic vein embolism
Hepatic vein for erflux
Hepatic vein for positive
Hunt and Hess scale
Hunt and Hess scale
Hypertensive cardiomyopathy
Hypertensive cardiomyopathy
Hypertensive creebrovascular disease
Hypotensive creebrovascular disease
Hypotensive crisis
Hypotensive crisis
Hypotensive crisis
Hypotensive crisis
Hypotricion
Iliac artery occlusion
Iliac artery occlusion
Iliac artery embolism
Iliac artery embolism
Iliac artery embolism
Iliac vein occlusion
Ilmoreased ventricular preload
Infarction
Infarction
Infarction
Infarction site thrombosis
Injection site thrombosis
Injection site thrombosis

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 26 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | , |
| Pre-defined MedDRA search | Preferred term | | | | | |

Inner ear infarction
Instillation site thrombosis
Internal capsule infarction
Internal carotid artery deformity
Intra-acrtic balloon placement
Intra-cerebral aneurysm operation
Intra-cardiac mass
Intra-cardiac pressure increased
Intra-cardiac pressure increased
Intra-cardiac pressure increased
Intra-cerebral haematoma evacuation
Intra-cranial haematoma evacuation
Intra-cranial aneurysm
Intra-cranial haematoma artery occlusion
Intra-cranial haematoma artery occlusion
Intra-cranial tumour haemorrhage
Intra-cranial mediomy
Ischaemic cardiomyopathy
Ischaemic cardiomyopathy
Ischaemic cardiomyopathy
Ischaemic stroke
Jugular vein distension
Ischaemic stroke
Jugular vein distension
Ischaemic stroke
Ischaemic stroke
Ischaemic cardiomal ectopic tachycardia
Kawasaki's disease
Isangerhans' cell histiocytosis
Isangerhans' cell histiocytosis
Isangerhans' cell histiocytosis
Isangerhans' cell histiocytosis
Isatraial wolume abnormal
Ieft atrial enlargement
Ieft atrial volume decreased
Ieft atrial volume increased
Ieft ventricular distation
Ieft ventricular distation

| NN9535 | Clinical Trial Report | Date: 04 | 4 December 2020 | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: 2 | 7 of 229 |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | |

Novo Nordisk

Cardiovascular disorders

Pre-defined MedDRA search

Left ventricular dysfunction
Left ventricular end-diastolic pressure decreased
Left ventricular end-diastolic pressure decreased
Left ventricular failure
Left ventricular heave
Lenegre's disease
Leriche syndrome
Long QT syndrome
Long QT syndrome
Long QT syndrome
Lower respiratory tract congestion
Magnetic resonance imaging thoracic abnormal
Madrial myocarditis
May-Thurner syndrome
Medical device site thrombosis
Medical device site vasculitis
Medical device site vasculitis
Mesenteric artery stent insertion
Mesenteric artery stent insertion
Mesenteric artery stent insertion
Mesenteric artery thrombosis
Mesenteric vascular insufficiency
Micrombolism
Micromodia Micromodia occlusion
Metabolic cardiomyopathy
Micromodia Gubler syndrome
Milard-Gubler syndrome

| Final Novo Nordisk | | |
|---|---|---|
| Fine | 28 of 229 | |
| Status | Page: | |
| 04 December 2020 | 1.0 | |
| Clinical Trial Report | 1 | f preferred terms |
| NN9535 | NN9535-4506 | Pre-defined MedDRA search - list of preferred t |

Cardiovascular disorders

Pre-defined MedDRA search

Modified Rankin score increased
Monoparesis
Monoparesis
Monopledia
Moyamoya disease
Multiple gated acquisition scan abnormal
Multiple gated acquisition syndrome
Multiple obscess
Mycardial calcification
Mycardial fibrosis
Mycardial librosis
Mycardial hypopertusion
Mycardial hypopertusion
Mycardial hypopertusion
Mycardial infarction
Mycardial increased
Mycardial necrosis marker increased
Mycardial necrosis marker increased
Mycardial stunning
Mycarditis hacterial
Mycarditis bacterial
Mycarditis bacterial
Mycarditis infectious
Mycarditis infectious
Mycarditis infectious
Mycarditis septic
Mycarditis septic
Mycarditis spotiitic
Mycarditis spotiilitic
Mycarditis spotiilitic
Mycarditis stoxoplasmal
Mycarditis toxoplasmal
Mycarditis toxoplasmal
Mycarditis score decreased
N-terminal prohormone brain natriuretic peptide
abnormal
N-terminal prohormone brain natriuretic peptide
Nceased scale score decreased
NH stroke scale score increased
NH stroke scale score increased
NH stroke scale score increased
NH stroke scale score increased
NH stroke scale score increased
NH stroke scale score fallure
Neonatal respiratory fallure
Neonatal respiratory fallure
Neonatal sinus bradycardia

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 29 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Neonatal sinus tachycardia
Neonatal tachyarrhythmia
Neonatal tachyarrhythmia
Neonatal tachyarrhythmia
Neoturia
Nocturia
Nocturia
Nodal arrhythmia
Nodal arrhythmia
Nodal arrhythmia
Nodal arrhythmia
Nodal rrhythm
Nodular vasculitis
Non-obstructive cardiomyopathy
Nonrassuring focatal heart rate pattern
Obssity cardiomyopathy
Nonrassuring focatal heart rate pattern
Obssity cardiomyopathy
Nonrassuring focatal heart rate pattern
Obstructive shock
Coular vasculitis
Ocdema due to cardiac disease
Ocdema blister
Ocdema blister
Ocdema blister
Ocdema blister
Ocdema brister
Ocdema cartery thrombosis
Ophthalmic artery thrombosis
Ophthalmic vein thrombosis
Ophthalmic vein thrombosis
Orthostations
Orthostatic hypotension
Ovarian vein thrombosis
Pacemaker syndrome
Pacemaker syndrome
Pacemaker syndrome
Pacemaker syndrome
Pacemaker syndrome
Papillary muscle disorder
Papillary muscle haemorrhage
Papillary muscle infarction
Parapolesis
Paraparesis
Paraparesis
Parasystole
Paresis

Paroxysmal arrhythmia

| Novo Nordisk | ı |
|---|---|
| Final 30 of 229 | |
| Status:<br>Page: | , |
| 04 December 2020<br>1.0 | |
| Date:<br>Version: | - |
| Clinical Trial Report | f preferred terms |
| NN9535<br>NN9535-4506 | Pre-defined MedDRA search - list of preferred terms |

Cardiovascular disorders

Pre-defined MedDRA search

Paroxysmal atrioventricular block
Pelvic venous thrombosis
Penile artery occlusion
Penile vein thrombosis
Perinatal stroke
Perinatal stroke
Perinatal atrevia andioplasty
Peripheral arterial reocclusion
Peripheral artery angioplasty
Peripheral artery angioplasty
Peripheral artery bypass
Peripheral artery bypass
Peripheral artery bypass
Peripheral artery bypass
Peripheral artery bypass
Peripheral artery thrombosis
Peripheral artery thrombosis
Peripheral artery thrombosis
Peripheral endarterectomy
Peripheral endarterectomy
Peripheral endarterectomy
Peripheral endarterection
Peripheral endarterection
Peripheral weelling
Peripheral wein occlusion
Peripheral woorscularisation
Peripheral woorscularisation
Peripheral woorscularisation
Plasama viscosity abnormal
Phebectomy
Pituitary infarction
Plasama viscosity abnormal
Pheumatic compression therapy
Polyarteritis nodosa
Polymyalgia rheumatica
Polymyalgia rheumatica
Polymyalgia rheumatica
Polymyalgia rheumatica
Portal vein cavernous transformation
Portal vein cavernous
Portal vein thrombosis
Port vendiac arrest syndrome
Portal vein thrombosis
Post angioplasty restenosis
Post syndrome
Post procedural myocardial infarction

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred | -<br> preferred terms | version. | 0:1 | 1 480. | 677 10 16 | |

Cardiovascular disorders

Pre-defined MedDRA search

Post procedural pulmonary embolism
Post procedural stroke
Post stroke depression
Post thrombotic syndrome
Post thrombotic syndrome
Postinfarction angina
Postpartum thrombosis
Postpartum thrombosis
Postpartum thrombosis
Postpartum thrombosis
Procerebral artery thrombosis
Procerebral artery thrombosis
Profundaplasty
Prohormone brain natriuretic peptide increased
Prosthetic cardiac valve thrombosis
Prosthetic cardiac valve thrombosis
Prosthetic cardiac valve thrombosis
Pulmonary artery thrombosis
Pulmonary artery thrombosis
Pulmonary artery thrombosis
Pulmonary endarterectomy
Pulmonary congestion
Pulmonary congestion
Pulmonary microemboli
Pulmonary microemboli
Pulmonary thrombosis
Pulmonary venous thrombosis
Pulmonary veno coclusive disease
Pulmonary veno coclusive disease
Pulmonary veno coclusive disease
Pulmonary veno coclusive disease
Pulmonary veno coclusive disease
Pulmonary veno coclusive disease
Pulmonary veno coclusive disease
Pulmonary veno starivity
Pulmonary veno coclusive disease
Pulmonary veno coclusive

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| IN9535-4506 | | Version: | 1.0 | Page: | 32 of 229 | |
| Pre-defined MedDRA search - list of preferrec | : preferred terms | | | | | |

Cardiovascular disorders

Pre-defined MedDRA search

Radiation associated cardiac failure
Radiation myocarditis
Radiation wasculitis
Radiation vasculitis
Rebound tachycardia
Renal artery occlusion
Renal artery thrombosis
Renal artery thrombosis
Renal vasculitis
Renal vasculitis
Renal vasculitis
Renal vasculitis
Renal vain embolism
Renal vain embolism
Renal vain embolism
Renal vain embolism
Renal vain embolism
Renal vain embolism
Renal vain embolism
Renal vain embolism
Renal vain embolism
Renal vain enthythmia magnitude decreased
Respiratory sinus arrhythmia magnitude decreased
Respiratory sinus arrhythmia magnitude increased
Respiratory sinus surhythmia magnitude increased
Respiratory sinus surhythmia magnitude increased
Respiratory endomosis
Retinal artery brombosis
Retinal artery thrombosis
Retinal vein occlusion
Retinal vein occlusion
Retinal vein occlusion
Retinal vein occlusion
Retinal vein occlusion
Retinal vein occlusion

Respiratory sinus arrnythmia magnitude increased Restenosis
Restinal artery embolism
Retinal artery occlusion
Retinal artery thrombosis
Retinal infarction
Retinal vascular thrombosis
Retinal vascular thrombosis
Retinal vein occlusion
Retinal vein occlusion
Retinal vein occlusion
Retinal vein encounties
Retinal vein coclusion
Retinal vein incomposis
Retinal vein occlusion
Retinal vein occlusion
Retinal vein occlusion
Retinal vein occlusion
Retinal vein forcedure
Revascularisation procedure
Revasible cerebral vasoconstriction syndrome
Reversible cerebral vasoconstriction Right atrial dilatation
Right atrial dilatation
Right atrial pressure increased
Right ventricle outflow tract obstruction
Right ventricle outflow tract obstruction
Right ventriclar dilatation
Right ventriclar dilatation

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 33 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Right ventricular dysfunction
Right ventricular ejection fraction
Right ventricular enlargement
Right ventricular fallure
Right ventricular fallure
Right ventricular heave
Right ventricular heave
Right ventricular systolic pressure decreased
Rught ventricular systolic pressure
Right ventricular systolic pressure
Right ventricular systolic pressure
Rught ventricular systolic pressure
Rught ventricular systolic pressure
Rught ventricular systolic pressure
Rught ventricular systolic pressure
Segmented hyalinising vasculitis
Segmented hyalinising vasculitis
Septic shock
Shock haemorrhagic
Shock haemorrhagic
Shock haemorrhagic
Shock hypoglycaemic
Spinal arrexy thrombosis
Spinal subdural haemorrhage
Spinal subdural haemorrhage
Spinal vascular disorder
Spinal subdural haemorrhage
Spinal vascular disorder
Spinal subdural haemorrhage
Spinal cord infarction
Spinal subdural haemorrhage
Spinal vessel confecutial anomaly
Spinal chrombosis
Splenic thrombosis
Splenic thrombosis

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 34 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ı |

Cardiovascular disorders

Superficial siderosis of central nervous system Subarachnoid haematoma Subarachnoid haematoma Subarachnoid haematoma Subarachnoid haemorrhage Bubclavian artery embolism Subclavian artery thrombosis Subclavian coronary steal syndrome Subclavian vein forclusion Subclavian vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Subdural haematoma evacuation Subdural haematoma evacuation Subdural haematoma evacuation Subdural haemorrhage neonatal Subendocardial ischeemia Superior sagittal sinus thrombosis Superior vena cava occlusion Superior vena cava syndrome Supraventricular extrasystoles Supraventricular tachyarrhythmia Splenic vein thrombosis Stoma site thrombosis Stress cardiomyopathy Stress echocardiogram abnormal Stroke in evolution Stroke volume decreased Sudden death

Systolic anterior motion of mitral valve Systolic dysfunction Tachycardia Tachycardia foetal Tachycardia induced cardiomyopathy Tachycardia paroxysmal Takayasu's arteritis Surgical vascular shunt Surgical ventricular restoration Susac's syndrome Tachyarrhythmia

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 35 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Temporal arteritis
Testicular infarction
Thalamus haemorrhage
Thandomotinis obliterans
Thromboembolectomy
Thromboembolectomy
Thrombophlebitis migrans
Thrombophlebitis menatal
Thrombophlebitis menatal
Thrombophlebitis neonatal
Thrombosis corpora cavernosa
Thrombosis in device
Thrombosis in device
Thrombosis prophylaxis
Thrombotic cerebral infarction
Thrombotic creepral infarction
Thrombotic diacretion
Thrombotic stroke
Thrombotic stroke
Thrombotic thrombotytopenic purpura
Thrombotic cardiomyopathy
Thrombotic stroke
Thrombotic stroke syndrome staphylococcal
Toxic shock syndrome staphylococcal
Toxic shock syndrome staphylococcal
Transient ischaemic attack
Transient ischaemic attack
Transient increased
Troponin I increased
Troponin I increased
Troponin I increased
Troponin I increased
Troponin I increased
Troponin I increased
Troponin I increased
Troponin thrombectomy
Tumour thrombectomy
Tumour thrombectomy
Tumour thrombectomy
Tumour thrombectomy
Tumour thrombectomy
Tumour thrombectomy
Ultrasound Opppler abnormal
Ultrasound coclusion

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | _ | Version: | 1.0 | Page: | 36 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Umbilical cord thrombosis
Vaccination site thrombosis
Vascular access site thrombosis
Vascular device occlusion
Vascular device occlusion
Vascular graft occlusion
Vascular graft thrombosis
Vascular predomeurysm thrombosis
Vascular predomeurysm thrombosis
Vascular predomeurysm thrombosis
Vascular predomeurysm thrombosis
Vascular stent occlusion
Vascular stent stenosis
Vascular stent stenosis
Vascular stent stenosis
Vascular stent stenosis
Vasculars nectotising
Vasculars nectotising
Vasculitis metrotisme
Vasculitis nectotising
Vasculitis nectotising
Vena cava filter insertion
Vena cava filter removal
Vena cava filter removal
Vena cava filter insertion
Venous angioplasty
Venous pressure jugular increased
Venous pressure jugular increased
Venous recanalisation
Venous recanalisation
Venous recanalisation
Venous thrombosis in pregnancy
Venous thrombosis neonatal
Ventricular arxipythmia

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 37 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Dro-dofined MedADBA sees | Draferrad to arm | | | | | I |

Ventricular asystole
Ventricular compliance decreased
Ventricular dysfunction
Ventricular dysfunction
Ventricular dyssynchrony
Ventricular enlargement
Ventricular enlargement
Ventricular fibrillation
Ventricular fibrillation
Ventricular hyperkinesia
Ventricular hyperkinesia
Ventricular parasystole
Ventricular parasystole
Ventricular parasystole
Ventricular remodelling
Ventricular remodelling
Ventricular remodelling
Ventricular recoparatia
Ventricular remodelling
Ventricular recoparatia
Ventricular recoparatia
Ventricular recoparatia
Ventricular recoparatia
Ventebral artery aneurysm
Vertebral artery occlusion
Vertebral artery perforation
Vertebral artery stenosis
Vertebral artery stenosis
Vertebrobasilar insulficiency
Vertebrobasilar stroke
Vertebro

| NN9535<br>NN9535-4506 | Clinical Trial Report | Date:<br>Version: | 04 December 2020 Status:<br>1.0 Page: | Final<br>38 of 229 | Final Novo Nordisk<br>f 229 |
|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | l 1 |

Diabetic retinopathy adverse events

Amaurosis
Visual acuity reduced transiently
Cystoid macular oedema
Diabetic blindness
Diabetic retinal oedema
Diabetic retinopathy
Diabetic retinopathy
Diabetic retinopathy
Macular ischaemia
Macular opedema
Macular opedema
Macular pseudohole
Macular pseudohole
Macular pseudohole
Macular pseudohole
Macular pseudohole
Retinal deposits
Retinal deposits
Retinal accomment
Retinal nemorrhage
Retinal neovascularisation
Retinal pallor
Retinal pallor
Retinal pallor
Retinal pallor
Retinal pallor
Retinal pallor
Retinal vascular occlusion
Retinopathy
Vitreal cells
Vitreal cells Vitreous detachment Vitreous haemorrhage Vitreous opacities

Bile output decreased Biliary ascites Biliary cirthosis Biliary cirthosis Biliary fibrosis Biliary conjugated abnormal

Bile output abnormal

Drug related hepatic disorders - comprehensive search (SMQ)  $\,$ 

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | 1.0 Page: | 39 of 229 |
| Pre-defined MedDRA search - list of preferred | of preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | |

Bilirubin conjugated increased

Jaundice cholestatic
Parenteral nutrition associated liver disease
Primary biliary cholangitis
Reynold's syndrome
X-ray hepatobiliary abnormal
Allergic hepatitis Suncleotidase increased
AST/ALT ratio abnormal
Acquired antithrombin III deficiency
Acquired factor IX deficiency
Acquired factor XI deficiency
Acquired hepatocerebral degeneration
Acquired protein S deficiency
Alanine aminotransferase abnormal
Ammonia abnormal
Ammonia increased
Anorectal varices Portal shunt procedure Portal vein cavernous transformation Bilirubin excretion disorder Blood bilirubin abnormal Blood bilirubin increased Immune-mediated cholangitis Cardiohepatic syndrome Congestive hepatopathy Hepatomegaly Hepatorenal failure Gallbladder varices Hepatitis cholestatic Hepatobiliary disease Hyperbilirubinaemia Cholestasis Jaundice Ascites Drug related hepatic disorders - comprehensive search (SMQ)
| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 40 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | 1 1 |

Anorectal varices haemorrhage

Drug related hepatic disorders - comprehensive search (SMQ)

Anti factor X activity abnormal
Anti factor X activity increased
Antithrombin III decreased
Aspartate aminotransferase abnormal
Aspartate aminotransferase abnormal
Aspartate aminotransferase abnormal
Aspartate aminotransferase increased
Aspartate aminotransferase abnormal
Aspartate aminotransferase increased
Asterixis
Autoimmune hepatitis
Bacteriacites
Benign hepatobiliary neoplasm
Benign hepatobiliary neoplasm
Benign hepatobiliary neoplasm
Bilirubin urine present
Blood alkaline phosphatase abnormal
Blood alkaline phosphatase increased
Blood alkaline phosphatase increased
Blood cholinesterase abnormal
Blood cholinesterase decreased
Blood thrombin abnormal
Blood thrombin abnormal
Blood thrombin decreased
Blood thrombin decreased
Blood thrombin abnormal
Child-Pugh-Turcotte score abnormal
Child-Pugh-Turcotte score increased
Cholangiosarcoma
Cholastatic liver injury
Cholestatic liver injury
Cholestatic liver injury
Cholestatic puritus
Chronic hepaticis
Coagulation factor IX level decreased
Coagulation factor IX level abnormal
Coagulation factor VI level abnormal
Coagulation factor VI level abnormal
Coagulation factor VI level abnormal
Coagulation factor VI level abnormal

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 41 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | E preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Coagulation factor X level decreased Drug related hepatic disorders - comprehensive search  $(\ensuremath{\mathsf{SMQ}})$ 

Coagulation factor decreased
Coma hepatic
Complications of transplanted liver
Computerised tomogram liver abnormal
Cryptogenic cirrhosis
Deficiency of bile secretion
Diabetic hepatopathy
Drug-induced liver injury
Drug-induced liver injury
Drug-induced liver injury
Coal nodular hyperplasia
Foctor hepaticuss abnormal
Galactose elimination capacity test decreased
Galactose elimination capaciton
Gastric varices lingation
Gastric varices haemorrhage
Gastric varices lingation
Gastric varices lingation
Gastric varices lingation
Gastric varices liver
Gastric varices liver
Gastric varices liver
Hemorrhagic accidences
Hemorrhagic decreased
Hemorrhagic decreased
Hepatic adenoma
Hepatic calcufication
Hepatic cancer metastatic
Hepatic cancer metastatic
Hepatic cancer recurrent
Hepatic cancer stage II

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 42 of 229 |
| Pre-defined MedDRA search - list of prefe | f preferred terms | | | | |

Final Novo Nordisk

Pre-defined MedDRA search

Preferred term

Hepatic cancer stage III Drug related hepatic disorders - comprehensive search (SMQ)

Hepatic neoplasm
Hepatic pain
Hepatic pain
Hepatic pain
Hepatic sequestration
Hepatic steatoriibrosis
Hepatic steatoriibrosis
Hepatic vascular resistance increased
Hepatic venous pressure gradient abnormal
Hepatic venous pressure gradient increased
Hepatitis acute
Hepatitis acute
Hepatitis chronic active
Hepatitis chronic persistent
Hepatitis toxio
Hepatitis toxio
Hepatitis toxic
Hepatobiliary cancer
Hepatobiliary cancer
Hepatobiliary cancer
Hepatobiliary cancer
Hepatobiliary cancer Hepatic cyst ruptured
Hepatic cyst ruptured
Hepatic encephalopathy
Hepatic encephalopathy prophylaxis
Hepatic enzyme abnormal
Hepatic enzyme increased
Hepatic failure
Hepatic fibrosis marker abnormal
Hepatic fibrosis marker increased
Hepatic fibrosis marker increased
Hepatic fibrosis marker increased
Hepatic fibrosis marker increased
Hepatic function abnormal
Hepatic haemangioma rupture
Hepatic haemangioma rupture
Hepatic haemangioma rupture
Hepatic haematoma
Hepatic lasion
Hepatic lesion
Hepatic lesion
Hepatic lesion Hepatic cancer stage IV Hepatic cirrhosis Hepatic cyst Hepatic mass Hepatic necrosis

| NN9535 | Clinical Trial Report | Date: 0 | 4 December 2020 Status: | tatus: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 P | Page: | 43 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Dre-defined MedARA | Drafarrad tarm | | | | | |

Drug related hepatic disorders - comprehensive Hepatobiliary neoplasm search (SMQ)

Hepatobiliary scan abnormal
Hepatoblastoma
Hepatoblastoma recurrent
Hepatocellular carcinoma
Hepatocellular injury
Hepatocellular injury
Hepatocellular injury
Hepatorenal syndrome
Hepatorenal syndrome
Hepatorenal syndrome
Hepatorenicity
Hypercholia
Hypercholia
Hypertibrinolysis
Hypertransaminasaemia
Hypertransaminasaemia
Hyportransaminasaemia
Hypothromboplastinaemia
Hypothromboplastinal
International normalised ratio increased
International normalised ratio increased
International varices
Jaundice hepatoitis
Jaundice hepatoitis
Jaundice hepatoitis
Jaundice hepatoitis
Jaundice hepatoitos

| NN9535<br>NN9535-4506 | Clinical Trial Report | Date: | 04 December 2020 8 | 20 Status:<br>1.0 Page: | Final<br>44 of 229 | Final <b>Novo Nordisk</b><br>rf 229 |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Mitochondrial aspartate aminotransferase increased Mixed hepatocellular cholangiocarcinoma Mixed hiver injury
Model for end stage liver disease score abnormal Model for the stage liver disease score increased Molar ratio of total branched-chain amino acid to Liver opacity
Liver parloads
Liver parloads
Liver scan abnormal
Liver transplant failure
Liver transplant rejection
Liver transplant rejection Liver injury Liver iron concentration abnormal Liver iron concentration increased Periportal oedema
Peritoneal fluid protein abnormal
Peritoneal fluid protein decreased
Peritoneal fluid protein increased
Peritoneovenous shunt
Perencoliia Nodular regenerative hyperplasia Non-alcoholic steatohepatitis Non-cirrhotic portal hypertension Nonalcoholic fatty liver disease Ocular icterus
Oedema due to hepatic disease
Oesophageal varices haemorrhage
Perihepatic discomfort tyrosine Multivisceral transplantation Peripancreatic varices Liver induration measurement Drug related hepatic disorders - comprehensive search (SMQ)

| NN9535<br>NN9535-4506 | Clinical Trial Report | Date:<br>Version: | 04 December 2020 Status:<br>1.0 Page: | 20 Status:<br>0 Page: | Final<br>45 of 229 | Final <b>Novo Nordisk</b><br>f 229 |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Drug related hepatic disorders - comprehensive Portal fibrosis search (SMQ)

Portal hypertension
Portal hypertensive colopathy
Portal hypertensive enteropathy
Portal hypertensive gastropathy
Portal hypertensive gastropathy
Portal hypertensive gastropathy
Portal lyein filammation
Portal vein filatation
Portal vein filatation
Portal vein flow decreased
Portopulmonary hypertension
Protein S abnormal
Protein S abnormal
Prothrombin level abnormal
Prothrombin time abnormal
Prothrombin time prolonged
Prothrombin time abnormal
Prothrombin time abnormal
Prothrombin time ratio increased
Prothrombin time ratio increased
Rediation hepatitis
Regenerative siderotic hepatic nodule
Real and liver transplant
Retinol binding protein decreased
Retrograde portal vein flow
Retye's syndrome
Spienc syndrome
Spienc naevus
Spienc varices haemorrhage
Splenorenal shunt procedure
Spienc varices haemorrhage
Splenorenal shunt
Splenic varices haemorrhage
Splenorenal shunt

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 Page: | 46 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | |
| | | | | | ı |
| Pre-defined MedDRA search | Preferred term | | | | |
| | | | | | I |

Transaminases abnormal

Drug related hepatic disorders - comprehensive search  $(\ensuremath{\mathsf{SMQ}})$ 

Transaminases increased
Ultrasound liver abnormal
Urine bilirubin increased
Urobilinogen urine decreased
Varices oesophageal
V

Intestinal infarction
Mesenteric arterial occlusion
Mesenteric arteriosclerosis
Mesenteric artery embolism
Mesenteric artery thrombosis
Mesenteric artery thrombosis
Mesenteric vascular insufficiency
Mesenteric veacular insufficiency
Mesenteric vein thrombosis
Mesenteric vein thrombosis
Mesenteric vein thrombosis
Mesenteric infarction

Haemorrhoids thrombosed

Ascites

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 47 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | l I |

Thrombosis mesenteric vessel
Truncus coeliacus thrombosis
Vasculitis gastrointestinal
Visceral venous thrombosis
Anorectal varices
Anorectal varices
Anorectal varices
Gastric varices
Gastric varices
Gastric varices haemorrhage
Haemorrhagic ascites
Intestinal varices haemorrhage
Peripanoreatic varices
Intestinal varices
Fortal hypertensive enteropathy
Portal hypertensive enteropathy
Portal hypertensive enteropathy
Varices oesophageal
Varices oesophageal
Varices veins of abdominal wall
White nipple sign
Abdominal disconfort
Abdominal disconfort
Abdominal hernia obstructive
Abdominal hernia obstructive
Abdominal hernia perforation
Abdominal hernia perforation
Abdominal pain lower
Abdominal pain lower
Abdominal rebound tenderness
Abdominal rebound tenderness
Abdominal rebound tenderness
Abdominal repound tenderness
Abdominal repound tenderness
Abdominal symptom
Abdominal tenderness
Abdominal wall disorder
Abdominal wall disorder
Abdominal wall haematoma
Abdominal wall haematoma
Abdominal wall haemorrhage

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 48 of 229 | |
| Pre-defined MedDRA search - list of preferred | : preferred terms | | | | | |

Gastrointestinal adverse events

Pre-defined MedDRA search

Abdominal wall mass
Abdominal wall oedema
Abnormal faeces
Acetonaemic vomiting
Achlorhydria
Acid peptic disease
Acquired enamel hypoplasia
Acquired macroglossia
Acquired macroglossia
Acquired backen
Acute abdomen
Acute backen
Acute oesophageal web
Acute oesophageal web
Acute oesophageal web
Acute pancreatitis
Alcoholic pancreatitis
Alcoholic pancreatitis
Alcoholic pancreatitis
Alcoholic pancreatitis
Alcoholic pancreatitis
Alcoholic pancreopathy
Alveolar bone resorption
Amalgam tattoo

Amoullary polyp
Anaesthesia oral
Anal blister
Anal dilatation
Anal fissure
Anal fissure
Anal fisture
Anal fisture
Anal hypoaesthesia
Anal incontinence
Anal inflammation
Anal leukoplakia
Anal leukoplakia
Anal paraesthesia
Anal paraesthesia

Anal prolapse
Anal prolapse
Anal skin tags
Anal spasm
Anal sphincter atony
Anal sphincter hypertonia
Anal stenosis
Anal trichiasis
Anal ulcer
Anal ulcer
Anal ulcer Anastomotic ulcer perforation polyp prolapse pruritus skin tags

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 49 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Anastomotic ulcer, obstructive
Angina bullosa haemorrhagica
Annyloglossia acquired
Anorectal discomfort
Anorectal discomfort
Anorectal sensory loss
Anorectal stenosis
Anorectal stenosis
Anorectal stenosis
Anorectal stenosis
Anorectal stenosis
Anorectal succent of istula
Anorectal ulcer
Anorectal ulcer
Anorectal stenosis
Anorectal stenosis
Anorectal ulcer
Anorectal stenosis
Appendic colonopathy
Appendic colonopathy
Appendic glossitis
Atrophic glossitis
Autoimmune colitis
Autoimmune pancreatitis
Burcillotemporal syndrome
Autoimmune pancreatitis
Barcett's oesophagus
Barcett's oesophagus
Barcett's oesophagus
Breath odour
Bloody peritoneal effluent
Breath odour
Breath odour
Brunner's gland hyperplasia
Buccal polyp
Buccoglossal syndrome
Cardiospasm
Cascade stomach
Cemento osseous dysplasia
Cascade stomach
Cemento osseous dysplasia

| Novo Nordisk | |
|-------------------------|-----------------------------------------------|
| Final 50 of 229 | |
| Status:<br>Page: | |
| 04 December 2020<br>1.0 | |
| Date: | |
| Clinical Trial Report | f preferred terms |
| NN9535<br>NN9535-4506 | Pre-defined MedDRA search - list of preferred |

Gastrointestinal adverse events

Pre-defined MedDRA search

Chapped lips
Cheilitis
Cheilitis granulomatosa
Cheilitis granulomatosa
Cheilosis
Chilaiditi's syndrome
Chronic cheek biting
Chronic gastrointestinal bleeding
Chronic gastrointestinal bleeding
Chronic gastrointestinal bleeding
Chronic gastrointestinal bleeding
Coating in mouth
Coble stone tongue
Coaliac artery aneurysm
Coeliac artery stenosis
Coeliac artery stenosis
Colitis artery stenosis
Colitis ischaemic
Colitis ischaemic
Colitis ischaemic
Colitis ischaemic
Colitis increative
Colitis increative
Colitis increative
Colitis increative
Colitis increative
Colitis increative
Colonic fistula
Colonic fistula
Colonic fistula
Colonic fistula
Colonic baematoma
Constipation
Constipa

| NN9535 | Clinical Trial Report | Date: 0 | 4 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 51 of 229 | |
| Pre-defined MedDRA search - list of preferred | f preferred terms | | | | | |

Pre-defined MedDRA search

Preferred term

Duodenal pelyp Duodenal stenosis Duodenal ulcer Duodenal ulcer haemorrhage Duodenal ulcer perforation Duodenal ulcer perforation Duodenal ulcer, obstructive Duodenal vascular ectasia Duodenitis haemorrhagic Duodenitis haemorrhagic Duodenogastric reflux Dieulacy's vascular malformation Discoloured vomit Distal intestinal obstruction syndrome Diverticular fistula Diverticular hernia Diverticular perforation Diverticulitis oesophageal Diverticulum
Diverticulum gastric
Diverticulum intestinal
Diverticulum intestinal
Diverticulum cesophageal
Dolichocolon acquired
Douglas' pouch mass Dental pulp disorder
Diabetic enteropathy
Diabetic gastroenteropathy
Diabetic gastroparesis
Diabetic gastropathy
Diaphragmatic hernia
Diaphragmatic hernia
Diaphragmatic hernia, obstructive
Diarrhoea
Diarrhoea heemorrhagic
Diarrhoea neonatal
Diastema Dumping syndrome Duodenal obstruction Duodenal papillitis Duodenal perforation Dry mouth

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | 1000 |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | ) Page: | 52 of 229 | |
| Pre-defined MedDRA search - list of preferred | oreferred terms | | | | | |

Gastrointestinal adverse events

Pre-defined MedDRA search

Dyschezia
Dysphagia
Dysphagia
Dysphagia lusoria
Ectopic gastric mucosa
Ectopic gastric mucosa
Ectopic gastric mucosa
Enamel anomaly
Encapsulating peritoneal sclerosis
Enterit neuropathy
Enterochomafin cell hyperplasia
Enterocolitis haemorrhagic
Enterocolitis haemorrhagic
Enterocolitis paemorrhagic
Enterocolitis
Enterocolit

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final Novo |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 53 of 229 |
| Pre-defined MedDRA search - list of preferred | f preferred terms | | | | |

Gastrointestinal adverse events

Frequent bowements
Functional gastrointestinal disorder
Gastric atony
Gastric cyst
Gastric dilatation
Gastric disorder
Gastric disorder
Gastric distula
Gastric fibrosis
Gastric haemorrhage
Gastric hypertonia
Gastric hypertonia
Gastric hypertonia
Gastric hypertonia
Gastric mucosal earthema
Gastric mucosal calcinosis
Gastric mucosal lesion
Gastric perforation
Gastric perforation
Gastric perforation
Gastric ulcer haemorrhage
Gastric ulcer perforation
Gastric ulcer perforation Flatulence Fluorosis dental Food poisoning Frequent bowel movements

Nordisk

Pre-defined MedDRA search

| N9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 54 of 229 | |
| Pre-defined MedDRA search - list of preferred t | preferred terms | | | | | |

Gastrointestinal adverse events

Pre-defined MedDRA search

Gastroduodenal ulcer
Gastroenteritis eosinophilic
Gastrointestinal amyloidosis
Gastrointestinal angiectasia
Gastrointestinal angiedysplasia
Gastrointestinal disorder
Gastrointestinal disorder
Gastrointestinal fistula
Gastrointestinal haemorrhage
Gastrointestinal hypormotility
Gastrointestinal hypormotility
Gastrointestinal inflammation
Gastrointestinal inflammation
Gastrointestinal ischaemia
Gastrointestinal melanosis

1 mucosa hyperaemia 1 mucosal disorder 1 mucosal exfoliation 1 mucosal necrosis 1 necrosis

Gastrointestinal Gastrointestinal Gastrointestinal

Gastrointestinal

obstruction

oedema

Gastrointestinal Gastrointestinal

pain

Gastrointestinal

motility disorder

mucocoele

Gastrointestinal Gastrointestinal Gastrointestinal Perforation | polyp | polyp haemorrhage | scarring | sounds abnormal

Gastrointestinal Gastrointestinal Gastrointestinal stenosis

Gastrointestinal Gastrointestinal

Gastrointestinal

Gastrointestinal toxicity
Gastrointestinal tract irritation
Gastrointestinal tract mucosal discolouration
Gastrointestinal tract mucosal pigmentation
Gastrointestinal ulcer
Gastrointestinal ulcer perforation
Gastrointestinal vascular malformation
Gastrointestinal vascular malformation
Haemorrhagic
Gastrointestinal wall abnormal
Gastrointestinal wall thickening

| NN9535<br>NN9535-4506 | Clinical Trial Report | Date:<br>Version: | 04 December 2020 Status: | Status:<br>Page: | Final<br>55 of 229 | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | '<br>of preferred terms | | - | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Gastrointestinal wall thinning
Gastrolithiasis
Gastrooesophageal reflux disease
Gastrooesophageal sphincter insufficiency
Gastropleural fistula Gastrosplenic fistula Gastrosplenic fistula Giant cell epulis Gingival atrophy Gingival bleeding Gingival blister Gingival discolouration Gingival disconfert Gingival discomfert Gingival erosion Gingival hypertiquentation Gingival hypertiophy Gingival hypertrophy Gingival pain Gingival pain Gingival pain Gingival pain Gingival pain Gingival pain Gingival recession Gingival ulceration Gingival ulceration Gingivitis ulcerative Glossitis Glossodynia Gastroptosis

Hernial eventration
Heyde's syndrome
Hiatus hernia strangulated
Hiatus hernia strangulated
Hiatus hernia, obstructive Haemorrhoids

Haemoperitoneum Haemorrhagic erosive gastritis Haemorrhagic necrotic pancreatitis Haemorrhoidal haemorrhage

Glossoptosis Glycogenic acanthosis Gut fermentation syndrome

Haematochezia

Haematemesis

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 56 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Dre-defined MedDRA search | Draferrad torm | | | | | ı |

Hyperaesthesia teeth
Hypercomentosis
Hypercomnoris
Hypercomnoris
Hypercomploy anal papilla
Hypercostrinaemia
Hypercostrinaemia
Hypercostrinaemia
Hypoaesthesia oral
Hypoaesthesia oral
Hypoaesthesia teeth
Ileal perforation
Ileal stenosis
Ileal ulcer perforation
Ileal ulcer perforation
Ileas sparalytic
Ileus paralytic
Ileus spatic
Ileus spa

| Final Novo Nordisk | f 229 | |
|---|---|---|
| H | 57 of 229 | |
| Status: | Page: | |
| 04 December 2020 | 1.0 | |
| Clinical Trial Report | | of preferred terms |
| NN9535 | NN9535-4506 | Pre-defined MedDRA search - list of preferred |

Gastrointestinal adverse events

Pre-defined MedDRA search

Intestinal haemorrhage
Intestinal mass
Intestinal mass
Intestinal macosal intestinal mucosal atrophy
Intestinal mucosal tear
Intestinal mucosal tear
Intestinal polyporestinal perforation
Intestinal prolyporestinal statosis
Intestinal statosis
Intestinal stanosis
Intestinal alocer perforation
Intestinal ulcer perforation
Intestinal ulcer perforation
Intestinal ulcer perforation
Intestinal ulcer perforation
Intestinal ulcer perforation
Intra-abdominal haematoma
Ischaemic centeritis
Ischaemic pancreatitis
Ischaemic pancreaticis
Intestinal ulcer perforation
Israe intestinal ulcer perforation
Israe intestinal ulcer perforation
Israe int

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 58 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | : preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ı |

Lip blister
Lip discolouration
Lip discolouration
Lip dry
Lip erosion
Lip erosion
Lip extfoliation
Lip extfoliation
Lip haemorrhage
Lip pain
Lip pain
Lip pruritus
Lip pruritus
Lip pruritus
Lip pruritus
Lip pruritus
Lip pruritus
Lip prostrointestinal haemorrhage
Lower gastrointestinal perforation
Lower gastrointestinal perforation
Lower gastrointestinal perforation
Lumbar hernia
Lupus pencreatitis
Lupus pencreatitis
Lupus pencreatitis
Lupus percreatitis
Lupus pencreatitis
Lupus pencre Leukoplakia oesophageal Leukoplakia oral Levator syndrome Lichenoid dysplasia Meconium cyst Meconium ileus

Meconium peritonitis
Meconium plug syndrome
Megacolon
Melaena
Melaena neonatal
Melanoplakia oral

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 59 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Mesenteric artery aneurysm
Mesenteric cyst
Mesenteric fibrosis
Mesenteric panniculitis
Mesenteric panniculitis
Mesenteric panniculitis
Mesenteric panniculitis
Mesenteric panniculitis
Mesenteritic
Mesenteritis
Mikulicz's disease
Mikulicz's disease
Mikulicz's syndrome
Mucosal prolapse syndrome
Mucosal prolapse syndrome
Mucosal prolapse syndrome
Necrotising colitis
Necrotising dastritis
Necrotising dastritis
Necrotising dastritis
Necrotising dastritis
Necrotising dastritis
Neonatal dastrointestinal haemorrhage
Neonatal intestinal dilatation
Neonatal intestinal obstruction
Neonatal intestinal dilatation
Neuropenic colitis
Neonatal intestinal dilatation
Neutropenic colitis
Noninfective gingivitis
Noninfective gastric
Obstructive defacecation
Obstructive defacecation
Obstructive pencreatitis
Occophageal achalasia
Occophageal achalasia
Occophageal compression
Occophageal dilatation

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 60 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ı |
| | | | | | | I |

Oesophageal discomfort
Oesophageal disorder
Oesophageal fibrosis
Oesophageal fibrosis
Oesophageal fibrosis
Oesophageal haemorthage
Oesophageal intramural haematoma
Oesophageal intriation
Oesophageal mucosal bister
Oesophageal mucosal bister
Oesophageal mucosal bister
Oesophageal stone
Oesophageal mucosal bister
Oesophageal stone
Oesophageal bolto
Oesophageal obstruction
Oesophageal stensis
Oesophageal stensis
Oesophageal ulcer haemorrhage
Oesophageal ulcer perforation
Oesophageal ulcer beforation
Oesophageal ulcer perforation
Oesophageal ulcer perforation
Oesophagitis
Oesophagitis ulcerative
Oesophagitis ulcerative
Oesophagitis fiatula
Omental infarction
Omental infarction
Omental infarction
Omental infarction
Omental discondert
Oral discondert
Oral discondert
Oral discondert
Oral discondert
Oral discondert
Oral discondert

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | 1.0 Page: | 61 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I I |

Oral hyperaesthesia
Oral lichen planus
Oral lichen planus
Oral lichen planus
Oral lichenoid reaction
Oral mucosa atrophy
Oral mucosa lescolouration
Oral mucosal blistering
Oral mucosal blistering
Oral mucosal erythema
Oral mucosal erythema
Oral mucosal erythema
Oral mucosal erythema
Oral mucosal scab
Oral mucosal scab
Oral papule
Oral papul

| NN9535 | Clinical Trial Report | Date: 04 | December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 62 of 229 | |
| Pre-defined MedDRA search - list of prefe | : preferred terms | | | | | |

Pre-defined MedDRA search

Preferred term

Pancreatic mass
Pancreatic necrosis
Pancreatic phegomon
Pancreatic pseudocyst
Pancreatic pseudocyst haemorrhage
Pancreatic pseudocyst haemorrhage
Pancreatic pseudocyst rupture
Pancreatitis pseudocyst rupture
Pancreatitis catoosis
Pancreatitis acute
Pancreatitis acute
Pancreatitis necrotising
Pancreatitis relapsing
Pancreatitis relapsing
Pancreatitis necrotising
Pancreatitis necrotising
Pancreatitis necrotising
Pancreatitis necrotising
Pancreatitis chonic
Pancreatitis relapsing
Pancreatitis necrotising
Pancreatitis necrotising
Pancreatitis necrotising
Pancreatitis necrotising
Pancreatitis necrotising
Pancreatitis necrotising
Parcreatitis necrotising
Parcreatitis necrotising
Parcreatitis necrotising
Parcreatitis necrotising
Parcreatitis of Vater stenosis
Parcrid gland enlargement
Parcrid gland haemorrhage
Pertic ulcer perforation
Peptic ulcer perforation
Peptic

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 63 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | : preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Peritoneal necrosis
Peritoneal perforation
Peritonecutaneous fistula
Peritonicus lupus
Peritonis lupus
Pharyngo-oesophageal diverticulum
Pigmentation lip
Plicated tongue
Pneumatosis intestinalis
Pneumatosis intestinalis
Pneumoperitoneum
Poor dental condition
Portal venous gas
Post-tussive vomiting
Prochitis
Precoparalysis
Proctalysis
Proctitis haemorrhagic
Proctitis haemorrhagic
Proctitis ulcerative
Proctitis ulcerative
Proctitis standing
Proctitis baemorrhagic
Proctitis standing
Proctitis standing
Proctitis baemorrhagic
Procticis ulcerative
Proctitis standing
Proctitis ulcerative
Proctitis standing
Proctitis ulcerative
Proctitis ulcerative
Proctitis standing
Proctitis ulcerative
Proctitis standing
Proctitis ulcerative
Proctitis standing
Procticis sphincter insufficiency
Pylorospasm
Pylorospasm
Pylorospasm
Pylorospasm
Pylorospasm
Pylorospasm
Pylorospasm
Pylorospasm
Pylorospasm
Rectal discharge
Rectal discharge
Rectal discharge
Rectal lesion
Rectal polyp

| NN9535<br>NN9535-4506 | Clinical Trial Report | Date: | 04 December 2020 5 | Status:<br>Page: | Final<br>64 of 229 | Final <b>Novo Nordisk</b><br>f 229 |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ı |

Rectal prolapse
Rectal stenosis
Rectal ulcer
Rectal ulcer haemorrhage
Rectal ulcer haemorrhage
Rectourethral fistula
Retioux gastritis
Reducgitation
Retroperitoneal leffusion
Retroperitoneal haematoma
Retroperitoneal haematoma
Retroperitoneal haematoma
Retroperitoneal haematoma
Retroperitoneal laematoma
Salivary duct inflammation
Salivary gland atrophy
Salivary gland eleculus
Salivary gland eleculus
Salivary gland miss

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 65 of 229 | |
| Pre-defined MedDRA search - list of preferred | preferred terms | | | | | |

Gastrointestinal adverse events

Pre-defined MedDRA search

Sialectasia
Sialocele
Sialocochitis fibrinosa
Sialocochitis fibrinosa
Sialometaplasia
Sideropenic dysphagia
Sideropenic dysphagia
Sideropenic dysphagia
Sideropenic dysphagia
Sideropenic dysphagia
Sideropenic dysphagia
Sideropenic dysphagia
Small intestinal berforation
Small intestinal ulcer perforation
Sprinc artery aneurysm
Splenic vein aneurysm
Splenic vein aneurysm
Splenic vein desenterios
Stomach mass
Stomach mass
Stomach is becontatis necrotising
Strawberry tongue

| NN9535 | Clinical Trial Report | Date: 0 | 4 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 66 of 229 | |
| Pre-defined MedDRA search - list of preferred | f preferred terms | | | | | |

Pre-defined MedDRA search

Gastrointestinal adverse events

Tongue pigmentation
Tongue prunitus
Tongue polyp
Tongue vough
Tongue spasm
Tongue ulceration
Tongue ulceration
Tooth ankylosis
Tooth demineralisation
Tooth development disorder
Tooth discolouration
Tooth discolouration
Tooth discolouration
Tooth pulp haemorrhage
Tooth pulp haemorrhage
Tooth socket haemorrhage
Tooth socket haemorrhage
Tooth coclusion
Tooth socket in testine
Tooth socket in testine
Tooth socket in testine
Tooth socket haemorrhage
Tooth socket haemorrhage
Tooth socket haemorrhage
Tooth socket haemorrhage
Tooth socket in testine
Transient lingual papillitis
Tranmatic occlusion
Tranmatic ulcerative granuloma with stromal essinophilia
Trichoglossia
Ulcerative duodenitis
Ulcerative gastritis Tongue ex.
Tongue ex.
Tongue peograp.
Tongue haematoma
Tongue haemorrhage
Tongue infarction
Tongue inforction
Tongue necvenent disturbance
Tongue peograpiantation

oblyp discomfort disorder Tongue discomfort
Tongue disorder
Tongue dry
Tongue dryplasia
Tongue eruption
Tongue eruptiom dysplasia

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 67 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Ultrafiltration failure
Umbilical hernia perforation
Umbilical hernia, obstructive
Upper gastrointestinal hemorrhage
Upper gastrointestinal perforation
Uraemic gastropathy
Urinary ascites
Uvulitis
Varicose veins sublingual

Gastrointestinal adverse events

Injection site reactions

Volunting of small bowel Vomiting projectile Wischnewsky spots

Visceroptosis Volvulus Administration site dermatitis
Administration site eczema
Administration site hypersensitivity
Administration site recall reaction
Administration site urticaria
Administration site urticaria
Application site dermatitis
Application site dermatitis
Application site tash
Application site recall reaction
Application site rash
Application site recall reaction
Application site recall reaction
Application site recall reaction
Application site recall reaction
Infusion site eczema
Infusion site eczema
Infusion site eczema
Infusion site rash
Infusion site recall reaction
Infusion site recall reaction
Infusion site recall reaction
Infusion site urticaria
Infusion site recall reaction
Infusion site urticaria
Infusion site recall reaction
Infusion site dermatitis
Injection site dermatitis
Injection site recall reaction
Injection site recall reaction
Injection site recall reaction
Injection site recall reaction

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 68 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Injection site urticaria
Injection site urscaria
Injection site vasculitis
Instillation site rash
Instillation site urticaria
Vessel puncture site rash
Vessel puncture site vesicles
Administration site thrombosis
Injection site thrombosis
Embolia cutis medicamentosa
Infusion site thrombosis
Injection site thrombosis
Injection site thrombosis
Instillation site thrombosis
Instillation site thrombosis
Vessel puncture site occlusion
Vessel puncture site occlusion
Vessel puncture site coclusion
Vessel puncture site occlusion
Administration site anaesthesia
Administration site atrophy
Administration site calcification
Administration site calcification
Administration site calcification
Administration site calcification
Administration site discolouration
Administration site discolouration
Administration site discolouration
Administration site discolouration
Administration site extravasation
Administration site extravasation
Administration site fibrosis
Administration site fibrosis
Administration site hyperaesthesia
Administration site hypertrichosis
Administration site hypertrichosis
Administration site hypertrichosis
Administration site hypertrichosis
Administration site hypertrichosis
Administration site hypertrichon

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 Page: | age: | 69 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Injection site reactions
Administration site in Administration site in Administration site in Administration site in

Administration site induration
Administration site infection
Administration site inflammation
Administration site inflammation
Administration site ischaemia
Administration site joint effusion
Administration site joint effusion
Administration site joint fifammation
Administration site joint inflammation
Administration site joint inflammation
Administration site joint warmth
Administration site joint warmth
Administration site joint warmth
Administration site joint warmth
Administration site point warmth
Administration site macule
Administration site macule
Administration site movement impairment
Administration site movement impairment
Administration site pailor
Administration site scab
Administration site scab
Administration site scab
Administration site scab
Administration site scab
Administration site scab
Administration site scap
Administration site scap
Administration site wealting
Administration site wealting
Administration site warmth
Administration site warmth
Administration site warmth
Administration site warmth
Administration site warmth

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 70 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Application site abscess sterile
Application site acne
Application site acne
Application site alopecia
Application site arrophy
Application site burins
Application site calcification
Application site calcification
Application site collulitis
Application site collulitis
Application site discondration
Application site discondration
Application site fibrosis
Application site extravasation
Application site fibrosis
Application site fibrosis
Application site fibrosis
Application site haematoma
Application site haematoma
Application site haematon
Application site hyperaesthesia
Application site hypertrophy
Application site hypertrophy
Application site inflammation
Application site inflammation
Application site inflammation
Application site inflammation
Application site infection
Application site inflammation
Application site joint effusion
Application site joint erythema
Application site joint erythema
Application site joint inflammation

| Novo Nordisk | | 1 |
|---|---|---|
| Final | 71 of 229 | |
| Status: | Page: | |
| 04 December 2020 | 1.0 | |
| Clinical Trial Report | 1 | f preferred terms |
| | | h - list o |
| NN9535 | NN9535-4506 | Pre-defined MedDRA search - list of preferred terms |

Injection site reactions

Pre-defined MedDRA search

Application site joint pain Application site joint swelling Application site joint warmth Application site joint warmth Application site laceration Application site macule Application site macule Application site mass Application site mass Application site nerve damage Application site nodule Application site parant odule Application site odour Application site paulor Application site pruritus Application site pruritus Application site pruritus Application site prusura Application site pusules Application site scab Application site swelling Application site telangiectasia Application site telangiectasia Application site warmth Application site abscess sterile Infusion site abscess sterile Infusion site anaesthesia Infusion site anaesthesia Infusion site callification Infusion site callification Infusion site callification Infusion site callification Infusion site cellulitis Infusion site cellulitis

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 72 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ı |

Infusion site cyst
Infusion site discharge
Infusion site discolouration
Infusion site disconfort
Infusion site discomfort
Infusion site dysaesthesia
Infusion site erosion
Infusion site erosion
Infusion site extravasation
Infusion site extravasation
Infusion site haematoma
Infusion site haematoma
Infusion site haematoma
Infusion site hypertrichosis
Infusion site hypertrichosis
Infusion site hypertrichosis
Infusion site inflammation
Infusion site inflammation
Infusion site inflammation
Infusion site inflammation
Infusion site inflammation
Infusion site joint discomfort
Infusion site joint effusion
Infusion site joint inflammation
Infusion site joint inflammation
Infusion site joint inflammation
Infusion site joint movement impairment
Infusion site joint movement infusion site joint swalling
Infusion site joint pain
Infusion site joint swalling
Infusion site inflammation
Infusion site joint swalling
Infusion site laceration
Infusion site macule
Infusion site mecule
Infusion site mecule
Infusion site mecule
Infusion site nerve damage
Infusion site nerve damage
Infusion site nerve damage
Infusion site nerve damage
Infusion site nerve damage
Infusion site oedema

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 73 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | E preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Infusion site pain
Infusion site pallor
Infusion site pallor
Infusion site photosensitivity reaction
Infusion site photosensitivity reaction
Infusion site plaque
Infusion site pustule
Infusion site pustule
Infusion site scab
Infusion site scab
Infusion site scab
Infusion site swelling
Infusion site swelling
Infusion site scar
Infusion site scab
Infusion site and star a
Infusion site and star a
Infusion site and star a
Infusion site alopecia
Injection site alopecia
Injection site calcification
Injection site calcification
Injection site calcification
Injection site deformation
Injection site deformation
Injection site deformation
Injection site discolouration
Injection site extravasation
Injection site extravasation
Injection site parametoma
Injection site haemacoma

| NN9535<br>NN9535-4506 | Clinical Trial Report | Date:<br>Version: | 04 December 2020 Status: | Status:<br>Page: | Final<br>74 of 229 | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | ist of preferred terms | _ | | ) | - | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Injection site hypertrichosis
Injection site hypertrophy
Injection site hypertrophy
Injection site indentation
Injection site indentation
Injection site inflammation
Injection site inflammation
Injection site inflammation
Injection site inflammation
Injection site joint effusion
Injection site joint effusion
Injection site joint effusion
Injection site joint inflammation
Injection site joint movement impairment
Injection site joint warmth
Injection site joint warmth
Injection site joint warmth
Injection site joint warmth
Injection site joint warmth
Injection site joint warmth
Injection site point warmth
Injection site point warmth
Injection site pallor
Injection site pallor
Injection site pallor
Injection site pallor
Injection site pallor
Injection site pallor
Injection site palnor
Injection site palnor
Injection site pallor
Injection site palnor
Injection site palnor
Injection site palnor
Injection site paraesthesia
Injection site phrebitis
Injection site publicis
Injection site public
Injection

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | 1.0 Page: | 75 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | l I |

Injection site telangiectasia
Injection site ulcer
Injection site ulcer
Injection site warmth
Instillation site abscess
Instillation site arrophy
Instillation site atrophy
Instillation site burn
Instillation site complication
Instillation site complication
Instillation site discomfort
Instillation site discomfort
Instillation site discomfort
Instillation site discomfort
Instillation site discomfort
Instillation site exfoliation
Instillation site exfoliation
Instillation site infection
Instillation site infection
Instillation site infection
Instillation site infection
Instillation site inflammation
Instillation site inflammation
Instillation site inflammation
Instillation site inflammation
Instillation site inflammation
Instillation site papules
Instillation site papules
Instillation site papules
Instillation site papules
Instillation site paraesthesia
Instillation site paraesthesia
Instillation site paraesthesia
Instillation site purritus
Instillation site purritus
Instillation site scab
Instillation site swelling
Instillation site swelling
Instillation site warmth
| NN9535<br>NN9535-4506 | Clinical Trial Report | Date:<br>Version: | 04 December 2020 Status: 1.0 Page: | Final 76 of 229 | Final <b>Novo Nordisk</b> f 229 |
|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | |

Injection site reactions

Malabsorption from administration site
Malabsorption from application site
Oral administration complication site
Oral administration complication
Puncture site abscess
Puncture site discharge
Puncture site discharge
Puncture site haematoma
Puncture site haematoma
Puncture site haemacrian
Puncture site harnia
Puncture site infection
Puncture site infection
Puncture site infection
Puncture site infection
Puncture site infection
Puncture site eodema
Puncture site swalling
Puncture site pain
Puncture site pain
Puncture site pain
Puncture site swalling
Systemic leakage
Vessel puncture site anaesthesia puncture site erythema 1 puncture site haematoma 1. puncture site haemorrhage 2. puncture site hypoaesthesia 2. puncture site infaration 3. puncture site inflammation puncture site injury
puncture site pain
puncture site paraesthesia
puncture site paraesthesia
puncture site phlebitis puncture site bruise puncture site cellulitis puncture site discharge reaction swelling puncture site puncture site Vessel | Ves Vessel Vessel Vessel Vessel

Malignant tumours (SMQ)

Cholangiosarcoma Hepatic angiosarcoma Hepatic cancer

Final Novo Nordisk 77 of 229 04 December 2020 | Status: 1.0 Page: Version: Date: Clinical Trial Report Pre-defined MedDRA search - list of preferred terms NN9535-4506 NN9535

Pre-defined MedDRA search

Preferred term

Malignant tumours (SMQ)

Hepatocellular carcinoma Mixed hepatocellular cholangiocarcinoma Hepatobiliary cancer Hepatobiliary cancer in situ Hepatic cancer metastatic
Hepatic cancer recurrent
Hepatic cancer stage I
Hepatic cancer stage III
Hepatic cancer stage III Hepatoblastoma Hepatoblastoma recurrent Hepatic cancer stage IV

5q minus syndrome Abdominal wall neoplasm malignant Acinar cell carcinoma of pancreas Acinic cell carcinoma of salivary gland

Acral lentiginous melanoma Acral lentiginous melanoma stage I Acral lentiginous melanoma stage II Acral lentiginous melanoma stage III Acral lentiginous melanoma stage IVI Acute bilineal leukaemia Acute biphenotypic leukaemia Acute erythroid leukaemia Acute leukaemia

Acute megakaryocytic leukaemia (in remission) Acute leukaemia in remission Acute lymphocytic leukaemia Acute lymphocytic leukaemia in remission) Acute lymphocytic leukaemia recurrent Acute lymphocytic leukaemia refractory Acute megakaryocytic leukaemia

Acute monocytic leukaemia
Acute monocytic leukaemia
Acute monocytic leukaemia
Acute myeloid leukaemia (in remission)
Acute myeloid leukaemia recurrent
Acute myeloid leukaemia recurrent
Acute myeloid leukaemia refractory
Acute myeloid leukaemia refractory
Acute promyelocytic leukaemia
Acute undifferentiated leukaemia
Adenocarcinoma

Adenocarcinoma gastric

| NN9535 | Clinical Trial Report | Date: 04 | December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 78 of 229 | |
| Pre-defined MedDRA search - list of preferre | f preferred terms | | | | | |

pre

Pre-defined MedDRA search

Malignant tumours (SMQ)

Preferred term

Adenoid cystic carcinoma of the cervix
Adenoid cystic carcinoma of the cervix
Adenosquamous carcinoma of the cervix
Adenosquamous carcinoma of vagina
Adenosquamous cell carcinoma
Adenosquamous cell lung cancer recurrent
Adenosquamous cell lung cancer stage 0
Adenosquamous cell lung cancer stage II
Adrenal gland cancer metastatic
Adrenocortical carcinoma
Adult T-cell lymphoma/leukaemia refractory
Adult T-cell lymphoma/leukaemia stage II
Adult T-cell lymphoma/leukaemia stage II
Adult T-cell lymphoma/leukaemia stage II
Adult T-cell lymphoma/leukaemia stage II
Adult T-cell lymphoma/leukaemia stage II Alveolar soft part sarcoma Alveolar soft part sarcoma metastatic Alveolar soft part sarcoma recurrent Ameloblastic carcinoma Adenocarcinoma metastatic
Adenocarcinoma of appendix
Adenocarcinoma of colon
Adenocarcinoma of salivary gland
Adenocarcinoma of the cervix Alveolar rhabdomyosarcoma Anal cancer metastatic
Anal cancer recurrent
Anal cancer stage I
Anal cancer stage II
Anal cancer stage III
Anal cancer stage III
Anal cancer stage III Aesthesioneuroblastoma Aleukaemic leukaemia cancer Anal

04 December 2020 | Status: Version: Date: Clinical Trial Report NN9535-4506

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Malignant tumours (SMQ)

types refractory
Anaplastic large cell lymphoma T and null-cell
types stage I
Anaplastic large cell lymphoma T and null-cell
types stage II
Anaplastic large cell lymphoma T and null-cell
types stage II
Anaplastic large cell lymphoma T and null-cell
types stage II
Anaplastic large-cell lymphoma T and null-cell
types stage IV
Anaplastic large-cell lymphoma
Anaplastic charge-cell lymphoma
Anaplastic chycoid cancer
Andiocentric lymphoma recurrent
Andiocentric lymphoma stage II
Andiocentric lymphoma stage II
Andiocentric lymphoma stage II
Andioimmunoblastic T-cell lymphoma stage II
Andioimmunoblastic T-cell lymphoma stage II Anal squamous cell carcinoma Anaplastic astrocytoma Anaplastic large cell lymphoma T- and null-cell types recurrent Anaplastic large cell lymphoma T- and null-cell Anaplastic large cell lymphoma T- and null-cell Angiosarcoma non-metastatic Angiosarcoma recurrent Apocrine breast carcinoma Appendix cancer Astrocytoma Angiosarcoma metastatic Astrocytoma malignant Angiosarcoma

Final Novo Nordisk


Preferred term

NN9535

Final Novo Nordisk 80 of 229 04 December 2020 Status: 1.0 Page: Version: Date: Preferred term | Clinical Trial Report Pre-defined MedDRA search - list of preferred terms Pre-defined MedDRA search NN9535-4506 NN9535

Malignant tumours (SMQ)

Atypical teratoid/rhabdoid tumour of CNS
B precursor type acute leukaemia
B-cell lymphoma recurrent
B-cell lymphoma refractory
B-cell lymphoma stage II
B-cell lymphoma stage II
B-cell lymphoma stage II
B-cell lymphoma stage II
B-cell lymphoma stage II
B-cell lymphoma stage II
B-cell lymphoma stage II
B-cell small lymphocytic lymphoma refractory
B-cell small lymphocytic lymphoma stage II
B-cell duct action a metastatic
Basal cell carcinoma
Basso cute leukaemia
Basal cell carcinoma
Basso cute action a metastatic
Basosquamous carcinoma of skin
Bile duct adenocarcinoma carcinoma
Bile duct cancer stage II
Bile duct cancer stage III
Bile duct cancer stage III
Bile duct cancer stage III
Bile duct cancer stage III
Bile duct cancer stage III
Bilader adenocarcinoma stage III
Bladder adenocarcinoma stage III

81 of 229 04 December 2020 | Status: 1.0 | Page: Version: Date: | Clinical Trial Report NN9535-4506 NN9535

Pre-defined MedDRA search - list of preferred terms Pre-defined MedDRA search

Preferred term

Bladder cancer recurrent
Bladder cancer stage 0, with cancer in situ
Bladder cancer stage 1, with cancer in situ
Bladder cancer stage 1, with cancer in situ
Bladder cancer stage 1, without cancer in situ
Bladder cancer stage II
Bladder cancer stage II
Bladder cancer stage IV
Bladder squamous cell carcinoma recurrent
Bladder squamous cell carcinoma stage I
Bladder squamous cell carcinoma stage II
Bladder squamous cell carcinoma stage II
Bladder squamous cell carcinoma stage II
Bladder squamous cell carcinoma stage II
Bladder squamous cell carcinoma stage II
Bladder squamous cell carcinoma stage II
Bladder squamous cell carcinoma stage II
Bladder transitional cell carcinoma metastatic
Bladder transitional cell carcinoma stage II
Bladder transitional cell carcinoma stage II
Bladder transitional cell carcinoma stage II
Bladder transitional cell carcinoma stage II
Bladder transitional cell carcinoma stage II
Bladder transitional cell carcinoma stage II
Bladder transitional cell carcinoma stage II
Bladder transitional cell carcinoma stage III
Bladder transitional cell carcinoma stage III Blast crisis in myelogenous leukaemia Blastic plasmacytoid dendritic cell neoplasia Bone cancer Bone giant cell tumour malignant Bone marrow leukaemic cell infiltration Bone marrow tumour cell infiltration Breast angiosarcoma Breast angiosarcoma metastatic Breast cancer Breast cancer female Breast cancer in situ Bone sarcoma Bowen's disease Brain cancer metastatic Brain neoplasm malignant Bone cancer metastatic Blast cell crisis Brain stem glioma Brain sarcoma

Final Novo Nordisk

Malignant tumours (SMQ)

| NN9535<br>NN9535-4506 | Clinical Trial Report | Date:<br>Version: | 04 December 2020 Status:<br>1.0 Page: | Final $ 82 \text{ of } 229 $ | Novo Nordisk |
|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred | f preferred terms | | | | |

Pre-defined MedDRA search

Malignant tumours (SMQ)

Preferred term

Breast sarcoma metastatic

Carcinoid tumour of the appendix
Carcinoid tumour of the caecum
Carcinoid tumour of the caecum
Carcinoid tumour of the gastrointestinal tract
Carcinoid tumour of the partial tract
Carcinoid tumour of the parcial
Carcinoid tumour of the parcial
Carcinoid tumour of the prostate
Carcinoid tumour of the prostate
Carcinoid tumour of the stomach
Carcinoid tumour of the stomach
Carcinoid tumour of the stomach
Carcinoid tumour of the stomach
Carcinoid tumour of the stomach
Carcinoid tumour of the stomach
Carcinoma in situ of eye
Carcinoma in situ of eye
Carcinoma in situ of skin
Carcinoma in situ of skin
Carcinoma in situ of skin
Carcinoma in situ of trachea

Breast cancer male
Breast cancer metastatic
Breast cancer recurrent
Breast cancer stage I
Breast cancer stage II
Breast cancer stage III
Breast cancer stage III
Breast implant-associated anaplastic large cell
Iymphoma
Breast sarcoma

Breast sarcoma recurrent
Bronchial carcinoma
Bronchioloalveolar carcinoma
Burkitt's leukaemia
Burkitt's lymphoma recurrent
Burkitt's lymphoma refractory
Burkitt's lymphoma stage II
Burkitt's lymphoma stage II
CNS germinoma

| NN9535<br>NN9535-4506 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final 83 of 229 | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | . of preferred terms | | | , Sp. 1 | 11 10 00 | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Cardiac neoplasm malignant
Central nervous system leukaemia
Central nervous system leukaemia
Central nervous system melanoma
Central nervous system melanoma
Cervix carcinoma stage IC
Cervix carcinoma stage II
Cervix carcinoma stage II
Cervix carcinoma stage II
Cervix carcinoma stage II
Cervix carcinoma stage II
Cervix carcinoma stage II
Cervix carcinoma stage IV
Chloroma
(in remission)
Choroma
(in remission)
Choroma
(in remission)
Choroma
Choroma metastatic
Chondrosarcoma metastatic
Chondrosarcoma metastatic
Choroma in remission)
Choroma in remission
Choroid melanoma
Choroid melanoma
Choroid melanoma
Choroid melanoma
Choroid plexus carcinoma
Choroid plexus carcinoma
Choroid leukaemia in remission)
Chronic leukaemia in remission)
Chronic lumphocytic leukaemia stage 1
Chronic lymphocytic leukaemia stage 2
Chronic lymphocytic leukaemia stage 3
Chronic myeloid leukaemia transformation Chronic myeloid leukaemia transformation Chronic myeloid leukaemia transformation Chronic myeloid leukaemia transformation Chronic myeloid leukaemia transformation Chronic myeloid leukaemia chronic myeloid leukaemia chronic myeloid leukaemia transformation Chronic myeloid leukaemia chronic myeloid leukaemia chronic

| NN9535<br>NN9535-4506 | Clinical Trial Report | Date:<br>Version: | 04 December 2020 Status: | Status:<br>Page: | Final<br>84 of 229 | Final <b>Novo Nordisk</b> of 229 |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | ist of preferred terms | | _ | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Ciliary body melanoma of cervix
Clear cell carcinoma of cervix
Clear cell endometrial carcinoma
Clear cell sarcoma of the kidney
Clear cell sarcoma of the kidney
Colon cancer metastatic
Colon cancer rage II
Colon cancer stage II
Colon cancer stage II
Colon cancer stage III
Colon cancer stage III
Colon cancer stage III
Colon cancer stage III
Colon cancer stage III
Colon cancer stage III
Colorectal adenocarcinoma
Colorectal cancer metastatic
Colorectal cancer stage II
Colorectal lymphoma stage II
Cutaneous T-cell lymphoma stage II
Cutaneous T-cell lymphoma stage IV
Cystadenocarcinoma pancreas
Dedifferentiated liposarcoma
Dermatofibrosarcoma protuberans
Dermatofibrosarcoma protuberans
Dermatofibrosarcoma protuberans
Dermatofibrosarcoma protuberans
Dermatofibrosarcoma protuberans metastatic
Desmoplastic mesothelioma

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final Novo | Novo |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | 1.0 Page: | 85 of 229 | |
| Pre-defined MedDRA search - list of preferred | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Malignant tumours (SMQ)

Desmoplastic small round cell tumour
Diffuse large B-cell lymphoma recurrent
Diffuse large B-cell lymphoma refractory
Diffuse large B-cell lymphoma stage II
Diffuse large B-cell lymphoma stage II
Diffuse large B-cell lymphoma stage II
Diffuse large B-cell lymphoma stage II
Diffuse large B-cell lymphoma stage III
Diffuse large B-cell lymphoma stage IV
Dissented large cell lymphoma
Double hit lymphoma
Double hit lymphoma
Ductal adenocarcinoma of pancreas Ependymoma malignant
Epididymal cancer
Epididymal cancer
Epithelioid mesothelioma
Epithelioid sarcoma metastatic
Epithelioid sarcoma recurrent
Epstein-Barr virus associated lymphoma
Erythraemic myelosis (in remission)
Ewing's sarcoma metastatic
Ewing's sarcoma metastatic Enteropathy-associated T-cell lymphoma Embryonal rhabdomyosarcoma Endocrine neoplasm malignant Endometrial adenocarcinoma Endometrial cancer Endometrial cancer metastatic Endometrial cancer recurrent Endometrial cancer stage I Endometrial cancer stage II Endometrial cancer stage II Endometrial cancer stage II Endometrial cancer stage II Endometrial cancer stage II Endometrial cancer stage IV Endometrial sarcoma metastatic Endometrial sarcoma recurrent Endometrial stromal sarcoma Endotheliomatosis Ear neoplasm malignant Eosinophilic leukaemia Eccrine carcinoma

o Nordisk

1.0 Page: Version: Date: Clinical Trial Report NN9535-4506 NN9535

04 December 2020 | Status:

Final Novo Nordisk 86 of 229

Pre-defined MedDRA search - list of preferred terms

Malignant tumours (SMQ)

Pre-defined MedDRA search

Ewing-like sarcoma
External ear neoplasm malignant
Extra-osseous Ewing's sarcoma metastatic
Extra-osseous Ewing's sarcoma recurrent

Preferred term

Extragonadal primary embryonal carcinoma Extragonadal primary germ cell tumour Extragonadal primary germ cell tumour mixed Extragonadal primary germ cell tumour mixed

Extragonadal primary germ cell tumour mixed stage

Extragonadal primary germ cell tumour mixed stage

malignant teratoma Extragonadal Extragonadal

non-seminoma primary n primary r primary r

Extragonadal primary non-seminoma stage I Extragonadal primary non-seminoma stage II Extragonadal primary non-seminoma stage II Extragonadal primary non-seminoma stage III Extragonadal primary seminoma (pure) Extragonadal primary seminoma (pure) stage I Extragonadal primary seminoma (pure) stage II Extragonadal primary seminoma (pure) stage II Extragonadal primary seminoma (pure) stage II Extramandal primary seminoma (pure) stage II Extramandal primary seminoma (pure) stage IV Extramammary Paget's disease

type) Extranodal marginal zone B-cell lymphoma (MALT type)

(MALT (MALT (MALT (MALT

Extranodal marginal zone B-cell lymphoma

Extranodal marginal zone B-cell lymphoma type) refractory Extranodal marginal zone B-cell lymphoma type) recurrent

type) stage II Extranodal marginal zone B-cell lymphoma (MALT type) stage I Extranodal marginal zone B-cell lymphoma

type) stage III Extranodal marginal zone B-cell lymphoma (MALT type) stage IV Extracoular retinoblastoma

04 December 2020 | Status: Version: Date: Clinical Trial Report NN9535-4506 NN9535

Preferred term

Final Novo Nordisk


Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Malignant tumours (SMQ)

Fallopian tube cancer metastatic Fallopian tube cancer stage I Fallopian tube cancer stage II Fallopian tube cancer stage II Fallopian tube cancer stage III Fallopian tube cancer stage IV Fallopian tube cancer stage IV Familial medullary thyroid cancer Female reproductive tract carcinoma in situ Fibrosarcoma lymphoma recurrent
Follicle centre lymphoma diffuse small cell
lymphoma refractory
Lymphoma stage I
Lymphoma stage I
Follicle centre lymphoma diffuse small cell
Follicle centre lymphoma diffuse small cell cell Follicle centre lymphoma diffuse small cell Extraskeletal chondrosarcoma metastatic Extraskeletal chondrosarcoma recurrent Extraskeletal myxoid chondrosarcoma Extraskeletal osteosarcoma metastatic Extraskeletal osteosarcoma metastatic Follicle centre lymphoma diffuse small Fibrosarcoma metastatic .ymphoma

lymphoma stage II Follicle centre lymphoma diffuse small cell lymphoma stage III Follicle centre lymphoma diffuse small cell lymphoma stage IV Follicle centre lymphoma, follicular grade I, II,

Follicle centre lymphoma, follicular grade I, II, III recurrent Follicle centre lymphoma, follicular grade I, II,

III refractory Follicle centre lymphoma, follicular grade I, II,

III stage I Follicle centre lymphoma, follicular grade I, III stage II Follicle centre lymphoma, follicular grade I, III stage III

II,

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 88 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I I |

Follicle centre lymphoma, follicular grade I, II, Follicular dendritic cell sarcoma Follicular dendritic cell sarcoma Follicular thyroid cancer Gallbladder adenocarcinoma Gallbladder adenocarcinoma Gallbladder cancer metastatic Gallbladder cancer recurrent Gallbladder cancer recurrent Gallbladder cancer stage I Gallbladder cancer stage II Gallbladder cancer stage II Gallbladder cancer stage II Gallbladder cancer stage II Gallbladder cancer stage II Gallbladder cancer stage IV Gallbladder cancer stage IV Gallbladder cancer stage II Gallbladder cancer stage II Gastric cancer stage II Gastric cancer stage IV Gastric cancer stage II Gastric cancer stage IV Gastric cancer male accinoma Gastrointestinal adenocarcinoma Gastrointestinal adenocarcinoma Gastrointestinal stromal tumour Gastrointestinal stromal tumour Gastrointestinal accinoma Gastrointestinal cancer male Gastrointestinal Gastro

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: 8 | 89 of 229 |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | |

Novo Nordisk

Malignant tumours (SMQ)

Gestational trophoblastic tumour
Gingival cancer
Glioblastcoma multiforme
Glioblastcoma multiforme
Gliomatosis cerebri
Gliomatosis cerebri
Gliomatosis cerebri
Gliomatosis cerebri
Gliomangioperioytoma
Glounangioperioytoma
Gloudangioperioytoma
Gloudangioperioytoma
Gloudangioperioytoma
HERZ positive breast cancer
HERZ positive breast cancer
HERZ positive gastric cancer
HERZ positive breast cancer
HERZ positive breast cancer
HERZ positive breast cancer
HERZ positive breast cancer
HERZ positive breast cancer
HERZ positive gastric cancer
Head and neck cancer stage II
High grade B-cell lymphoma Burkitt-like lymphoma
stage II
High grade B-cell lymphoma Burkitt-like lymphoma
stage II
High grade B-cell lymphoma Burkitt-like lymphoma
stage III

| ns: | ë: | |
|-----------------------|-------------|-----------------------------|
| Stat | Page | |
| 04 December 2020 | 1.0 | |
| Clinical Trial Report | | - list of preferred terms |
| NN9535 | NN9535-4506 | Pre-defined MedDRA search - |

Pre-defined MedDRA search

Preferred term

Histiocytic medullary reticulosis
Histiocytic sarcoma
Hodgkin's disease
Hodgkin's disease lymphocyte depletion stage I
site unspecified

Hodgkin's disease lymphocyte depletion stage

 $\vdash$ 

subdiaphragm Hodgkin's disease lymphocyte depletion stage supradiaphragm Hodgkin's disease lymphocyte depletion stage

Hodgkin's disease lymphocyte depletion stage site unspecified

ΙΙ Η

ΙΙ

subdiaphragm
Hodgkin's disease lymphocyte depletion stage supradiaphragm
Hodgkin's disease lymphocyte depletion type recurrent

refractory Hodgkin's disease lymphocyte depletion type stage Hodgkin's disease lymphocyte depletion type

Hodgkin's disease lymphocyte depletion type stage Hodgkin's disease lymphocyte depletion type stage Hodgkin's disease lymphocyte predominance stage I unspecified

subdiaphragm Hodgkin's disease lymphocyte predominance stage I site unspec Hodgkin's disease lymphocyte predominance stage Hodgkin's disease lymphocyte predominance stage supradiaphragm

II subdiaphragm Hodgkin's disease lymphocyte predominance II supradiaphragm Hodgkin's disease lymphocyte predominance II site unspec Hodgkin's disease lymphocyte predominance

recurrent
Hodgkin's disease lymphocyte predominance type
refractory
stage lliis disease lymphocyte predominance type
stage llii

Final Novo Nordisk


| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Fir |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 91 of 2 |
| Pre-defined MedDRA search - list of | f preferred terms | | | | |

Preferred term

inal Novo Nordisk

Malignant tumours (SMQ)

Pre-defined MedDRA search

Hodgkin's disease lymphocyte predominance type stage IV
Hodgkin's disease lymphocyte predominance type stage unspecified
Hodgkin's disease mixed cellularity refractory Hodgkin's disease mixed cellularity stage I site unspecified Hodgkin's disease mixed cellularity stage I subdiaphragmatic
Hodgkin's disease mixed cellularity stage I subdiaphragmatic
Hodgkin's disease mixed cellularity stage II supradiaphragmatic
Hodgkin's disease mixed cellularity stage II subdiaphragmatic
Hodgkin's disease mixed cellularity stage II hodgkin's disease mixed cellularity stage III Hodgkin's disease modular sclerosis refractory Hodgkin's disease nodular sclerosis stage II Hodgkin's disease stage II Hodgkin's

Final Novo Nordisk 92 of 229 04 December 2020 | Status: 1.0 Page: Version: Date: Preferred term Clinical Trial Report Pre-defined MedDRA search - list of preferred terms NN9535-4506 NN9535

Malignant tumours (SMQ)

Pre-defined MedDRA search

Hypopharyngeal cancer stage II Hypopharyngeal cancer stage III Hypopharyngeal cancer stage IV Immune reconstitution inflammatory syndrome associated Kaposi's sarcoma Immunoblastic lymphoma

Inflammatory carcinoma of breast recurrent Inflammatory carcinoma of breast stage III Inflammatory carcinoma of breast stage III inflammatory carcinoma of breast stage IV Inflammatory carcinoma of breast stage IV Inflammatory malignant fibrous histiocytoma Inflammatory myofibroblastic tumour Intestinal T-cell lymphoma refractory Intestinal T-cell lymphoma stage II Intestinal T-cell lymphoma stage IV Intestinal T-cell lymphoma stage IV

Intracranial germ cell tumour Intracranial meningioma malignant Intraductal papillary breast neoplasm Intraductal papillary-mucinous carcinoma of Intestinal metastasis

pancreas

Intraductal proliferative breast lesion Intracoular melanoma Invasive breast carcinoma Invasive ductal breast carcinoma Invasive lobular breast carcinoma Invasive papillary breast carcinoma

Juvenile chronic myelomonocytic leukaemia Kaposi's sarcoma

ris melanoma

Kaposi's sarcoma AIDS related Kaposi's sarcoma classical type Keratinising squamous cell carcinoma of

nasopharynx
Keratoacanthoma
Langerhans cell sarcoma
Large cell lung cancer metastatic
Large cell lung cancer metastatic

| NN9535<br>NN9535-4506 | Clinical Trial Report | Date:<br>Version: | 04 December 2020 Status: | Status:<br>Page: | Final<br>93 of 229 | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | ist of preferred terms | | | D | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Large cell lung cancer stage 0
Large cell lung cancer stage II
Large cell lung cancer stage II
Large cell lung cancer stage II
Large cell lung cancer stage III
Large cell lung cancer stage III
Laryngeal cancer metastatic
Laryngeal cancer recurrent
Laryngeal cancer stage II
Lentigo maligna recurrent
Lentigo maligna stage II
Lentigo maligna stage II
Lentigo maligna stage II
Lentiaemia cutis
Leukaemia cutis
Leukaemia cutis
Leukaemic infiltration gingiva
Leukaemic infiltration pulmonary
Leukaemic infiltration renal
Leukaemic infiltration renal
Leukaemic infiltration renal
Leukaemic retinopathy
Leukaemic retinopathy
Leukaemic retinopathy
Leukaemic retinopathy
Leukaemic retinopathy

04 December 2020 | Status: 1.0 | Page: Version: Date: | Clinical Trial Report NN9535-4506 NN9535

Preferred term

Pre-defined MedDRA search - list of preferred terms

Malignant tumours (SMQ)

Lip and/or oral cavity cancer
Lip and/or oral cavity cancer stage I
Lip and/or oral cavity cancer stage I
Lip and/or oral cavity cancer stage II
Lip and/or oral cavity cancer stage III
Lip and/or oral cavity cancer stage III
Lip and/or oral cavity cancer stage III
Lip neoplasm malignant stage unspecified
Liposarcoma metastatic
Liposarcoma metastatic
Liposarcoma recurrent
Liposarcoma recurrent
Liposarcoma recurrent
Linum adenocarcinoma stage III
Linum adenocarcinoma stage III
Linum adenocarcinoma stage III
Linum adenocarcinoma stage III
Lium adenocarcinoma stage III
Lium adenocarcinoma capa III
Lium adenocarcinoma capa III
Lium adenocarcinoma capa III
Lium carcinoma call type unspecified stage II
Lium carcinoma cell type unspecified stage II
Lium carcinoma cell type unspecified stage III
Liung carcinoma cell type unspecified stage III
Liung squamous cell carcinoma recurrent squamous cell carcinoma stage 0 squamous cell carcinoma stage I squamous cell carcinoma stage II squamous cell carcinoma stage III squamous cell carcinoma stage III Lymphangiosis carcinomatosa Lymphocytic leukaemia Lymphocytic lymphoma Lymphoid leukaemia (in remission) ymphangiosarcoma Lung Lung Lung Lung Lung Lung

Lymphoma AIDS related

Final Novo Nordisk


Pre-defined MedDRA search

Final Novo Nordisk 95 of 229 04 December 2020 | Status: 1.0 Page: Version: Date: | Clinical Trial Report Pre-defined MedDRA search - list of preferred terms NN9535-4506 NN9535

Preferred term

Malignant tumours (SMQ)

Pre-defined MedDRA search

Lymphoplasmacytoid lymphoma/immunocytoma
Lymphoplasmacytoid lymphoma/immunocytoma
Lymphoplasmacytoid lymphoma/immunocytoma
refractory
Lymphoplasmacytoid lymphoma/immunocytoma stage II
Malignant fibrous histiocytoma metastatic
Malignant fibrous histiocytoma metastatic
Malignant fibrous histiocytoma metastatic
Malignant fibrous histiocytoma metastatic
Malignant haemangiopericytoma metastatic
Malignant haemangiopericytoma metastatic
Malignant haemangiopericytoma metastatic
Malignant lymphoma unclassifiable high grade
Malignant lymphoma unclassifiable low grade
Malignant melanoma of eyelid
Malignant melanoma stage II
Malignant melanoma stage II
Malignant melanoma stage II
Malignant melanoma stage II
Malignant melanoma stage II
Malignant melanoma stage II
Malignant melanoma stage II
Malignant mesenchymoma metastatic
Malignant mesenchymoma metastatic
Malignant mesenchymoma recurrent

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 96 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Malignant tumours (SMQ)

Malignant mesenteric neoplasm
Malignant middle ear neoplasm
Malignant muscle neoplasm
Malignant neoplasm of ampulla of Vater
Malignant neoplasm of choroid
Malignant neoplasm of conjunctiva
Malignant neoplasm of eyelid
Malignant neoplasm of islets of Langerhans
Malignant neoplasm of islets of Langerhans
Malignant neoplasm of lacrimal gland
Malignant neoplasm of paraurethral glands
Malignant neoplasm of placenta
Malignant neoplasm of placenta
Malignant neoplasm of placenta
Malignant neoplasm of placenta
Malignant neoplasm of pleura metastatic
Malignant neoplasm of seminal vesicle
Malignant neoplasm of seminal orda
Malignant neoplasm of seminal orda
Malignant neoplasm of seminal orda
Malignant neoplasm of thorax
Malignant neoplasm of thorax
Malignant neoplasm of thorax
Malignant neoplasm of threina adnexa
Malignant neoplasm of threina adnexa
Malignant neoplasm of threina
Malignant neoplasm of unknown primary site
Malignant neoplasm of theria adnexa
Malignant neoplasm of thorax
Malignant neoplasm of unknown primary site
Malignant nipple neoplasm
Malignant placentanolysm
Malignant placentanolysm
Malignant pericardial neoplasm
Malignant pericardial neoplasm
Malignant pericardial neoplasm
Malignant respiratory tract neoplasm
Malignant respiratory tract neoplasm
Malignant transformation
Malignant urinary tract neoplasm
Malignant transformation
Malignant urinary tract neoplasm

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 97 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | : preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Mantle cell lymphoma recurrent
Mantle cell lymphoma refractory
Mantle cell lymphoma stage I
Mantle cell lymphoma stage II
Mantle cell lymphoma stage II
Mantle cell lymphoma stage III
Mantle cell lymphoma stage III
Marginal zone lymphoma recurrent
Marginal zone lymphoma refractory
Marginal zone lymphoma stage II
Marginal zone lymphoma stage II
Marginal zone lymphoma stage II
Marginal zone lymphoma stage II
Marginal zone lymphoma stage II
Marginal zone lymphoma stage II
Marginal zone lymphoma stage IV
Marginal zone in pregnancy
Mature B-cell type acute leukaemia
Medullary carcinoma of breast
Medullary thyroid cancer
Medulloblastoma recurrent Metastases to central nervous system Metastases to chest wall Metastases to diaphragm Mesothelioma malignant
Mesothelioma malignant recurrent
Metaplastic breast carcinoma
Metastases to Eustachian tube
Metastases to abdominal cavity
Metastases to abdominal wall Metastases to adrenals
Metastases to biliary tract
Metastases to bone
Metastases to bone
Metastases to bone marrow
Metastases to bonesta Meningioma malignant Metastases to e Metastases to f Metastases to g

to fallopian tube to gallbladder to gastrointestinal tract

Metastases

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 98 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

o perineum
o peripheral nervous system
o peripheral vascular system
o peritoneum
o pharynx
o pituitary gland the mediastinum the respiratory system rectum reproductive organ retroperitoneum salivary gland mouth muscle nasal sinuses nervous system oesophagus skin soft tissue spinal cord lymph nodes meninges ovary pancreas pelvis placenta pleura prostate testicle spine spleen stomach thorax thyroid tonsils trachea heart kidney larynx liver penis neck lung t t t t t けつ 4444 to t t t t to to 2 2 2 2 2 2 to to to to たり to to けつ Metastasses
Metastasses
Metastasses Metastases t Metastases

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 99 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | l I |

Metastases to urinary tract
Metastases to uterus
Metastasis
Metastatic vagina
Metastatic bronchial carcinoma
Metastatic carcinoma of the bladder
Metastatic carcinoma of the bladder
Metastatic carcinoma of the bladder
Metastatic glioma
Metastatic glioma
Metastatic lymphoma
Metastatic lymphoma
Metastatic lymphoma
Metastatic neoplasm
Metastatic neoplasm
Metastatic neoplasm
Metastatic coular melanoma
Metastatic coular melanoma
Metastatic coular melanoma
Metastatic coular melanoma
Metastatic coular melanoma
Metastatic coular melanoma
Metastatic levious system neoplasm
Metastatic salivary gland cancer
Metastatic salivary gland cancer
Metastatic uterine cancer
Metastatic uterine cancer
Metastatic levious coll carcinoma
Mixed-type liposarcoma
Mixed-type liposarcoma
Mixed-type liposarcoma
Mucinous breast carcinoma of appendix
Mucinous cystedenocarcinoma of appendix
Mucinous cystedenocarcinoma of salivary gland
Musculoskeletal cancer
Myeloid leukaemia

Final Novo Nordisk 100 of 229 04 December 2020 | Status: 1.0 Page: Version: Date: | Clinical Trial Report Pre-defined MedDRA search - list of preferred terms NN9535-4506 NN9535

Preferred term

Malignant tumours (SMQ)

Pre-defined MedDRA search

Nasopharyngeal cancer metastatic
Nasopharyngeal cancer recurrent
Nasopharyngeal cancer stage 0
Nasopharyngeal cancer stage 1
Nasopharyngeal cancer stage 11
Nasopharyngeal cancer stage 11
Nasopharyngeal cancer stage 11
Nasopharyngeal cancer stage 11
Nasopharyngeal cancer stage 11
Nasopharyngeal cancer stage 11
Natural killer-cell leukaemia
Natural killer-cell leukaemia
Neonatal leukaemia
Neonatal leukaemia
Neonatal neuroblastoma
Neoplasm malignant
Neurochocrine carcinoma
Neurochocrine carcinoma
Neurochocrine carcinoma of prostate
Neurochocrine carcinoma of the skin
Neurochocrine carcinoma of the bladder
Neurochocrine carcinoma of the bladder
Neurochocrine tumour of the lung metastatic
Neurochocrine tumour of the lung metastatic
Neurochocrine tumour of the lung metastatic
Neurochocrine tumour of the lung metastatic
Neurofibrosarcoma metastatic
Neurofibrosarcoma recurrent
Nodal marginal zone B-cell lymphoma stage II
Non-Hodgkin's lymphoma refractory
Non-Hodgkin's lymphoma refractory
Non-Hodgkin's lymphoma stage II
Non-Hodgkin's lymphoma stage III

04 December 2020 | Status: Version: Clinical Trial Report Pre-defined MedDRA search - list of preferred terms NN9535-4506 NN9535

Preferred term

Malignant tumours (SMQ)

indolent stage IV

Non-renal cell carcinoma of kidney

Non-small cell lung cancer metastatic

Non-small cell lung cancer recurrent

Non-small cell lung cancer stage 0

Non-small cell lung cancer stage II

Non-small cell lung cancer stage II

Non-small cell lung cancer stage II

Non-small cell lung cancer stage III

Non-small cell lung cancer stage III

Non-small cell lung cancer stage IIIA

Non-small cell lung cancer stage IIIA

Non-small cell lung cancer stage IIIA

Non-small cell lung cancer stage IIIA

Non-small cell lung cancer stage IIIA

Non-small cell lung cancer stage IIIA

Non-small cell lung cancer stage IIIA

Non-small cell lung cancer stage IV

Nongerminomatous germ cell tumour of the CNS

Nonkeratinising carcinoma of nasopharynx indolent stage I Non-Hodgkin's lymphoma unspecified histology indolent stage II Non-Hodgkin's lymphoma unspecified histology indolent stage III Non-Hodgkin's lymphoma unspecified histology Non-Hodgkin's lymphoma stage IV Non-Hodgkin's lymphoma transformed recurrent Non-Hodgkin's lymphoma unspecified histology aggressive refractory
Non-Hodgkin's lymphoma unspecified histology
aggressive stage I
Non-Hodgwin's lymphoma unspecified histology
aggressive stage II
Non-Hodgkin's lymphoma unspecified histology aggressive stage III Non-Hodgkin's lymphoma unspecified histology aggressive stage IV Non-Hodgkin's lymphoma unspecified histology aggressive recurrent Non-Hodgkin's lymphoma unspecified histology aggressive Non-Hodgkin's lymphoma unspecified histology Non-Hodgkin's lymphoma unspecified histology Ocular cancer metastatic Ocular haemangiopericytoma Ocular lymphoma Oesophageal adenocarcinoma indolent

Final Novo Nordisk


Pre-defined MedDRA search

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Novo N |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 102 of 229 | |
| Pre-defined MedDRA search - list of preferred | f preferred terms | | | | | |
| | | | | | | ı |
| Pre-defined MedDRA search | Preferred term | | | | | |

Nordisk

Malignant tumours (SMQ)

Oesophageal adenocarcinoma stage 0
Oesophageal adenocarcinoma stage 1
Oesophageal adenocarcinoma stage II
Oesophageal adenocarcinoma stage II
Oesophageal adenocarcinoma stage III
Oesophageal adenocarcinoma stage III
Oesophageal adenosquamous carcinoma
Oesophageal cancer metastatic
Oesophageal carcinoma recurrent
Oesophageal carcinoma stage 0
Oesophageal squamous cell carcinoma metastatic
Oesophageal squamous cell carcinoma recurrent
Oesophageal squamous cell carcinoma stage 0
Oesophageal squamous cell carcinoma stage 1
Oesophageal squamous cell carcinoma stage II
Oesophageal squamous cell carcinoma stage II
Oesophageal squamous cell carcinoma stage II
Oesophageal squamous cell carcinoma stage II
Oesophageal squamous cell carcinoma stage III
Oesophageal squamous cell carcinoma stage III
Oesophageal squamous cell carcinoma stage III
Oesophageal squamous cell carcinoma stage IV
Oliqoastrocytoma

Oligoastrocytoma
Oligoastrocytoma
Oligodendroglioma
Optic glioma
Oral cavity cancer metastatic
Oropharyngeal cancer stage I
Oropharyngeal cancer stage II
Oropharyngeal cancer stage II
Oropharyngeal cancer stage II
Oropharyngeal cancer stage II
Oropharyngeal cancer stage II
Oropharyngeal lymphoepithelioma
Oropharyngeal lymphoepithelioma
Oropharyngeal lymphoepithelioma
Oropharyngeal squamous cell carcinoma
Osteosarcoma
Osteosarcoma
Osteosarcoma
Osteosarcoma recurrent
Otic cancer metastatic
Ovarian cancer metastatic
Ovarian cancer metastatic
Ovarian cancer recurrent
Ovarian cancer stage II
Ovarian cancer stage II
Ovarian cancer stage III
Ovarian cancer stage III
Ovarian cancer stage III
Ovarian cancer stage III

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Sta | itus: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 Pa | ge: | 103 of 229 | |
| Pre-defined MedDRA search - list of preferred | f preferred terms | | | | | |

Pre-defined MedDRA search

Malignant tumours (SMQ)

clear cell carcinoma

Preferred term

Ovarian embryonal carcinoma ovarian embryonal carcinoma ovazian embryonal carcinoma ovazian embryonal carcinoma ovazian epithelial cancer metastatic
Ovarian epithelial cancer stage II
Ovarian epithelial cancer stage II
Ovarian epithelial cancer stage II
Ovarian epithelial cancer stage II
Ovarian epithelial cancer stage II
Ovarian germ cell cancer stage II
Ovarian germ cell cancer stage II
Ovarian germ cell choriocarcinoma stage II
Ovarian germ cell choriocarcinoma stage II
Ovarian germ cell choriocarcinoma stage II
Ovarian germ cell embryonal carcinoma stage II
Ovarian germ cell endodermal sinus tumour stage II
Ovarian germ cell endodermal sinus tumour stage II Ovarian germ cell endodermal sinus tumour stage IV Ovarian germ cell polyembryoma stage I Ovarian germ cell polyembryoma stage I Ovarian germ cell polyembryoma stage II Ovarian germ cell polyembryoma stage III Ovarian germ cell polyembryoma stage IV Ovarian germ cell teratoma stage IV Ovarian germ cell teratoma stage I Ovarian germ cell teratoma stage II Ovarian clear cell carcinoma
Ovarian dysgerminoma stage I
Ovarian dysgerminoma stage II
Ovarian dysgerminoma stage III
Ovarian dysgerminoma stage IV
Ovarian dysgerminoma stage unspecified

| NN9535<br>NNIO628 4506 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| 000+0006 | 1 | v etstorii. | 0.1 | rage. | 10+01 773 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Dre-defined MedhRA search | Drafarrad tarm | | | | | |

Ovarian germ cell teratoma stage III
Ovarian germ cell teratoma stage IV
Ovarian germ cell teratoma stage IV
Ovarian granulosa-theca cell tumour
Ovarian pranulosa-theca cell tumour
Ovarian melanoma
Ovarian stromal cancer
Paget's disease of penis
Paget's disease of penis
Paget's disease of penis
Paccatic carcinoma stage II
Pancreatic carcinoma stage II
Pancreatic carcinoma stage II
Pancreatic carcinoma stage IV
Pancreatic neuroendocrine tumour metastatic
Parceatic neuroendocrine tumour metastatic
Pancreatic neuroendocrine tumour pancreatic neuroendocrine tumour metastatic
Pancreatic sarcoma
Papillary renal call carcinoma
Papillary thyroid cancer
Paranasal sinus and nasal cavity malignant neoplasm stage II
Paranasal sinus and nasal cavity malignant neoplasm stage II
Paranasal sinus and nasal cavity malignant neoplasm stage III

| NN9535 | Clinical Trial Report | Date: 0 | 4 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 105 of 229 | |
| Pre-defined MedDRA search - list of preferred | f preferred terms | | | | | |

Preferred term

Malignant tumours (SMQ)

Pre-defined MedDRA search

Penile squamous cell carcinoma
Penis carcinoma metastatic
Penis carcinoma stage II
Penis carcinoma stage II
Penis carcinoma stage III
Penis carcinoma stage III
Penis carcinoma stage III
Penis carcinoma stage III
Penis carcinoma stage III
Penis carcinoma stage III
Penis carcinoma stage III
Periotal mesothelioma malignant recurrent
Periotaral T-cell lymphoma unspecified recurrent
Peripheral T-cell lymphoma unspecified recurrent
Peripheral T-cell lymphoma unspecified stage II
Peripheral T-cell lymphoma unspecified stage II
Peripheral T-cell lymphoma unspecified stage II
Peripheral neuroepithelioma of bone metastatic
Peripheral neuroepithelioma of bone metastatic
Peripheral pruncopithelioma of bone recurrent
Peripheral primitive neuroectodermal bone tumour

Peritoneal carcinoma metastatic
Peritoneal mesothelioma malignant
Peritoneal ascone
Pritoneal sarcoma
Phaeochromocytoma malignant recurrent
Pharyngeal cancer
Pharyngeal cancer recurrent
Pharyngeal cancer recurrent
Pharyngeal cancer stage 0
Pharyngeal cancer stage 1
Pharyngeal cancer metastatic
Pituitary cancer metastatic
Pituitary neoplasm malignant recurrent
Plasma cell leukaemia

soft tissue

04 December 2020 | Status: 1.0 Page: Version: Date: Clinical Trial Report NN9535-4506 NN9535

Preferred term

Final Novo Nordisk


Pre-defined MedDRA search - list of preferred terms

Malignant tumours (SMQ)

Pre-defined MedDRA search

Plasma cell leukaemia in remission Plasma cell myeloma Plasma cell myeloma in remission Plasma cell myeloma recurrent Plasma cell myeloma refractory Plasmablastic lymphoma Plasmacytoma

Pleomorphic leiomyosarcoma Pleomorphic liposarcoma Pleomorphic malignant fibrous histiocytoma Pleural mesothelioma malignant Pleural mesothelioma malignant recurrent Pleural mesothelioma

Pleural sarcoma Pleuropulmonary blastoma Poorly differentiated thyroid carcinoma

Porocarcinoma

Postcricoid cancer
Precursor B-lymphoblastic lymphoma recurrent
Precursor B-lymphoblastic lymphoma refractory
Precursor B-lymphoblastic lymphoma stage I
Precursor B-lymphoblastic lymphoma stage II
Precursor B-lymphoblastic lymphoma stage II
Precursor B-lymphoblastic lymphoma stage II
Precursor B-lymphoblastic lymphoma stage III
Precursor B-lymphoblastic lymphoma stage IV
Precursor T-lymphoblastic lukaemia acute
Precursor T-lymphoblastic lukaemia lukaemia

Precursor T-lymphoblastic lymphoma/leukaemia Precursor T-lymphoblastic lymphoma/leukaemia refractory

recurrent

Precursor T-lymphoblastic lymphoma/leukaemia stage II Precursor T-lymphoblastic lymphoma/leukaemia stage III

Precursor T-lymphoblastic lymphoma/leukaemia

Primary breast lymphoma
Primary cardiac lymphoma
Primary effusion lymphoma
Primary gastrointestinal follicular lymphoma

| JN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| 9535-4506 | | Version: | 1.0 | Page: | 107 of 229 | |
| Pre-defined MedDRA search - list of preferred | preferred terms | | | | | |

Preferred term

Malignant tumours (SMQ)

Pre-defined MedDRA search

Primary mediastinal large B-cell lymphoma recurrent Primary mediastinal large B-cell lymphoma recurrent Primary mediastinal large B-cell lymphoma stage In Primary mediastinal large B-cell lymphoma stage II Primary mediastinal large B-cell lymphoma stage II Primary mediastinal large B-cell lymphoma stage II Primary mediastinal large B-cell lymphoma stage II Primary pulmonary melanoma Primitive neuroectodermal tumour Prostate cancer stage II Rectal cancer stage II Rectosigmoid cancer stage II Recto

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 108 of 229 | |
| Pre-defined MedDRA search - list of preferre | preferred terms | | | | | |

Preferred term

Malignant tumours (SMQ)

Pre-defined MedDRA search

Renal cancer metastatic
Renal cancer recurrent
Renal cancer stage II
Renal cancer stage II
Renal cancer stage II
Renal cancer stage III
Renal cancer stage IV
Renal cell carcinoma recurrent
Renal cell carcinoma stage II
Renal cell carcinoma stage II
Renal cell carcinoma stage II
Renal cell carcinoma stage II
Renal cell carcinoma stage II
Renal cell carcinoma stage II
Renal cell carcinoma stage II
Respiratory tract carcinoma in situ
Retinoblastoma

Retroperitoneal cancer
Retroperitoneal neoplasm metastatic
Rhabdoid tumour
Rhabdomyosarcoma
Rhabdomyosarcoma recurrent
Richter's syndrome
Round cell liposarcoma
Salivary gland cancer recurrent
Salivary gland cancer stage 0
Salivary gland cancer stage 1
Salivary gland cancer stage 1
Salivary gland cancer stage 1
Salivary gland cancer stage 1
Salivary gland cancer stage 1
Salivary gland cancer stage 11
Salivary gland cancer stage 11
Salivary gland cancer stage 11
Salivary gland cancer stage 11
Salivary gland cancer stage 11
Salivary gland cancer stage 11

Sarcoma metastatic
Sarcoma metastatic
Sarcoma of skin
Sarcoma therus
Sarcomatoid carcinoma
Sarcomatoid carcinoma
Sarcomatoid mesothelioma

Sarcomatold carcinoma of the Sarcomatold mesothelioma Sarcomatosis Scrotal cancer Sebaceous carcinoma Second primary malignancy Seminoma

109 of 229 04 December 2020 | Status: 1.0 | Page: Version: Date: Preferred term | Clinical Trial Report Pre-defined MedDRA search - list of preferred terms Pre-defined MedDRA search NN9535-4506 NN9535

Malignant tumours (SMQ)

Soft Lissue sarcoma Solid pseudopapillary tumour of the pancreas Spermatocytic seminoma Spinal meningioma malignant Spinal meningioma malignant Spinale cell sarcoma Splenic marginal zone lymphoma recurrent Splenic marginal zone lymphoma refractory Splenic marginal zone lymphoma stage I Splenic marginal zone lymphoma stage II Splenic marginal zone lymphoma stage II Splenic marginal zone lymphoma stage II Splenic marginal zone lymphoma stage II Splenic marginal zone lymphoma stage II Splenic marginal zone lymphoma stage IV Skin cancer metastatic
Skin cancer metastatic
Skin squamous cell carcinoma metastatic
Skin squamous cell carcinoma recurrent
Small cell carcinoma of the cervix
Small cell lung cancer extensive stage
Small cell lung cancer metastatic
Small cell lung cancer metastatic
Small cell lung cancer metastatic
Small intestine adenocarcinoma
Small intestine carcinoma metastatic
Small intestine carcinoma stage 0
Small intestine carcinoma stage 1
Small intestine carcinoma stage 1
Small intestine carcinoma stage 11
Small intestine carcinoma stage 11
Small intestine carcinoma stage 11
Small intestine carcinoma stage 11
Small intestine carcinoma stage 11
Small intestine carcinoma stage 11 Squamous cell breast carcinoma
Squamous cell carcinoma
Squamous cell carcinoma of head and neck
Squamous cell carcinoma of lung
Squamous cell carcinoma of pharynx
Squamous cell carcinoma of skin Serous cystadenocarcinoma ovary Signet-ring cell carcinoma Sinus cancer metastatic Skin angiosarcoma

Final Novo Nordisk

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | ģ |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 110 of 229 | |
| Pre-defined MedDRA search - list of preferred | : preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Squamous cell carcinoma of the cervix
Squamous cell carcinoma of the hypopharynx
Squamous cell carcinoma of the parotid gland
Squamous cell carcinoma of the parotid gland
Squamous cell carcinoma of the tongue
Squamous cell carcinoma of the vagina
Squamous cell carcinoma of the vagina
Squamous cell carcinoma of the valva
Squamous cell carcinoma of the valva
Squamous cell carcinoma
Squamous cell carcinoma
Squamous cell carcinoma
Squamous cell carcinoma
Squamous cell carcinoma
Squamous cell carcinoma
Squamous cell carcinoma
Squamous call carcinoma
Squamous stage II
Superficial spreading melanoma stage III
Superficial spreading melanoma
Squamous carcoma
Squamous carcoma
Squamous stage II
T-cell lymphoma
T-cell lymphoma
T-cell lymphoma
Stage II
T-cell lymphoma
Stage III
T-cell lymphoma
Stage II
T-cell lymphoma
Stage III
T-cell lymphoma
Stage II
T-cell lymphoma
Stage II
T-cell lymphoma
Stage III
T-cell lymphoma
Stage III
T-cell lymphoma
T-cell lymphoma
Stage III
T-cell lymphoma
Stage III
T-cell lymphoma
Stage III
T-cell lymphoma
Stage III
T-cell lymphoma
Stage II
T-cell lymphoma
Stage III
T-cel Testicular cancer metastatic
Testicular choriocarcinoma recurrent
Testicular choriocarcinoma stage I
Testicular choriocarcinoma stage I
Testicular choriocarcinoma stage II
Testicular embryonal carcinoma
Testicular embryonal carcinoma stage II
Testicular embryonal carcinoma stage II
Testicular embryonal carcinoma stage II
Testicular embryonal carcinoma stage II
Testicular embryonal carcinoma stage II
Testicular germ cell cancer
Testicular germ cell cancer metastatic
Testicular germ cell cancer metastatic
Testicular germ cell tumour mixed
Testicular germ cell tumour mixed

ovo Nordisk

| NN9535 | Clinical Trial Report | Date: ( | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 111 of 229 | |
| Pre-defined MedDRA search - list of preferred | preferred terms | | | | | |

Preferred term

Malignant tumours (SMQ)

Pre-defined MedDRA search

Testicular germ cell tumour mixed stage II
Testicular malignant teratoma
Testicular malignant teratoma stage III
Testicular malignant teratoma stage III
Testicular malignant teratoma stage III
Testicular seminoma (pure)
Testicular seminoma (pure) stage III
Testicular seminoma (pure) stage III
Testicular seminoma (pure) stage III
Testicular seminoma (pure) stage III
Testicular seminoma (pure) stage III
Testicular yolk sac tumour stage III
Testicular yolk sac tumour stage III
Testicular yolk sac tumour stage III
Thymoma malignant
Testis cancer
Thymoma malignant
Thymoma malignant recurrent
Thymoma malignant recurrent
Thymoid cancer stage III
Thyroid cancer stage III
Thyroid cancer metastatic
Tongue carcinoma stage II
Tongue neoplasm malignant stage unspecified
Tongue carcinoma stage II
Tongue carcinoma stage III
Tongue carcin
| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 112 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | - | | I |

Malignant tumours (SMQ)

Transitional cell cancer of renal pelvis and ureter metastatic
Transitional cell cancer of the renal pelvis and ureter
Transitional cell cancer of the renal pelvis and ureter localised
Transitional cell cancer of the renal pelvis and ureter recurrent
Transitional cell cancinoma metastatic
Transitional cell carcinoma metastatic
Transitional cell carcinoma urethra
Transitional cell carcinoma urethra
Transitional cell carcinoma urethra
Transitional cell carcinoma urethra
Triple hit lymphoma
Triple hit lymphoma
Triple positive breast cancer
Triple positive breast cancer
Triple positive breast cancer
Triple positive breast cancer
Triple positive breast cancer
Triple cancer ascopharyngeal carcinoma
Undifferentiated carcinoma
Undifferentiated sarcoma
Ureteric cancer recurrent
Ureteric cancer recurrent
Ureteric cancer recurrent
Ureterial cancer recurrent
Urethral cancer recurrent
Urethral cancer metastatic
Urethral melanoma metastatic

Urinary bladder sarcoma Urinary tract carcinoma in situ Uterine cancer

Uterine carcinoma in situ Uterine leiomyosarcoma

Uveal melanoma

Vaginal adenocarcinoma Vaginal cancer Vaginal cancer metastatic Vaginal cancer recurrent Vaginal cancer stage 0

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 113 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | 1 1 |

Vaginal cancer stage II
Vaginal cancer stage III
Vaginal cancer stage III
Vaginal cancer stage IVA
Vaginal cancer stage IVB
Vulval cancer metastatic
Vulval cancer recurrent
Vulval cancer stage II
Vulval cancer stage II
Vulval cancer stage II
Vulval cancer stage II
Vulval cancer stage III
Vulval cancer stage III
Vulval cancer stage III
Vulval cancer stage III
Vulval cancer stage IV
Vulval cancer stage III
Vulval cancer stage III
Vulval cancer stage IV
Vulval cancer stage IV
Vulvar basal cell carcinoma
Waldenstrom's macroglobulinaemia refractory
Waldenstrom's macroglobulinaemia stage II
Waldenstrom's macroglobulinaemia stage II
Waldenstrom's macroglobulinaemia stage II
Waldenstrom's macroglobulinaemia stage III
Waldenstrom's macroglobulinaemia stage III
Waldenstrom's macroglobulinaemia stage III
Waldenstrom's macroglobulinaemia stage III Medication error overdose Malignant tumours (SMQ)

Documented hypersensitivity to administered

product

Accidental device ingestion
Accidental device ingestion by a child
Accidental exposure to product
Accidental exposure to product by child
Accidental exposure to product packaging
Accidental exposure to product packaging by child
Accidental overdose
Accidental poisoning
Accidental underdose
Accidental underdose
Accidental use of placebo
Assisted suicide

device use error
Circumstance or information capable of leading to medication error
Completed suicide
Contraindicated device used Booster dose missed Circumstance or information capable of leading to  $\ensuremath{\mathsf{C}}$ 

| NN9535 Clinical Trial Report Date: 04 December 2020 Status: NN9535-4506 - 1.0 Page: |
|---|

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Pre-defined MedDRA search

Medication error overdose

Drug dose omission by device
Drug dose titration not performed
Drug monitoring procedure incorrectly performed
Drug monitoring procedure not performed
Drug minitation error Device monitoring procedure not performed Device placement issue Device programming error Device use confusion Device use error Contraindicated product administered Contraindicated product prescribed Contraindication to medical treatment Contraindication to vaccination Dietary supplement prescribing error Discontinued product administered Dopamine dysregulation syndrome Dose calculation error Drug administered in wrong device Drug delivery system issue Drug delivery system malfunction Drug dependence dispensed to wrong patient Drug use disorder, antepartum Drug use disorder, postpartum Duplicate therapy error Expired device used Expired product administered Device-device incompatibility Drug dependence, antepartum Drug dependence, postpartum Drug dispensed to wrong pati dependence antepartum Device difficult to use Device dispensing error Device infusion issue Device maintenance issue Device malfunction Device monitoring procedur Device placement issue Device programming error Device use confusion connection issue difficult to use dispensing error infusion issue Device adhesion issue Deprescribing error Device use issue Drug abuser Drug abuse Device

| NN9535 | Clinical Trial Report | Date: ( | 94 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 115 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |

Medication error overdose

Pre-defined MedDRA search

Exposure to contaminated device
Exposure via contaminated device
Exposure via contaminated device
Exposure via direct contact
Exposure via indestion
Exposure via ingestion
Exposure via ingestion
Exposure via ingestion
Exposure via ingestion
Exposure via ingestion
Exposure via ingestion
Exposure via ingestion
Exposure via okin contact
Exposure via uknown route
Exposure via okin contact
Exposure via uknown route
Exposure via okin contact
Exposure via skin contact
Exposure via skin contact
Exposure via uknown route
Exposure via okin contact
Exposure via uknown route
Exposure via okin contact
Incomplete course of vaccination
Incorrect dosage administered
Incorrect dosage administered
Incorrect dosage administered by product
Incorrect dosage administered by product
Incorrect product doministered by product
Incorrect product doministered by device
Incorrect product formulation administered
Incorrect product formulation administered
Intentional device misses
Intentional device misses
Intentional solf-injury
Intercepted medication error
Intercepted product misuse
Intercepted product dispensing error
Intercepted product ministration error
Intercepted product prescribing error
Intercepted product prescribing error
Intercepted product prescribing error
Intercepted product selected
Intercepted product selected
Intercepted product selected

| NN9535 | Clinical Trial Report | Date: 04 D | 04 December 2020 Status: | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | .0 Page: 116 | 116 of 229 |
| Pre-defined MedDRA search - list of prefer | f preferred terms | | | | |

Novo Nordisk

Medication error overdose

Pre-defined MedDRA search

Interchange of vaccine products
Labelled drug-disease interaction medication error
Labelled drug-disease interaction medication error
Labelled drug-food interaction medication error
Lack of administration site rotation
Lack of injection site rotation
Lack of injection site rotation
Lack of injection site rotation
Lack of injection site rotation
Lack of injection site rotation
Maternal use of illicit drugs
Medicatlon error
Medication error
Medication error
Multiple use of single-use product
Needle issue
Neodle issue
Neodle issue
Neodle issue
Neodle issue
Neodle issue
Neodle issue
Por quality product use product
Occupational exposure to radiation
Out of specification product use
Nerdose
Personne enhanistration
Performance enhanistration
Performed deliberate
Poor quality product administered to patient of inappropriate
Product administered to patient of inappropriate
Product administeration interrupted
Product administeration interrupted
Product administration interrupted
Product administration interrupted
Product administration interrupted
Product administration issue
Product communication
Product design confusion
Product design confusion
Product design confusion
Product dispensing error
Product dispensing error
Product dosage form confusion
Product dosage form confusion
Product dosage form confusion
Product dosage form confusion

| NN9535 | Clinical Trial Report | Date: 04 | 14 December 2020 Status: | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 17 of 229 |
| Pre-defined MedDRA search - list of preferr | f preferred terms | | | | |

Medication error overdose

Product dose omission
Product dropper issue
Product label confusion
Product label confusion
Product label issue
Product label issue
Product label on wrong product
Product monitoring error
Product monitoring error
Product packaging confusion
Product packaging difficult to open
Product preparation error
Product preparation issue
Product prescribing issue
Product prescribing issue
Product prescribing issue
Product prescribing issue
Product selection error
Product selection error
Product substitution error
Product use complaint
Product use complaint
Product use in unapproved therapeutic environment
Product use in unapproved therapeutic Therapeutic drug monitoring analysis not performed Transcription medication error Transfusion with incompatible blood Therapeutic drug monitoring analysis incorrectly Radiation underdose Recalled product administered Single component of a two-component product administered Suicide attempt Suspected suicide Suspected suicide attempt Substance use disorder Substance dependence Radiation overdose Substance abuser Substance abuse Syringe issue performed

Underdose

Novo Nordisk

Pre-defined MedDRA search

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo No |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | 1.0 Page: | 118 of 229 | |
| Pre-defined MedDRA search - list of preferred to | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ı |

Unintentional medical device removal Unintentional use for unapproved indication Vaccination error Wrong dosage form
Wrong dosage form
Wrong dosage formulation
Wrong dosage formulation
Wrong drug
Wrong patient received product
Wrong product administered
Wrong product procured
Wrong product stored
Wrong rate
Wrong schedule
Wrong strength
Wrong strength
Wrong technique in device usage process
Wrong technique in product usage process Medication error overdose Neoplasm

Cerebral cyst hammorrhage
Inferior vena cava syndrome
Intracranial tumour hammorrhage
Langerhans' cell histiocytosis
Multiple gated acquisition scan abnormal
Paraneoplastic thrombosis
Pulmonary tumour thrombotic microangiopathy Benign hepatic neoplasm
Benign hepatobiliary neoplasm
Biopsy liver abnormal
Cholangiosarcoma
Computerised tomogram liver abnormal
Focal nodular hyperplasia Scan myocardial perfusion abnormal Superior vena cava occlusion Superior vena cava syndrome Thrombophlebitis migrans Biopsy bile duct abnormal Biopsy gallbladder abnormal Malignant biliary obstruction Acquired Cl inhibitor deficiency Biopsy heart abnormal Tumour thrombectomy Tumour thrombosis

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 119 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Hepatic angiosarcoma
Hepatic angiosarcoma
Hepatic cancer
Hepatic cancer metastatic
Hepatic cancer stage II
Hepatic cancer stage II
Hepatic cancer stage II
Hepatic cancer stage II
Hepatic cancer stage II
Hepatic cancer stage IV
Hepatic cancer stage IV
Hepatic cancer stage IV
Hepatic cancer stage IV
Hepatic cancer stage IV
Hepatic hamartoma
Hepatic hamartoma
Hepatic hamartoma
Hepatic hamartoma
Hepatic hamartoma
Hepatic neoplasm
Hepatobiliary cancer
Hepatobiliary cancer
Hepatobiliary cancer
Hepatobiliary neoplasm
Hepatobiliary neoplasm
Hepatobiliary neoplasm
Hepatobiliary neoplasm
Hepatobiliary cancer
Hepatobiliary cancer
Hepatobiliary peoplasm
Hepatobiliary peoplasm
Hepatobiliary carcinoma recurrent
Hepatobiliary peoplasm
Hepatobiliary peoplasm
Inver ablation
Liver acronoma ruptured
Liver acronoma ruptured
Liver acronoma ruptured
Liver acronoma la lud postor
Ampullary polyp
Anal leukoplakia
Anal leukoplakia
Anal leukoplakia
Colon dysplasia
Colon dysplasia
Colon dysplasia
Colon dysplasia
Colon dysplasia
Colon dysplasia
Duodenal polyp
Epulis Haemangioma of liver Haemorrhagic hepatic cyst Hepatectomy

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 120 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ı |

Neoplasm

Gastric cyst
Gastric dysplasia
Gastric dysplasia
Gastrointestinal dysplasia
Gastrointestinal polyp
Gastrointestinal polyp
Gastrointestinal polyp
Gastrointestinal polyp
Gastrointestinal polyp
Gastrointestinal polyp
Intestinal polyp
Intestinal polyp
Intestinal polyp
Intestinal polyp
Intestinal cyst
Intestinal polyp
Intestinal polyp
Intestinal cyst
Intestinal polyp
Intestinal polyp
Intestinal polyp
Intestinal polyp
Intestinal polyp
Intestinal dysplasia
Malignant dysplasia
Malignant gastrointestinal obstruction
Mesenteric cyst
Mouth cyst
Oesophageal polyp
Palatal polyp
Palatal polyp
Palatal polyp
Palatal polyp
Parceatic cyst
Precancerous lesion of digestive tract
Precancerous lesion of digestive tract Rectal dysplasia
Rectal polyp
Retroperitoneum cyst
Salivary gland cyst
Salivary gland induration
Small intestine polyp
Terminal ileitis Tongue polyp Administration site cyst Application site cyst Infusion site cyst Injection site cyst 5q minus syndrome Tongue cyst Tongue dysplasia

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final / |
|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 121 of 229 |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | |
| Tro-dofined Mediber | し しょうしょうしょう しょうしょう しょう | | | | |

Novo Nordisk

Neoplasm

Abdominal wall neoplasm malignant
Actinar cell carcinoma of pancreas
Actinar cell carcinoma of pancreas
Actinic cell carcinoma of salivary gland
Acral lentiginous melanoma stage II
Acral lentiginous melanoma stage II
Acral lentiginous melanoma stage III
Acral lentiginous melanoma stage III
Acral lentiginous melanoma stage III
Acral lentiginous melanoma stage III
Acral lentiginous melanoma stage IV
Acute biphenotypic leukaemia
Acute leukaemia
Acute leukaemia in remission
Acute lymphocytic leukaemia (in remission)
Acute lymphocytic leukaemia refractory
Acute megakaryocytic leukaemia
Acute monocytic leukaemia (in remission)
Acute monocytic leukaemia (in remission)
Acute myeloid leukaemia (in remission)
Acute myeloid leukaemia (in remission)
Acute myeloid leukaemia (in remission)
Acute myeloid leukaemia refractory
Acute myeloid leukaemia concurent
Acute myeloid leukaemia refractory
Acute myeloid leukaemia of neukaemia
Acute myeloid satiacemia acturent
Acute myeloid satiacemia acturent
Acute myeloid satiacemia Acute myeloid sativary gland
Adenocarcinoma of appendix
Adenocarcinoma of salivary gland
Adenocarcinoma of the cervix
Adenocarcinoma of the cervix
Adenocarcinoma of salivary gland
Adenocarcinoma of salivary gland
Adenocarcinoma carcinoma of the cervix
Adenocarcinoma carcinoma of vagina
Adenosquamous carcinoma of vagina
Adenosquamous cell lung cancer recurrent
Adenosquamous cell lung cancer

04 December 2020 | Status: 1.0 Page: Version: Date: Clinical Trial Report NN9535-4506 NN9535

Final Novo Nordisk


Pre-defined MedDRA search - list of preferred terms

Preferred term Pre-defined MedDRA search

Neoplasm

Anal cancer stage 0
Anal cancer stage I
Anal cancer stage II
Anal cancer stage III
Anal cancer stage IV
Anal cancer stage IV
Anal squamous cell carcinoma
Anaplastic astrocytoma
Anaplastic large cell lymphoma T- and null-cell types refractory
Anaplastic large cell lymphoma T- and null-cell
types stage I
Anaplastic large cell lymphoma T- and null-cell
types stage II Anaplastic large cell lymphoma T- and null-cell Adenosquamous cell lung cancer stage 0
Adenosquamous cell lung cancer stage II
Adenosquamous cell lung cancer stage III
Adenosquamous cell lung cancer stage III
Adenosquamous cell lung cancer stage III
Adrenal gland cancer metastatic
Adrenal gland cancer metastatic
Adrenal gland cancer metastatic
Adrenocutical carcinoma
Adult T-cell lymphoma/leukaemia recurrent
Adult T-cell lymphoma/leukaemia stage II
Adult T-cell lymphoma/leukaemia stage II
Adult T-cell lymphoma/leukaemia stage II
Adult T-cell lymphoma/leukaemia stage II
Adult T-cell lymphoma/leukaemia stage II
Adult T-cell lymphoma/leukaemia stage III
Adult T-cell lymphoma/leukaemia stage III
Adult T-cell lymphoma/leukaemia stage III
Adult T-cell lymphoma/leukaemia stage III
Acthesioneuroblastoma Aleukaemic leukaemia Alveolar rhabdomyosarcoma Alveolar soft part sarcoma Alveolar soft part sarcoma metastatic Alveolar soft part sarcoma recurrent Ameloblastic carcinoma Anal cancer metastatic Anal cancer recurrent Anal cancer types

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final / |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 123 of 229 |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | |
| dysees Manham hearited | Drafarrad + | | | | |

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Neoplasm

Anaplastic large cell lymphoma T-

Anaplastic large cell lymphoma T- and null-cell types stage III
Anaplastic large cell lymphoma T- and null-cell types stage IV
Anaplastic large-cell lymphoma Anaplastic meningioma
Anaplastic chycid cancer
Anaplastic thyrioid cancer
Anaplastic thyrioid cancer
Angiocentric lymphoma recurrent
Angiocentric lymphoma recurrent
Angiocentric lymphoma stage II
Angiocentric lymphoma stage III
Angiocentric lymphoma stage II
Angiocentric lymphoma stage III
Angiocentric lymphoma stage III
Angioimmunoblastic T-cell lymphoma stage II
Angioimmunoblastic T-cell lymphoma stage II
Angioimmunoblastic T-cell lymphoma stage II
Angiosarcoma metastatic
Angiosarcoma metastatic
Angiosarcoma metastatic
Angiosarcoma recurrent
Angiosarcoma recurrent
Angiosarcoma analignant
Appendix cancer
Appendix cancer
Appendix cancer
Astrocytoma
Astrocy

Final Novo Nordisk 124 of 229 04 December 2020 | Status: 1.0 | Page: Version: Preferred term | Clinical Trial Report Pre-defined MedDRA search - list of preferred terms Pre-defined MedDRA search NN9535-4506 NN9535

Neoplasm

B-cell small lymphocytic lymphoma refractory
B-cell small lymphocytic lymphoma stage I
B-cell small lymphocytic lymphoma stage II
B-cell small lymphocytic lymphoma stage II
B-cell small lymphocytic lymphoma stage III
B-cell unclassifiable lymphoma high grade
B-cell unclassifiable lymphoma high grade
B-cell unclassifiable lymphoma high grade
B-cell unclassifiable lymphoma high grade
B-cell unclassifiable lymphoma of grade
B-cell unclassifiable lymphoma of grade
B-cell unclassifiable lymphoma stage IV
B-cell carcinoma
B-cell carcinoma stage II
B-cell carcinoma stage III
B-cell cancer recurrent
B-cell cancer stage IV
B-cell cancer stage III
B-cell

| NN9535 | Clinical Trial Report | Date: 04 Dece | December 2020 | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: 125 | 25 of 229 |

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Preferred term

Neoplasm

Pre-defined MedDRA search

Bladder squamous cell carcinoma stage II
Bladder squamous cell carcinoma stage III
Bladder squamous cell carcinoma stage III
Bladder transitional cell carcinoma stage III
Bladder transitional cell carcinoma stage III
Bladder transitional cell carcinoma stage 0
Bladder transitional cell carcinoma stage II
Bladder transitional cell carcinoma stage II
Bladder transitional cell carcinoma stage II
Bladder transitional cell carcinoma stage II
Bladder transitional cell carcinoma stage III
Bladder transitional cell carcinoma stage III
Bladder transitional cell carcinoma stage IV
Blast crisis in myelogenous leukaemia
Blast crisis in myelogenous leukaemia
Bone cancer metastatic
Bone marrow leukaemic cell infiltration
Bone marrow tumour cell infiltration
Bone sarcoma
Bone sarcoma
Brain neoplasm malignant
Brain neoplasm malignant
Brain stem glioma
Breast angiosarcoma metastatic
Brast cancer female
Breast cancer metastatic
Breast cancer metastatic
Breast cancer textege II
Breast cancer stage II
Breast cancer stage III
Breast sarcoma
Breast sarcoma metastatic

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | <u> </u> | v ersion: | 0.1 | rage: | 170 01 776 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Carcer in remission
Carcinoid tumour of the appendix
Carcinoid tumour of the caecum
Carcinoid tumour of the duodenum
Carcinoid tumour of the gastrointestinal tract
Carcinoid tumour of the parcinoid tumour of the parcinoid tumour of the parcinoid cumour of the parcinoid tumour of the parcinoid tumour of the small bowel
Carcinoid tumour of the small bowel
Carcinoid tumour of the stomach
Carcinoid tumour of the stomach
Carcinoid tumour pulmonary
Carcinoma in situ of the stomach
Carcinoma in situ of eye
Carcinoma in situ of penis
Carcinoma in situ of penis
Carcinoma in situ of faxin
Carcinoma in situ of faxin
Carcinoma in situ of faxin
Carcinoma in situ of skin
Carcinoma in situ of skin Bronchial carcinoma
Bronchioloalveolar carcinoma
Burkitt's leukaemia
Burkitt's lymphoma
Burkitt's lymphoma recurrent
Burkitt's lymphoma refractory
Burkitt's lymphoma stage I
Burkitt's lymphoma stage II
Burkitt's lymphoma stage II
Burkitt's lymphoma stage II
Burkitt's lymphoma stage II
CNS Germinoma Cervix carcinoma recurrent Cervix carcinoma stage 0 Cervix carcinoma stage I Cervix carcinoma stage II Cervix carcinoma stage II

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 127 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Cervix carcinoma stage IV

Chloroma

Chloroma

Choloroma

Choloroma (in remission)

Cholangiocarcinoma

Chondrosarcoma metastatic

Chondrosarcoma metastatic

Chordrosarcoma metastatic

Chordrocarcinoma

Chordrocarcinoma

Chorid melanoma

Choroid plaxus carcinoma

Chronic laukaemia in remission)

Chronic laukaemia in remission)

Chronic lymphocytic leukaemia refractory

Chronic lymphocytic leukaemia stage 1

Chronic lymphocytic leukaemia stage 1

Chronic lymphocytic leukaemia stage 2

Chronic lymphocytic leukaemia stage 3

Chronic lymphocytic leukaemia stage 3

Chronic lymphocytic leukaemia stage 3

Chronic lymphocytic leukaemia stage 3

Chronic lymphocytic leukaemia stage 4

Chronic lymphocytic leukaemia stage 3

Chronic lymphocytic leukaemia stage 3

Chronic myeloid leukaemia choroic myeloid leukaemia choroic myeloid leukaemia choroic myeloid leukaemia coursent

Chronic myeloid leukaemia recurrent

Chronic myeloid leukaemia coursent

Clear cell sarcoma of the kidney

Colon cancer stage I

Colon cancer stage I

Colon cancer stage II

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 128 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | 1 1 |

Colon cancer stage III
Colorectal adenocarcinoma
Colorectal cancer metastatic
Colorectal cancer metastatic
Colorectal cancer stage II
Colorectal cancer stage II
Colorectal cancer stage III
Colorectal cancer stage III
Colorectal cancer stage III
Colorectal cancer stage III
Colorectal cancer stage III
Colorectal cancer stage III
Colorectal cancer stage III
Colorectal cancer stage IV
Colorectal cancer stage III
Colorectal cancer stage IV
Colorectal cancer stage III
Colorectal cancer stage III
Colorectal cancer stage III
Colorectal cancer stage III
Colorectal cancer stage IV
Congenital malignant neoplasm
Conjunctival melanoma
Conjunctival melanoma
Conjunctival melanoma
Coliumeous T-cell lymphoma stage II
Cutaneous T-cell lymphoma stage II
Cutaneous T-cell lymphoma stage III
Cutaneous I-cell lymphoma stage III
Cutaneous I-cell lymphoma stage III
Cutaneous I-cell lymphoma ovary
Cystadenocarcinoma pancreas
Defiferentiated liposarcoma
Dermatofibrosarcoma protuberans
Desmoplastic mesothelioma
Desmoplastic mesothelioma
Desmoplastic mesothelioma
Desmoplastic mesothelioma
Diffuse large B-cell lymphoma refractory
Diffuse large B-cell lymphoma stage III
Diffuse large B-cell lymphoma stage III
Diffuse large B-cell lymphoma stage III
Diffuse large B-cell lymphoma stage III
Diffuse large B-cell lymphoma stage III
Diffuse large B-cell lymphoma
Dutal adenocarcinoma of pancreas
Bar neoplasm malignant

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 129 of 229 |
| Pre-defined MedDRA search - list of prefer | f preferred terms | | | | |
| יייים מסתאיין סאר באסר סאר שאר סאר שאר סאר שאר סאר | 70<br>4 20<br>4 20<br>5 | | | | |

Novo Nordisk

Neoplasm

Eccrine carcinoma
Embryonal rhabdomyosarcoma
Embryonal rhabdomyosarcoma
Endocrine neoplasm malignant
Endometrial cancer metastatic
Endometrial cancer stage I
Endometrial cancer stage I
Endometrial cancer stage II
Endometrial cancer stage II
Endometrial cancer stage II
Endometrial cancer stage II
Endometrial cancer stage II
Endometrial sarcoma metastatic
Endometrial sarcoma metastatic
Endometrial sarcoma metastatic
Entorphilo: leukaemia sarcoma recurrent
Epidodyman analignant
Epithelioid sarcoma metastatic
Epithelioid sarcoma metastatic
Epithelioid sarcoma metastatic
Epithelioid sarcoma metastatic
Epithelioid sarcoma metastatic
Epithelioid sarcoma metastatic
Extra-osseous Ewing's sarcoma metastatic
Extra

| 79535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|
| 19535-4506 | 1 | Version: | 1.0 Page: | 130 of 229 | |

Preferred term pre Pre-defined MedDRA search

Neoplasm

Extragonadal primary malignant teratoma
Extragonadal primary non-seminoma
Extragonadal primary non-seminoma stage II
Extragonadal primary non-seminoma stage II
Extragonadal primary non-seminoma stage III
Extragonadal primary seminoma (pure)
Extragonadal primary seminoma (pure)
Extragonadal primary seminoma (pure) stage II
Extramammary Paget's disease
Extramodal marginal zone B-cell lymphoma (BALT Extragonadal primary germ cell tumour mixed stage (MALT type) Extranodal marginal zone B-cell lymphoma (MALT (MALT (MALT (MALT (MALT (MALT type) recurrent
Extranodal marginal zone B-cell lymphoma
type) refractory
Extranodal marginal zone B-cell lymphoma type) stage II Extranodal marginal zone B-cell lymphoma type) stage III Extranodal marginal zone B-cell lymphoma type) Extranodal marginal zone B-cell lymphoma type) stage I Extranodal marginal zone B-cell lymphoma Extraskeletal chondrosarcoma metastatic Extraskeletal chondrosarcoma recurrent Extraskeletal myxoid chondrosarcoma Extraskeletal osteosarcoma metastatic Extraskeletal osteosarcoma metastatic Extraskeletal osteosarcoma recurrent Fallopian tube cancer metastatic Fallopian tube cancer stage I Fallopian tube cancer stage II Fallopian tube cancer stage II Fallopian tube cancer stage III Fallopian tube cancer stage IV type) stage IV Extraocular retinoblastoma

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | | Novo Nordisk |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 Page: | 131 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | |

Neoplasm

Pre-defined MedDRA search

Familial medullary thyroid cancer
Female reproductive tract carcinoma in situ
Fibrosarcoma
Fibrosarcoma
Fibrosarcoma
Fibrosarcoma
Fibrosarcoma
Fibrosarcoma
Fibrosarcoma
Fibrosarcoma
Follicle centre lymphoma diffuse small cell
lymphoma recurrent
Follicle centre lymphoma diffuse small cell
lymphoma stage I
Follicle centre lymphoma diffuse small cell
lymphoma stage II
Follicle centre lymphoma diffuse small cell
lymphoma stage II
Follicle centre lymphoma diffuse small cell
lymphoma stage II
Follicle centre lymphoma, follicular grade I, II,
III recurrent
Follicle centre lymphoma, follicular grade I, II,
III refractory
Follicle centre lymphoma, follicular grade I, II,
III refractory
Follicle centre lymphoma, follicular grade I, II,
III stage II
Follicle centre lymphoma follicular grade I, II,
III stage II
Follicle centre lymphoma follicular grade I, II,
III stage II
Follicle centre lymphoma, follicular grade I, II,
III stage II
Follicle centre lymphoma, follicular grade I, II,
III stage II
Follicle centre lymphoma follicular grade I, II,
II

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 132 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Dre-defined Medines | りなったのかながら | | | | | |

Gallbladder cancer stage IV
Gallbladder squamous cell carcinoma
Ganglioglioma
Ganglioplioma
Ganglioplioma
Gastric cancer stage I
Gastric cancer stage II
Gastric cancer stage II
Gastric cancer stage II
Gastric cancer stage II
Gastric cancer stage IV
Gastric cancer stage IV
Gastric cancer stage IV
Gastrioner malignant
Gastrointestinal adenocarcinoma
Gastrointestinal acancer metastatic
Gastrointestinal lymphoma
Gastrointestinal melanoma
Gastrointestinal melanoma
Gastrointestinal stromal tumour
Gastrointestinal melanoma
Gastrointestinal melanoma
Gastrointestinal melanoma
Gastrointestinal melanoma
Gastrointestinal stromal tumour
Gastrointestinal melanoma
Gastrointestinal trophoblastic tumour
Genital cancer male
Genital cancer male
Genital cancer metastatic
Genital cancer melanoma
Germ cell cancer metastatic
Gestational trophoblastic tumour
Glioblastoma
Glioblastoma
Gliomatosis cerebri
Gliomatosis cerebri
Gliomatosis cerebri
Gliomatosis carcinoma
Gloutis carcinoma
Gloutis carcinoma
HERZ positive breast cancer

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | 133 |
|---|---|---|---|---|---|
| NN9535-4506 | - | Version: | 1.0 Page: | Page: | |
| Pre-defined MedDRA search - list of | preferred terms | | | | |

Final Novo Nordisk

Neoplasm

Pre-defined MedDRA search

HER2 positive gastric cancer Haemangiopericytoma of meninges Haemangiopericytoma of meninges Haemangiopericytoma of meninges Haemangiopericytoma of meninges Haemangiopericytoma of Haemangiopericytoma of Haemangiopericytoma of Haemangiopericytoma of Hairy cell leukaemia recurrent Head and neck cancer stage II High grade B-cell lymphoma Burkitt-like lymphoma reflactory becall lymphoma Burkitt-like lymphoma stage II High grade B-cell lymphoma Burkitt-like lymphoma stage II High grade B-cell lymphoma Burkitt-like lymphoma stage II High grade B-cell lymphoma Burkitt-like lymphoma stage II High grade B-cell lymphoma Burkitt-like lymphoma stage II High grade B-cell lymphoma burkitt-like lymphoma stage II High grade B-cell lymphoma burkitt-like lymphoma stage II High grade B-cell lymphoma burkitt-like lymphoma stage II High grade B-cell lymphocyte depletion stage II subclocytic sarcoma Hodgkin's disease lymphocyte depletion stage II subcadiaphragm Hodgkin's disease lymphocyte depletion stage II subcadiaphragm Hodgkin's disease lymphocyte depletion stage II subcadiaphragm Hodgkin's disease lymphocyte depletion stage II subcadiaphragm Hodgkin's disease lymphocyte depletion stage II subcadiaphragm Hodgkin's disease lymphocyte depletion stage II subcabiaphragm

| NN9535<br>NN9535-4506 | Clinical Trial Report<br> - | Date:<br>Version: | 04 December 2020 Status: 1.0 Page: | 1 | Final 34 of 229 | Final <b>Novo Nordisk</b><br>f 229 |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Hodgkin's disease lymphocyte depletion stage II supradiaphragm lymphocyte depletion type recurrent Hodgkin's disease lymphocyte depletion type stage II digkin's disease lymphocyte depletion type stage IV site unspecified lymphocyte depletion type stage I site unspecified lymphocyte predominance stage I subdiaphragm lymphocyte predominance stage I subdiaphragm lymphocyte predominance stage I subdiaphragm lymphocyte predominance stage I subdiaphragm lymphocyte predominance stage I subdiaphragm lymphocyte predominance stage II site unspecified lymphocyte predominance stage II subdiaphragm lymphocyte predominance type refractory disease lymphocyte predominance type refractory disease lymphocyte predominance type refractory disease lymphocyte predominance type refractory disease lymphocyte predominance type stage II subcaphragm lymphocyte predominance type stage II disease mixed cellularity recurrent Hodgkin's disease mixed cellularity stage I site unspecified Hodgkin's disease mixed cellularity stage I site Hodgkin's disease mixed cellularity stage I site unspecified Hodgkin's disease mixed cellularity stage I site Hodgkin's disease mixed cellularity stage I site Hodgkin's disease mixed cellularity stage I site

| NN9535 | Clinical Trial Report | Date: 0 | 34 December 2020 Status: | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 135 of 229 |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | |

Novo Nordisk

Neoplasm

Augykin's disease mixed cellularity stage III Hodgkin's disease mixed cellularity stage III Hodgkin's disease mixed cellularity stage IV wingspecified Hodgkin's disease nodular sclerosis recurrent Hodgkin's disease nodular sclerosis refractory Hodgkin's disease nodular sclerosis stage II Hodgkin's disease nodular sclerosis stage II Hodgkin's disease nodular sclerosis stage II Hodgkin's disease nodular sclerosis stage II Hodgkin's disease nodular sclerosis stage IV Hodgkin's disease refractory Hodgkin's disease refractory Hodgkin's disease stage II Hodgkin's disease stage IV Hodgkin's disease unclassifiable Hormone receptor positive breast cancer Hodgkin's disease mixed cellularity stage II subdiaphragmatic Hodgkin's disease mixed cellularity stage II Hypopharyngeal cancer stage II Hypopharyngeal cancer stage III Hypopharyngeal cancer stage IV Hypopharyngeal cancer stage IV associated Kaposi's sarcoma Inflammatory carcinoma of breast recurrent Inflammatory carcinoma of breast stage III Inflammatory carcinoma of breast stage IV Inflammatory carcinoma of the breast INflammatory malignant fibrous histocytoma Inflammatory myofibroblastic tumour Hormone-refractory prostate cancer
Huerthle cell carcinoma
Hypopharyngeal cancer
Hypopharyngeal cancer recurrent
Hypopharyngeal cancer stage 0
Hypopharyngeal cancer stage 1 Hormone-dependent prostate cancer Hormone refractory breast cancer Immunoblastic lymphoma supradiaphragmatic

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 136 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |
| | 4 | | | | | ı |

Preferred term Pre-defined MedDRA search Neoplasm

Intestinal T-cell lymphoma recurrent
Intestinal T-cell lymphoma refractory
Intestinal T-cell lymphoma stage I
Intestinal T-cell lymphoma stage II
Intestinal T-cell lymphoma stage III
Intestinal T-cell lymphoma stage IV
Intestinal denocarcinoma
Intestinal metastasis
Intracranial germ cell tumour
Intraductal papillary breast neoplasm
Intraductal papillary breast neoplasm Intraductal proliferative breast lesion
Intraocular melanoma
Invasive breast carcinoma
Invasive ductal breast carcinoma
Invasive popillary breast carcinoma
Invasive papillary breast carcinoma
Invasive papillary breast carcinoma
Invasive papillary breast carcinoma
Invasive papillary breast carcinoma of

Reratoacanthoma
Langerhans cell sarcoma
Large cell lung cancer metastatic
Large cell lung cancer metastatic
Large cell lung cancer recurrent
Large cell lung cancer stage 0
Large cell lung cancer stage I
Large cell lung cancer stage II
Large cell lung cancer stage II
Large cell lung cancer stage IV

Laryngeal cancer metastatic Laryngeal cancer recurrent Laryngeal cancer stage 0 Laryngeal cancer stage II Laryngeal cancer stage II Laryngeal cancer stage III

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 137 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Laryngeal cancer stage IV
Laryngeal squamous cell carcinoma
Leiomyosarcoma
Leiomyosarcoma metastatic
Leiomyosarcoma recurrent
Lentigo maligna
Lentigo maligna
Lentigo maligna stage II
Leutaemic infiltration pulmonary
Leutaemic infiltration pulmonary
Leutaemic infiltration renal
Leutaemic infiltration renal
Leutaemic infiltration renal
Leutaemic infiltration renal
Leutaemic Iymphoma
Leutaemic Iymphoma
Leutaemic Iymphoma
Leutaemic Infiltration renal
Leutaemic Infiltration
Leutaemic Infiltr

04 December 2020 | Status: 1.0 Page: Version: Date: | Clinical Trial Report NN9535-4506 NN9535

Final Novo Nordisk


Preferred term Pre-defined MedDRA search - list of preferred terms Pre-defined MedDRA search

Neoplasm

Lymphoma transformation Lymphoplasmacytoid lymphoma/immunocytoma Lymphoplasmacytoid lymphoma/immunocytoma recurrent Lymphoplasmacytoid lymphoma/immunocytoma Lung adenocarcinoma stage II

Lung adenocarcinoma stage III

Lung adenocarcinoma stage IV

Lung carcinoma cell type unspecified stage I

Lung carcinoma cell type unspecified stage I

Lung carcinoma cell type unspecified stage I

Lung carcinoma cell type unspecified stage II

Lung carcinoma cell type unspecified stage II

Lung carcinoma cell type unspecified stage II

Lung carcinoma cell type unspecified stage II

Lung carcinoma cell type unspecified stage II

Lung sacinoma cell type unspecified stage II

Lung squamous cell carcinoma metastatic

Lung squamous cell carcinoma stage I

Lung squamous cell carcinoma stage I

Lung squamous cell carcinoma stage II

Lung squamous cell carcinoma stage II

Lung squamous cell carcinoma stage II

Lung squamous cell carcinoma stage II

Lung squamous cell carcinoma stage III

Lung squamous cell carcinoma stage III

Lung squamous cell carcinoma stage III

Lung squamous cell carcinoma stage III

Lung squamous cell carcinoma stage III

Lung squamous cell carcinoma stage III

Lung squamous cell carcinoma stage III

Lung squamous cell carcinoma stage IV Lymphangiosarcoma Lymphangiosis carcinomatosa Lymphocytic leukaemia Lymphocytic lymphoma Lymphoid leukaemia (in remission) Lobular breast carcinoma in situ Lung adenocarcinoma Lung adenocarcinoma recurrent Lung adenocarcinoma stage 0
Lung adenocarcinoma stage I
Lung adenocarcinoma stage II
Lung adenocarcinoma stage III
Lung adenocarcinoma stage III ymphoma AIDS related ymphoma

Lymphoplasmacytoid lymphoma/immunocytoma stage I Lymphoplasmacytoid lymphoma/immunocytoma stage II Lymphoplasmacytoid lymphoma/immunocytoma stage II Lymphoplasmacytoid lymphoma/immunocytoma stage III Lymphoplasmacytoid lymphoma/immunocytoma stage IV Malignant anorectal neoplasm Malignant blue naevus Malignant connective tissue neoplasm

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| 000+-000 | <u> </u> | v cision. | 0.1 | rage. | 139 01 773 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | 1 1 |

Malignant cranial nerve neoplasm
Malignant fibrous histiocytoma metastatic
Malignant fibrous histiocytoma of bone
Malignant fibrous histiocytoma of bone
Malignant fibrous histiocytoma recurrent
Malignant genitourinary tract neoplasm
Malignant glint cell fibrous histiocytoma
Malignant paemangiopericytoma metastatic
Malignant haemangiopericytoma recurrent
Malignant haemangiopericytoma recurrent
Malignant haemangiopericytoma recurrent
Malignant hymphoid neoplasm
Malignant hymphoid neoplasm
Malignant hymphoid neoplasm
Malignant mediastinal neoplasm
Malignant mediastinal neoplasm
Malignant melanoma of eyelid
Malignant melanoma stage II
Malignant mesenchymoma metastatic
Malignant mesenchymoma metastatic
Malignant mesenchymoma recurrent
Malignant mesenchymoma metastatic
Malignant mesenchymoma recurrent
Malignant mesenchymoma recurrent
Malignant mesenchymoma recurrent
Malignant mesenchymoma metastatic
Malignant mesenchymoma recurrent
Malignant mesenchymoma recurrent
Malignant mesenchymoma metastatic
Malignant mesenchymoma
Malignant neoplasm of contea
Malignant neoplasm of contea
Malignant neoplasm of sevelid
Malignant neoplasm of sislets of Langerhans
Malignant neoplasm of lacrimal duct
Malignant neoplasm of lacrimal duct

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 140 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I I |

Malignant neoplasm of orbit
Malignant neoplasm of paraurethral glands
Malignant neoplasm of pleura
Malignant neoplasm of pleura metastatic
Malignant neoplasm of reinal
Malignant neoplasm of seminal vesicle
Malignant neoplasm of seminal vesicle
Malignant neoplasm of spinal cord
Malignant neoplasm of thorax
Malignant neoplasm of thorax
Malignant neoplasm of uterine adnexa
Malignant neoplasm of uterine adnexa
Malignant neoplasm of uterine adnexa
Malignant neoplasm of uterine adnexa
Malignant neoplasm of uterine adnexa
Malignant neoplasm system neoplasm
Malignant neoplasm papilla of Vater
Malignant neoplasm poplasm
Malignant nipple neoplasm
Malignant nipple neoplasm
Malignant plotonersolasm
Malignant plotonersolasm
Malignant pericardial neoplasm
Malignant pericardial neoplasm
Malignant polyp
Malignant polyp
Malignant polyp
Malignant sylenic neoplasm
Malignant transformation
Malignant transformation
Malignant urinary tract neoplasm
Malignant urinary tract neoplasm
Malignant urinary tract neoplasm
Malignant urinary tract neoplasm
Malignant urinary tract neoplasm
Malignant cell lymphoma stage II
Mantle cell lymphoma stage II
Mantle cell lymphoma stage II
Mantle cell lymphoma stage II
Mantle cell lymphoma stage II
Mantle cell lymphoma stage II
Marginal zone lymphoma refractory
Marginal zone lymphoma stage II
Marginal zone lymphoma stage II
Marginal zone lymphoma stage II

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo N |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | 1.0 Page: | 141 of 229 | |
| Pre-defined MedDRA search - list of preferred | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Nordisk

Neoplasm

Marginal zone lymphoma stage III
Marginal zone lymphoma stage IV
Marjolin's ulcer
Mastocytic leukaemia
Maternal cancer in pregnancy
Mature B-cell type acute leukaemia
Medullary carcinoma of breast
Medulloblastoma
Medulloblastoma recurrent
Medunoma recurrent central nervous system fallopian tube gallbladder gastrointestinal tract Metastases to bone marrow
Metastases to bone marrow
Metastases to abdominal wail
Metastases to abdominal cavity
Metastases to abdominal vall
Metastases to badominal wail
Metastases to badominal wail
Metastases to badominal wail
Metastases to bone
Metastases to bone
Metastases to bone
Metastases to bone
Metastases to bone
Metastases to bone
Metastases to bone
Metastases to bone
Metastases to bone marrow
Metastases to bone marrow
Metastases to central nervous syste to neck to nervous system to muscle to nasal sinuses lung lymph nodes chest wall diaphragm to meninges larynx liver kidney heart to mouth t t t t たり たり to けつ Metastases t Metastases t Metastases t Metastases t Metastases t Metastases t Metastases t Metastases

Metastases

| NN9535 | Clinical Trial Report | Date: 04 | December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | ı | Version: | 1.0 | Page: | 142 of 229 | |
| Pre-defined MedDRA search - list of preferrec | f preferred terms | | | | | |

Neoplasm

Pre-defined MedDRA search

o perineum
o peripheral nervous system
o peripheral vascular system
o peritoneum
o pharynx
o pituitary gland Metastases to uterus.
Metastases to vagina
Metastatis
Metastatic bronchial carcinoma
Metastatic carcinoma of the bladder
Metastatic choriocarcinoma
Metastatic gastric cancer
Metastatic galioma
Metastatic glucagonoma
Metastatic glucagonoma
Metastatic glucagonoma
Metastatic lymphoma o the mediastinum
o the respiratory system
o thorax
o thyroid
o tonsils
o trachea o rectum
co rectum
co reproductive organ
to retroperitoneum
to salivary gland
to skin
to skin
to spinal cord
s to spinal
s to spine
s to spleen
s to stomach
ss to testicle urinary tract oesophagus placenta pleura prostate rectum ovary pancreas pelvis penis t t 0 to to to t t to たり Metastases Metastases Metastases Metastases Metastases Metastases Metastasses Metastases t Metastases t Metastases t Metastases

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 143 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Metastatic malignant melanoma
Metastatic neoplasm
Metastatic nervous system neoplasm
Metastatic ocular melanoma
Metastatic coular melanoma
Metastatic salivary gland cancer
Metastatic salivary gland cancer
Metastatic uterine cancer
Metastatic uterine cancer
Minimal residual disease
Minimal residual disease
Mismatch repair cancer syndrome
Mixed adenoneurcendocrine carcinoma
Mixed-type liposarcoma of appendix
Mucinous breast carcinoma of appendix
Mucinous sedometrial carcinoma
Mucinous sedometrial carcinoma
Mucinous sedometrial carcinoma
Mucinous sedometrial carcinoma
Mucinous sedometrial carcinoma
Mucinous sedometrial carcinoma
Mucinous levasemia
Mucinous cystadenocarcinoma of salivary gland
Mucinous cystadenocarcinoma of salivary gland
Mucinous cystadenocarcinoma
Carcinoma
Myeloid leukaemia
Myeloid leukaemia
Myeloid leukaemia
Myeloid leukaemia in remission
Mysoloid leukaemia
Nasopharyngeal cancer metastatic
Nasopharyngeal cancer stage II

| status: | age: |
|-----------------------|-------------|
| 04 December 2020 | 1.0 |
| Clinical Trial Report | 1 |
| NN9535 | NN9535-4506 |

Final Novo Nordisk


Pre-defined MedDRA search - list of preferred terms

Preferred term

Neoplasm

Pre-defined MedDRA search

Neurofibrosarcoma metastatic
Neurofibrosarcoma metastatic
Neurofibrosarcoma recurrent
Nodal marginal zone B-cell lymphoma recurrent
Nodal marginal zone B-cell lymphoma refractory
Nodal marginal zone B-cell lymphoma stage I
Nodal marginal zone B-cell lymphoma stage I
Nodal marginal zone B-cell lymphoma stage II
Nodal marginal zone B-cell lymphoma stage II
Nodal marginal zone B-cell lymphoma stage II
Nodal marginal zone B-cell lymphoma stage IV
Nodal marginal zone B-cell lymphoma stage IV recurrent histology Neuroendocrine tumour of the lung metastatic aggressive Non-Hodgkin's lymphoma unspecified histology aggressive refractory
Non-Hodgkin's lymphoma unspecified histology
aggressive stage I
Non-Hodgkin's lymphoma unspecified histology
aggressive stage II Non-Hodgkin's lymphoma unspecified histology Neuroendocrine carcinoma of prostate Neuroendocrine carcinoma of the bladder Neuroendocrine carcinoma of the skin Neuroendocrine tumour Non-Hodgkin's lymphoma metastatic
Non-Hodgkin's lymphoma metastatic
Non-Hodgkin's lymphoma refractory
Non-Hodgkin's lymphoma stage II
Non-Hodgkin's lymphoma stage II
Non-Hodgkin's lymphoma stage II
Non-Hodgkin's lymphoma stage III
Non-Hodgkin's lymphoma stage IV
Non-Hodgkin's lymphoma transformed re
Non-Hodgkin's lymphoma transformed re Neuroendocrine carcinoma metastatic Neuroendocrine breast tumour Neuroendocrine carcinoma Neuroblastoma recurrent aggressive recurrent Nodular melanoma Nephroblastoma Neuroblastoma

| NN9535 | Clinical Trial Report | Date: 04 | 94 December 2020 Status: | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: 145 | 45 of 229 |
| Pre-defined MedDRA search - list of preferred | preferred terms | | | | |

Novo Nordisk

Neoplasm

Pre-defined MedDRA search

Non-Hodgkin's lymphoma unspecified histology aggressive stage III
Non-Hodgkin's lymphoma unspecified histology aggressive stage IV
Non-Hodgkin's lymphoma unspecified histology indolent stage IV
Non-Hodgkin's lymphoma unspecified histology indolent stage II
Non-Hodgkin's lymphoma unspecified histology indolent stage II
Non-Hodgkin's lymphoma unspecified histology indolent stage III
Non-manla cell ung cancer recurrent
Non-small cell lung cancer stage III
Ocsophageal adenocarcinoma stage III
Ocsophageal adenocarcinoma stage III
Ocsophageal adenocarcinoma stage III
Ocsophageal adenocarcinoma stage III
Ocsophageal carcinoma stage III
Ocsophageal adenocarcinoma stage III
Ocsophageal carcinoma stage III
Ocsopha

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 146 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Oesophageal squamous cell carcinoma metastatic Oesophageal squamous cell carcinoma recurrent Oesophageal squamous cell carcinoma stage 0 Oesophageal squamous cell carcinoma stage I Oesophageal squamous cell carcinoma stage II Oesophageal squamous cell carcinoma stage III Oesophageal squamous cell carcinoma stage IV Oligoastrocytoma Oligodendroglioma

Oral cavity cancer metastatic oropharyngeal cancer coropharyngeal cancer stage of oropharyngeal cancer stage I oropharyngeal cancer stage II oropharyngeal cancer stage II oropharyngeal cancer stage II oropharyngeal cancer stage II oropharyngeal lymphoepithelioma oropharyngeal squamous cell carcinoma osteosarcoma metastatic osteosarcoma recurrent

Optic glioma

Ovarian cancer metastatic
Ovarian cancer recurrent
Ovarian cancer stage II
Ovarian cancer stage III
Ovarian cancer stage IV Otic cancer metastatic Ovarian cancer

Ovarian clear cell carcinoma
Ovarian dysgerminoma stage I
Ovarian dysgerminoma stage III
Ovarian dysgerminoma stage III
Ovarian dysgerminoma stage IV
Ovarian dysgerminoma stage unspecified

Ovarian endometrioid carcinoma Ovarian epithelial cancer metastatic Ovarian epithelial cancer metastatic Ovarian epithelial cancer recurrent Ovarian epithelial cancer stage I Ovarian embryonal carcinoma

| NN9535 | Clinical Trial Report | Date: ( | 34 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 147 of 229 | |
| Pre-defined MedDRA search - list of preferred | preferred terms | | | | | |

Pre-defined MedDRA search

Preferred term

Neoplasm

Ovarian epithelial cancer stage II

Ovarian epithelial cancer stage III

Ovarian germ cell cancer stage IV

Ovarian germ cell cancer stage II

Ovarian germ cell cancer stage II

Ovarian germ cell cancer stage III

Ovarian germ cell cancer stage III

Ovarian germ cell cancer stage III

Ovarian germ cell choriocarcinoma stage II

Ovarian germ cell choriocarcinoma stage III

Ovarian germ cell choriocarcinoma stage III

Ovarian germ cell choriocarcinoma stage III

Ovarian germ cell embryonal carcinoma stage III

Ovarian germ cell endodermal sinus tumour stage III

Ovarian

Ovarian germ cell endodermal sinus tumour stage IV
Ovarian germ cell polyembryoma
Ovarian germ cell polyembryoma stage II
Ovarian germ cell polyembryoma stage III
Ovarian germ cell polyembryoma stage III
Ovarian germ cell polyembryoma stage IV
Ovarian germ cell teratoma
Ovarian germ cell teratoma
Ovarian germ cell teratoma stage II
Ovarian germ cell teratoma stage II
Ovarian germ cell teratoma stage II
Ovarian germ cell teratoma catage III
Ovarian germ cell teratoma catage IV
Ovarian germ cell teratoma catage IV
Ovarian germ cell teratoma catage IV
Ovarian germ cell teratoma catage IV
Ovarian germ cell teratoma cell tumour
Ovarian germ cell tumour mixed
Ovarian germ cell tumour mixed
Ovarian germ cell tumour mixed
Ovarian germ cell tumour mixed

Ovarian stromal cancer Paget's disease of nipple Paget's disease of penis Paget's disease of the vulva Pancoast's tumour Pancreatic carcinoma Ovarian melanoma
148 of 229 04 December 2020 Status: 1.0 Page: Version: | Clinical Trial Report NN9535-4506 NN9535

Final Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Neoplasm

Pre-defined MedDRA search

metastatic

Preferred term

Pericardial mesothelioma malignant
Pericardial mesothelioma malignant recurrent
Peripheral T-cell lymphoma unspecified
Peripheral T-cell lymphoma unspecified recurrent
Peripheral T-cell lymphoma unspecified recurrent Pancreatic carcinoma stage 0
Pancreatic carcinoma stage I
Pancreatic carcinoma stage II
Pancreatic carcinoma stage III
Pancreatic carcinoma stage III
Pancreatic carcinoma stage IV
Pancreatic neuroendocrine tumour
Pancreatic sarcoma
Pancreatoblastoma
Papillarv reassatic Papillary renal cell carcinoma
Papillary serous endometrial carcinoma
Papillary thyroid cancer
Paraganglion neoplasm malignant
Paranasal sinus and nasal cavity malignant neoplasm recurrent
Paranasal sinus and nasal cavity malignant
neoplasm stage 0
neoplasm stage 1
neoplasm stage I Paranasal sinus and nasal cavity malignant neoplasm stage  $\ensuremath{\mathrm{II}}$ Paranasal sinus and nasal cavity malignant neoplasm stage III Paranasal sinus and nasal cavity malignant neoplasm stage IV Paranasal sinus and nasal cavity malignant Penile squamous cell carcinoma Parathyroid tumour malignant Penis carcinoma metastatic Penis carcinoma recurrent Penis carcinoma stage I Penis carcinoma stage II Penis carcinoma stage III Penis carcinoma stage IV Pancreatic carcinoma m Pancreatic carcinoma r Pancreatic carcinoma s Pancreatic carcinoma s Penile cancer neoplasm

| | 14 | |
|--------------------------|-------------|-------------------------------------|
| 34 December 2020 Status: | 1.0 Page: | |
| 04 December | • • | |
| Date: | Version | |
| Clinical Trial Report | 1 | of preferred terms |
| NN9535 | NN9535-4506 | Pre-defined MedDRA search - list of |

Final Novo Nordisk


Neoplasm

Pre-defined MedDRA search

Peripheral T-cell lymphoma unspecified stage In Peripheral T-cell lymphoma unspecified stage IT Peripheral T-cell lymphoma unspecified stage IT Peripheral T-cell lymphoma unspecified stage IT Peripheral T-cell lymphoma unspecified stage IV Peripheral T-cell lymphoma unspecified stage IV Peripheral T-cell lymphoma of bone metastatic Peripheral neuroepithelioma of bone metastatic Peripheral primitive neuroectodermal bone tumour Peripheral primitive neuroectodermal bone tumour Peripheral primitive neuroectodermal bone tumour Peripheral primitive neuroectodermal tumour of soft tissue Peritoneal mesothelioma malignant recurrent Peritoneal mesothelioma malignant recurrent Pharyngeal cancer stage I Pharyngeal cancer stage II Pharyngeal cancer stage II Pharyngeal cancer stage IV Pharyngeal cancer metastatic Pharyngeal cancer metastatic Pharyngeal cancer stage IV Plumatrix carcinoma Pineal parenchymal neoplasm malignant recurrent Pineal barenchymal neoplasm malignant recurrent Plasma cell leukaemia in remission Plasma cell leukaemia Plasma cell myeloma recurrent Plasma cell myeloma relactory Plasmacollum plasma cell myeloma relactory Plasmacollum plasmacollum plasmacolum plasmacollum plasmacolum pl

04 December 2020 | Status: Version: Date: | Clinical Trial Report NN9535-4506 NN9535

Final Novo Nordisk


1.0 Page:

Pre-defined MedDRA search - list of preferred terms

Preferred term

Neoplasm

Pre-defined MedDRA search

Primary mediastinal large B-cell lymphoma stage I Primary mediastinal large B-cell lymphoma stage II Primary mediastinal large B-cell lymphoma stage Primary mediastinal large B-oell lymphoma stage IV Primary pulmonary melanoma Primitive neuroectodermal tumour Postcricoid cancer

Precursor B-lymphoblastic lymphoma recurrent
Precursor B-lymphoblastic lymphoma refractory
Precursor B-lymphoblastic lymphoma stage I
Precursor B-lymphoblastic lymphoma stage II
Precursor B-lymphoblastic lymphoma stage II
Precursor B-lymphoblastic lymphoma stage II
Precursor B-lymphoblastic lymphoma stage IV
Precursor I-lymphoblastic lymphoma stage IV
Precursor T-lymphoblastic leukaemia acute
Precursor T-lymphoblastic leukaemia Precursor T-lymphoblastic lymphoma/leukaemia stage I Precursor T-lymphoblastic lymphoma/leukaemia stage II Precursor T-lymphoblastic lymphoma/leukaemia stage IV
Primary breast lymphoma
Primary cardiac lymphoma
Primary effusion lymphoma
Primary gastrointestinal follicular lymphoma Precursor T-lymphoblastic lymphoma/leukaemia Precursor T-lymphoblastic lymphoma/leukaemia stage III Primary mediastinal large B-cell lymphoma Primary mediastinal large B-cell lymphoma recurrent Primary mediastinal large B-cell lymphoma refractory Pleural mesothelioma malignant recurrent Pleural sarcoma Poorly differentiated thyroid carcinoma Pleuropulmonary blastoma Porocarcinoma refractory recurrent

| NN9535<br>NN9535-4506 | Clinical Trial Report | Date:<br>Version: | 04 December 2020 Status:<br>1.0 Page: | Final<br>151 of 229 | Final Novo Nordisk<br>f 229 |
|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | I |

Primitive neuroectodermal tumour metastatic Prolymphocytic leukaemia Prostate cancer Prostate cancer metastatic Prostate cancer metastatic Prostate cancer stage 0 Prostate cancer stage I Prostate cancer stage II Prostate cancer stage IV

Pseudosarcoma

Queyrat erythroplasia
Rectal adenocarcinoma
Rectal cancer metastatic
Rectal cancer stage 0
Rectal cancer stage 11
Rectal cancer stage 11
Rectal cancer stage 11
Rectal cancer stage 11
Rectal cancer stage 11
Rectal cancer stage 11
Rectal cancer stage 11
Rectosigmoid cancer metastatic
Rectosigmoid cancer metastatic
Rectosigmoid cancer stage 0
Rectosigmoid cancer stage 1
Rectosigmoid cancer stage 1
Rectosigmoid cancer stage 1
Rectosigmoid cancer stage 11

Renal cancer Renal cancer Renal cancer Renal cancer Senal cancer Senal cancer Senal cancer Senal cell car Renal cell car

cancer metastatic
cancer recurrent
cancer stage I
cancer stage II
cancer stage III
cancer stage IV
call carcinoma
cell carcinoma stage II
cell carcinoma stage II

| Final Novo Nordisk<br>152 of 229 | |
|---|---|
| December 2020 Status:<br>1.0 Page: | |
| Date: 04 | |
| Clinical Trial Report | of preferred terms |
| NN9535<br>NN9535-4506 | Pre-defined MedDRA search - list of preferred terms |

Neoplasm

Pre-defined MedDRA search

Renal cell carcinoma stage IV
Respiratory tract carcinoma in situ
Retinal melaanoma
Retinoblastoma
Retroperitoneal cancer
Retroperitoneal neoplasm metastatic
Rhabdooid tumour
Rhabdooid tumour
Rhabdomyosarcoma
Rhabdomyosarcoma
Richter's syndrome
Round cell liposarcoma
Salivary gland cancer recurrent
Richter's syndrome
Round call liposarcoma
Salivary gland cancer stage II
Salivary gland cancer metastatic
Sarcoma of skin
Sarcomatoid carcinoma
Sarcomatoid mesothelioma
Sarcomatoid mesothelioma
Sarcomatoid carcinoma
Sarcomatoid mesothelioma
Sarcomatoid mesothelioma
Sarcomatoid mesothelioma
Sarcomatoid carcinoma
Sarcomatoid mesothelioma
Sarcomatoid carcinoma
Sarcomatoid carcinoma
Serious cystadenocarcinoma
Serious cystadenocarcinoma
Sinus cancer metastatic
Skin cancer metastatic
Skin cancer metastatic
Skin squamous cell carcinoma
Skin squamous cell carcinoma
Skin squamous cell carcinoma
Small cell carcinoma
Small cell lung cancer
Small cell lung cancer
Small cell lung cancer
Small cell lung cancer

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 153 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | : preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | 1 1 |

Neoplasm Small o

Small cell lung cancer limited stage
Small cell lung cancer metastatic
Small cell lung cancer metastatic
Small intestine carcinoma
Small intestine carcinoma metastatic
Small intestine carcinoma stage I
Small intestine carcinoma stage II
Small intestine carcinoma stage II
Small intestine carcinoma stage II
Small intestine carcinoma stage II
Small intestine carcinoma stage II
Small intestine carcinoma stage II
Small intestine leiomyosarcoma
Soft tissue sarcoma
Solid pseudopapillary tumour of the pancreas
Spiral meningiona malignant
Spinal meningiona malignant
Spinal merginal zone lymphoma refractory
Splenic marginal zone lymphoma stage II
Squamous cell carcinoma of the barotid gland
Squamous cell carcinoma of the barotid gland
Squamous cell carcinoma of the valva
Squamous cell carcinoma

| NN9535<br>NN9535-4506 | Clinical Trial Report | Date: ( | 34 December 2020 Status:<br>1.0 Page: | Status:<br>Page: | Final<br>154 of 229 | Final <b>Novo Nordisk</b><br>f 229 |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | c of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Superficial spreading melanoma stage IV
Superficial spreading melanoma stage unspecified
Synovial sarcoma metastatic
Synovial sarcoma metastatic
Synovial sarcoma metastatic
Synovial sarcoma recurrent
T-cell chronic lymphocytic leukaemia
T-cell lymphoma recurrent
T-cell lymphoma stage II
T-cell unclassifiable lymphoma high grade
T-cell prolymphocytic leukaemia
T-cell unclassifiable lymphoma low grade
T-cell unclassifiable lymphoma stage II
T-cell unclassifiable lymphoma (pure) stage II
T-cell unclassifiable lymphoma (pure) stage II
T-cell unclassifiable lymphoma (pure) stage III
T-cell unc

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 S | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 155 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |

Neoplasm

Pre-defined MedDRA search

Testicular yolk sac tumour stage I
Testicular yolk sac tumour stage II
Testis cancer
Testis cancer
Testis cancer recurrent
Thymicat cancer
Thymoma malignant recurrent
Thymoma malignant recurrent
Thyroid cancer stage II
Thyroid cancer metastatic
Tongue carcinoma stage II
Tongue carcin

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 156 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | 1 1 |

Transitional cell carcinoma urethra
Trichoblastic carcinoma
Triple hostive breast cancer
Triple positive breast cancer
Triple positive breast cancer
Tubular breast carcinoma
Undifferentiated carcinoma
Undifferentiated carcinoma
Undifferentiated carcinoma
Undifferentiated carcinoma
Uncteric cancer
Uretric cancer metastatic
Uretric cancer requinal
Uretric cancer regional
Uretric cancer recurrent
Uretrial cancer metastatic
Uretrial cancer metastatic
Uretrial cancer metastatic
Uretrial cancer metastatic
Uretrial cancer metastatic
Uretrial cancer recurrent
Uretrial cancer recurrent
Uretrial cancer metastatic
Uretrial cancer metastatic
Uretrial cancer metastatic
Uretrial cancer metastatic
Uretrial cancer stage II
Uretrial cancer stage II
Uretrial cancer stage II
Uretrial cancer stage IV
Uredinal cancer stage IV
Uredinal cancer stage II
Uretrial cancer stage II
Uretrial cancer stage IV

| NN9535 | Clinical Trial Report | Date: ( | 34 December 2020 Status: | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: 1 | 157 of 229 |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | |

Novo Nordisk

Neoplasm

Vulvar adenocarcinoma

Vulvar basal cell carcinoma

Waldenstrom's macroglobulinaemia refractory
Waldenstrom's macroglobulinaemia stage I
Waldenstrom's macroglobulinaemia stage II
Waldenstrom's macroglobulinaemia stage II
Waldenstrom's macroglobulinaemia stage II
Waldenstrom's macroglobulinaemia stage III
Waldenstrom's macroglobulinaemia stage III
Waldenstrom's macroglobulinaemia stage IV
ACTH-producing pituitary tumour
APUDoma
Abdominal wall neoplasm
Abdominal wall neoplasm
Abdominal wall neoplasm
Acanthoma
Acanthoma
Acanthoma
Acanthoma
Acanthoma
Acanthoma
Acanthomial cyst
Acquired chromosomal abnormality
Acquired thalassaemia
Actorired thalassaemia
Adenoma benign
Adenoma benign
Adenoma benign
Adenoma benign
Adenoma theri cyst
Adrenal rest tumour of the testis
Adrenal cyst
Adrenal cyst
Adrenal cyst
Adrenal cyst
Adrenal cyst
Adrenal cyst
Adrenal cest umour of the testis
Adrenal cyst
Albha I foetoprotein abnormal
Albha interferon therapy
Albha interferon therapy
Albha interferon therapy
Albha interferon therapy
Albha interferon therapy
Albha interferon therapy
Ampliation of penis
Amyloidoma
Amyloidoma
Amal neoplasm

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 158 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | l |

Anal polypectomy Anaplastic lymphoma kinase gene and nucleophosmin gene fusion overexpression

Androgen therapy Aneurysmal bone cyst

Angiofibroma Angiogenesis biomarker increased

Angiolipoma Angiomyofibroblastoma Angiomyolipoma

Angiomyxome
Angiomyxome
Anogenital warts
Anorectal haemangioma
Anti-NWDA antibody positive
Anti-vGCC antibody positive
Antiandrogen withdrawal syndrome
Antiandrogen therapy
Antioestrogen therapy
Antioestrogen therapy
Anschnoid cyst
Arschnoid cyst
Arsenical keratosis
Aspiration bone marrow abnormal
Astroblastoma

Astrocyana and a grade
Atypical fibroxanthoma
Aural cystadenoma
Aural polyp
Autologous bone marrow transplantation therapy
Autologous bone marrow transplant transplant
Axillary lymphadenectomy
B-cell depletion therapy
Bannayan-Riley-Ruvalcaba syndrome
Bartholin's cyst
Basal cell naevus syndrome
Becker's naevus
Bendom anorectal neoplasm
Benign anorectal neoplasm
Benign bone neoplasm
Benign beas t neoplasm
Benign cardiac neoplasm
Benign cardiac neoplasm

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 159 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

on endocrine neoplasm

In fallopian tube neoplasm

In female reproductive tract neoplasm

In gastric neoplasm

In gastrointestinal neoplasm

In genitourinary tract neoplasm

In hydatidiform mole Benign connective tissue neoplasm
Benign duodenal neoplasm
Benign ear neoplasm
Benign fallopian tube neoplasm
Benign fallopian tube neoplasm
Benign gastroin explasm
Benign gastroin neoplasm
Benign gastroin neoplasm
Benign gastroin neoplasm
Benign gastroin neoplasm
Benign joint neoplasm
Benign lumg neoplasm
Benign male reproductive tract neoplasm
Benign male reproductive tract neoplasm
Benign male reproductive tract neoplasm
Benign mesenteric neoplasm
Benign mesenteric neoplasm
Benign mescheliam
Benign mescheliam
Benign mecolasm of adrenal gland
Benign neoplasm of adrenal gland
Benign neoplasm of cervix uteri
Benign neoplasm of conjunctiva
Benign neoplasm of conjunctiva
Benign neoplasm of conjunctiva
Benign neoplasm of conjunctiva
Benign neoplasm of conjunctiva
Benign neoplasm of conjunctiva
Benign neoplasm of conjunctiva
Benign neoplasm of islets of Langerhans
Benign neoplasm of islets of Langerhans
Benign neoplasm of lacrimal gland
Benign neoplasm of lacrimal gland
Benign neoplasm of lacrimal gland
Benign neoplasm of obtit
Benign neoplasm of obtit
Benign neoplasm of obtit
Benign neoplasm of obtit
Benign neoplasm of obtit
Benign neoplasm of obtit
Benign neoplasm of obtit
Benign neoplasm of obtit scrotum seminal vesicle spinal cord prostate neoplasm of neoplasm of neoplasm of neoplasm of neoplasm of neoplasm of

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 160 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | E preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I I |

Benign neoplasm of testis
Benign neoplasm of thymus
Benign neoplasm of thyroid gland
Benign neoplasm of uretra
Benign neoplasm of uretra
Benign neoplasm of uretra
Benign neoplasm of uretra
Benign neoplasm of uretra
Benign pancreatic neoplasm
Benign pericardium neoplasm
Benign pericardium neoplasm
Benign pericardium neoplasm
Benign pericardium neoplasm
Benign pleural neoplasm
Benign pleural neoplasm
Benign small intestinal neoplasm
Benign small intestinal neoplasm
Benign small intestinal neoplasm
Benign spleen tumour
Benign syleen tumour
Benign variatory tract neoplasm
Benign varial neoplasm
Biliary ovst
Biliary ovst
Biliary padenoma
Biliary padenoma
Biliary padenoma
Biliary padenomial wall abnormal
Biopsy artery abnormal
Biopsy artery abnormal
Biopsy bone marrow abnormal
Biopsy bone marrow abnormal
Biopsy bone marrow abnormal
Biopsy breast abnormal

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 161 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ! |

Biopsy bronchus abnormal
Biopsy cartilage abnormal
Biopsy chest wall abnormal
Biopsy chest wall abnormal
Biopsy chest wall abnormal
Biopsy conformative abnormal
Biopsy cornea abnormal
Biopsy cornea abnormal
Biopsy endometrium abnormal
Biopsy epididymis abnormal
Biopsy epididymis abnormal
Biopsy feetal abnormal
Biopsy feetal abnormal
Biopsy feetal abnormal
Biopsy fighted abnormal
Biopsy fighted abnormal
Biopsy ligament abnormal
Biopsy ligament abnormal
Biopsy ligament abnormal
Biopsy ligament abnormal
Biopsy ligament abnormal
Biopsy lung abnormal
Biopsy palate abnormal
Biopsy palate abnormal
Biopsy palate abnormal
Biopsy palate abnormal
Biopsy palate abnormal
Biopsy parathyroid gland abnormal
Biopsy parathyroid gland abnormal
Biopsy pericardium abnormal
Biopsy pericardium abnormal
Biopsy pericardium abnormal
Biopsy pharynx abnormal
Biopsy pripheral nerve abnormal
Biopsy pripheral nerve abnormal
Biopsy prostate abnormal
Biopsy prostate abnormal
Biopsy prostate abnormal Biopsy salivary gland abnormal Biopsy sclera abnormal Biopsy seminal vesicle abnormal Biopsy site unspecified abnormal Biopsy skin abnormal Biopsy prostate abnormal Biopsy rectum abnormal Biopsy retina abnormal

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 162 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | l I |

Biopsy small intestine abnormal
Biopsy spleen abnormal
Biopsy stomach abnormal
Biopsy tendon abnormal
Biopsy testes abnormal
Biopsy thyroid gland abnormal
Biopsy thyroid gland abnormal
Biopsy trachea abnormal
Biopsy trachea abnormal
Biopsy urethra abnormal
Biopsy uterus abnormal
Biopsy vagina abnormal
Biopsy varina abnormal
Biopsy vulva abnormal
Biopsy vulva abnormal
Biopsy vulva abnormal
Biopsy vulva abnormal
Biopsy vocal cord abnormal
Biopsy volva abnormal
Biopsy volva abnormal
Biopsy volva abnormal
Biopsy volva abnormal
Biopsy volva abnormal
Biopsy volva abnormal
Biopsy volva abnormal
Biopsy volva abnormal
Bladder Cyst
Bladder neoplasm
Bladder neoplasm
Bladder neoplasm
Bladder papilloma
Bladder polypectomy
Blast cell count increased
Blast cell proliferation
Blast cell proliferation
Blast cell proliferation
Blast cell proliferation
Blone giant cell tumour benign
Bone giant cell tumour benign
Bone marrow reticulin fibrosis
Bone marrow reticulin fibrosis
Bone marrow infiltration
Bone marrow infiltration
Bone marrow infiltration
Bone marrow reticulin seronary
Borderline worrian tumour
Bone bonderline serous tumour of ovary
Boneonid papulosis

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 163 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I I |

Brachytherapy to eye
Brachytherapy to penis
Brachytherapy to tongue
Brachytherapy to tongue
Brain neoplasm
Brain neoplasm
Brain scan abnormal
Brain stem glioma benign
Brain teratoma
Brain tratoma
Brain tumour operation
Brachtal cyst
Brack adenoma
Brack adenoma
Breast calcifications
Breast conserving surgery
Breast conserving surgery
Breast proliferative
Breast libroma
Breast fibroma
Breast fibroma
Breast fibroma
Breast tumour excision
Breast tumour excision
Breast tumour excision
Breast tumour excision
Breast tumour excision
Breast tumour excision
CD20 antigen positive
CD20 antigen positive
CD25 antigen positive
CD25 antigen positive
CD30 expression
CLOVES syndrome
CSF lymphocyte count abnormal
CSF lymphocyte count increased
Cachexia
Cancer fatigue
Cancer hormonal therapy
Cancer pain
Cancer staging
Cancer surgery
Cancer surgery

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 164 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Carbohydrate antigen 15-3 increased
Carbohydrate antigen 19-9 increased
Carbohydrate antigen 57-9 increased
Carbohydrate antigen 572-4
Carbohydrate antigen 72-4
Carbohydrate antigen 72-4
Carbohydrate antigen 72-4
Carbohydrate antigen 72-4
Carbohydrate antigen 72-4
Carbohydrate antigen 72-4
Carcinoembryonic antigen increased
Carcinoembryonic antigen increased
Carcinoembryonic antigen increased
Carcinoembryonic antigen increased
Carcinoembryonic antigen increased
Carcinoembryonic antigen increased
Carcinoid crisis
Carcinoid crisis
Carcinoid heart disease
Carcinoid heart disease
Carcinomatous polyarthritis
Carcinoid heart disease
Carcinomatous polyarthritis
Carcino Anguer increased
Carcino Carcinoma
Carcino Carcinoma
Carcino Carcinoma
Carcino Carcinoma
Carcino Carcinoma
Carcino Carcinoma
Carcino Carcinoma
Carcino Carcinoma
Carcinomatous fibroelastoma
Carcinomatous system dermoid tumour
Cerebellar tumour
Cerebellar tumour
Cerebellar tumour
Cerebellar tumour
Cerebellopontine angle tumour

| Novo Nordisk | I |
|-----------------------------|-----------------------------------------------|
| Final 165 of 229 | |
| Status:<br>Page: | |
| 04 December 2020<br>1.0 | |
| Date: | |
| Clinical Trial Report<br> - | f preferred terms |
| NN9535<br>NN9535-4506 | Pre-defined MedDRA search - list of preferred |

Neoplasm

Pre-defined MedDRA search

Cervix tumour excision
Cervix warts
Chemical peel of skin
Chemotherapy
Chemotherapy
Chemotherapy cardiotoxicity attenuation
Chemotherapy stravasation management
Chemotherapy wiltiple agents systemic
Chemotherapy woultiple agents systemic
Chemotherapy sensitivity and resistance assay
Chemotherapy single agent systemic
Chemotherapy single agent systemic
Chemotherapy single agent systemic
Chemotherapy toxicity attenuation
Chemotherapy toxicity attenuation
Chemotherapy toxicity attenuation
Chemotherapy wrothelial toxicity attenuation
Chest wall cyst
Chest wall cyst
Cholastion
Cholasteran
Cholasteran
Cholasteran
Cholasteran
Cholasteran
Cholesterin granuloma
Cholesterin granuloma
Cholesterin granuloma
Cholesterin granuloma
Chondroblastoma
Chondroblastoma
Choroid neoplasm
Choroid plexus papilloma
Choroid plexus papilloma
Choroid beannosinusitis with nasal polyps
Cloral evolution
Colectomy
Colon seeplasm
Colon seeplasm
Colon seeplasm
Colon seeplasm
Colon seeplasm
Colon peoplasm

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 166 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Congenital benign neoplasm
Congenital cerebral cyst
Congenital cerebral haemangioma
Congenital chroid plexus cyst
Congenital cyst
Congenital cyst
Congenital cyst
Congenital syst
Congenital neevus
Congenital neoplasm
Congenital neoplasm
Congenital vaginal cyst
Congenital vaginal cyst
Congenital vaginal cyst
Congenital vaginal cyst
Congenital vaginal cyst
Congenital vaginal cyst
Conjunctival primary acquired melanosis
Congenital vaginal cyst
Conjunctival primary acquired melanosis
Conjunctival primary acquired melanosis
Conjunctival primary acquired melanosis
Conjunctival cyst
Conjunctival primary acquired melanosis
Conjunctival primary acquired melanosis
Conjunctival primary acquired melanosis
Conjunctival primary acquired melanosis
Conferential cyst
Cyst rupture
Cyst rupture
Cyst congenital
Cystic engiomatosis
Cyst rupture
Cystic engiomatosis
Cystic lymphangioma
Cyst congenital B increased
Cystoprostatectomy
Cytokeratin 18 increased
Dermoid cyst
Dermoid

| N9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| 35-4506 | | Version: | 1.0 | Page: | 167 of 229 | |
| Pre-defined MedDRA search - list of preferred | preferred terms | | | | | |

Eastern Cooperative Oncology Group performance Eastern Cooperative Oncology Group performance Dysplasia Dysplastic naevus Dysplastic naevus syndrome Ear neoplasm

Ectopic ACTH syndrome
Ectopic and diduretic hormone secretion
Ectopic antiduretic hormone secretion
Ectopic calcitonin production
Ectopic calcitonin production
Ectopic continuing gonadotrophin secretion
Ectopic crowth hormone secretion
Ectopic parathyroid hormone production
Electron radiation therapy to blood
Electron radiation therapy to breast
Electron radiation therapy to colon
Electron radiation therapy to liver
Electron radiation therapy to lung
Electron radiation therapy to lung
Electron radiation therapy to skin
Electron radiation therapy to soft tissue
Electron radiation therapy to soft tissue
Electron radiation therapy to soft tissue
Electron radiation therapy to uterus

Encephalitis autoimmune

Enchondromatosis

Endobronchial lipoma Endocervical mucosal thickening

Endocrine neoplasm
Endometrial adenoma
Endometrial dysplasia
Endometrial hyperplasia

Pre-defined MedDRA search

Preferred term

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 Page: | 168 of 229 | |
| Pro-defined MedDRA search - list of preferred terms | f preferred terms | | | | |

Neoplasm

Pre-defined MedDRA search

Epithelioma adenoides cysticum Epstein Barr virus positive mucocutaneous ulcer Epstein-Barr virus associated lymphoproliferative Eyelid naevus
Eyelid naevus
Eyelid seborrhoeic keratosis
Eyelid tumour
Fallopian tube leiomyoma
Fallopian tube leiomyoma
Familial acromegaly
Familial haemophagocytic lymphohistiocytosis
Femilial multiple lipomatosis
Femilial multiple lipomatosis
Femilial multiple lipomatosis Epidermal naevus syndrome
Epidermodysplasia verruciformis
Epididymal cyst
Epiglottic cyst
Epiglottic mass
Epiglottic mass Fibromatosis Fibromatosis colli of infancy Erythroplasia of lip
Erythroplasia of lip
Erythroplasia of penis
Erythroplasia of vulva
Essential thrombocythaemia
Ex vivo gene therapy
Exploratory operation
Extended radical mastectomy Fibroadenoma of breast Fibrocystic breast disease disorder Erdheim-Chester disease Endometrial neoplasm Extradural neoplasm Ependymoma Ependymoma benign Eye haemangioma Eye naevus

| inical Trial Report Date: 04 December 2020 Status: | Version: 1.0 Page: | eferred terms |
|---|---|---|
| NN9535 Clinical | 49535-4506 | Pre-defined MedDRA search - list of prefer |

Final Novo Nordisk


Neoplasm

Pre-defined MedDRA search

Fractor of prostate-specific antigen increased Free prostate-specific antigen positive Fractor wound Gallbladder adenoma Gallbladder adenoma Gallbladder polyp Gamma interferon therapy to blood Gamma radiation therapy to blood Gamma radiation therapy to blood Gamma radiation therapy to blood Gamma radiation therapy to brain Gamma radiation therapy to brain Gamma radiation therapy to colon Gamma radiation therapy to colon Gamma radiation therapy to colon Gamma radiation therapy to colon Gamma radiation therapy to colon Gamma radiation therapy to plung Gamma radiation therapy to plura Gamma radiation therapy to pleura Gamma radiation therapy to pleura Gamma radiation therapy to pleura Gamma radiation therapy to prostate Gamma radiation therapy to soft tissue Gamma radiation therapy to soft tissue Gamma radiation therapy to styroid Gamma radiation therapy to thyroid Gamma radiation therapy to thyroid Gamma radiation therapy to thyroid Gamma radiation therapy to thyroid Gamma radiation therapy to thyroid Fibrous cortical defect
Fibrous histiocytoma
Fiducial marker placement
Fms-like tyrosine kinase 3 positive Foetal cystic hygroma Follicular cystitis

Gastric adenoma Gastric haemangioma Gammopathy Ganglioneuroma Garcin syndrome Gastrectomy

Gastric lelomyowa Gastric neoplasm Gastric polypectomy Gastric stent insertion Gastrin-releasing peptide precursor increased

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | .0 Page: 1 | 170 of 229 |
| Pre-defined MedDRA search - list of prefe | f preferred terms | | | | |

Novo Nordisk

Neoplasm

Pre-defined MedDRA search

Hemipelvectomy
Hepatic cyst infection
Hereditary multiple osteochondromas
Hereditary non-polyposis colorectal cancer Granular cell tumour Granulosa cell tumour of the testis Growth hormone-producing pituitary tumour Haemangioblastoma Haematopoietic neoplasm
Haemophagocytic lymphohistiocytosis
Haemophilic pseudotumour
Haemorrhagic breast cyst
Haemorrhagic cyst
Haemorrhagic cyst
Haemorrhagic thyroid cyst
Haemorrhagic thyroid cyst
Haemorrhagic tumour necrosis
Hair follicle tumour benign Haemangioma rupture Haemangioma-thrombocytopenia syndrome Gastrinoma
Gastrointestinal neoplasm
Gastrointestinal submucosal tumour
Gastrointestinal tract adenoma Germ cell neoplasm Giant cell tumour of tendon sheath Glomus tumour Glossectomy Genitourinary tract neoplasm Haemangioma of bone Haemangioma of breast Haemangioma of retina Haemangioma of skin Haemangioma of spleen Haemangioma congenital Heavy chain disease Hamartoma vascular Hemicorporectomy Gorham's disease Good syndrome Genital cyst Haemangioma syndrome

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 171 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

High frequency ablation
High intensity focused ultrasound
Histiocytic necrotising lymphadenitis
Histiocytosis
Hormone suppression therapy
Hormone therapy
Hormone suppression therapy
Hormone scretching ovarian tumour
Horner's syndrome
Human chorionic gonadotropin positive
Human chorionic gonadotropin positive
Human chorionic gonadotropin positive
Human chorionic gonadotropin positive
Hypercalcaemia of malignancy
Hypercalcitoninaemia benign monoclonal
Hypercalcitoninaemia benign monoclonal
Hyperreactio luteinalis
Hyperreactio luteinalis
Hyperreactio luteinalis
Hyperreactio luteinalis
Hyperreactio luteinalis
Hyperreactio seteomathropathy
Hyperreactio luteinalis
Hyperreactio seteomalacia
Hypopharyngeal neoplasm benign
Hypopharyngeal neoplasm benign
Hypopharyngeal neoplasm benign
Hypopharyngeal neoplasm
Hypopharynge

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 172 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | |

Infected lymphocele
Infected neavus
Infected neavus
Infected neavus
Infected neavus
Infected neoplasm
Inflammatory pseudotumour
Insulinoma
Interleukin therapy
Intestinal angioma
Intestinal polypectomy
Intracabdominal haemangioma
Intracabdominal haemangioma
Intracabdominal haemangioma
Intracabdominal haemangioma
Intracabdominal haemangioma
Intracacanial haemangioma
Intracacseous angiloma of breast
Intraductal papillary mucinous neoplasm
Intracoseous meningioma
Intracoseous meningioma
Intracoseous meningioma
Intracoseous meningioma
Intravescular lipoma
Intravescular lipoma
Intravescular lipoma
Intravescular papillary endothelial hyperplasia
Intravescular papillary endothelial out neoplasm
Incommal gland neoplasm
Inace intestinal polypectomy
Inace intestinal polypectomy
Inace intestinal polypectomy
Inace intestinal polypectomy
Inace intestinal dout neoplasm
Inace intestinal polypectomy
Inace intestinal polypectomy
Inace intestinal dout neoplasm
Inace intestinal dout neoplasm
Inace intestinal polypectomy
Inace intestinal polypectomy
Inace intestinal polypectomy
Inace intestinal dout neoplasm
Inace intestinal dout neoplasm
Inace intestinal polypectomy
Inace intestinal plandandal dysplasia

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 173 of 229 |
| Pre-defined MedDRA search - list of pref | f preferred terms | | | | |

Novo Nordisk

Neoplasm

Pre-defined MedDRA search

Laryngeal neoplasm
Laryngeal papilloma
Laryngeal polypectomy
Laryngeal polypectomy
Laryngeal polypectomy
Laryngectomy
Leukoplakia of penis
Leukoplakia of penis
Leukoplakia of penis
Leukoplakia of penis
Leukoplakia of penis
Liphot encephalitis
Liphotoplasm
Liphotoplasm
Liphotoma
Lipodermoid tumour
Lipodermoid tumour
Lipodermoid tumour
Lipodermoid tumour
Lipodermoid tumour
Lipodermoid tumour
Lipoma
Lipodermoid tumour
Liphotoplasm
Liphotoplasm
Lung lobectomy
Lung lobectomy
Lung lobectomy
Lung neoplasm surgery
Lung neoplasm surgery
Lung neoplasm surgery
Lung neoplasm surgery
Lung neoplasm
Lymphatic system neoplasm
Lymphocyte adoptive therapy
Lymphocyte adoptive disorder in remission
Lymphoproliferative disorder in
Lymphoproliferative disorder in
Lymphoproliferative disorder
Lymphoproliferative disorder
Lymphoproliferative assites
Malignant exophthalmos
Malignant exophthalmos
Malignant exophthalmos
Malignant exophthalmos

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NIN9333-4300 | 1 | v ersion: | 0.1 | rage: | 1/4 01 229 | |
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| | | | | | | ! |
| Pre-defined MedDRA search | Preferred term | | | | | |

Malignant pleural effusion
Malignant psoas syndrome
Malignant urinary tract obstruction
Marignant urinary tract obstruction
Mastectomy
Mastectomy
Mastocid cyst
Mastoid cyst
Mastoid cyst
Maxillofacial sinus neoplasm
Maxillofacial sinus neoplasm
Maxillofactial sinus neoplasm
Mediastinal biopsy abnormal
Mediastinal cyst
Mediastinal cyst
Mediastinal cyst
Mediastinal cyst
Mediastinal cyst
Mediastinal cyst
Mediastinal cyst
Mediastinal syndrome
Medical device site cyst
Mediastinal neoplasm
Medical device site cyst
Medical device site cyst
Medical neoplasm
Meningeal neoplasm
Meningioma benign
Meningioma benign
Mesonteric neoplasm
Mesonephic duct cyst
Mesonephic duct cyst
Mesonephic skin surgery
Mesotratic bone disease prophylaxis
Metastatic bone disease prophylaxis
Metastatic pulmonary embolism
Metastatic pulmonary embolism
Metastatic pulmonary embolism
Mutcontal gammopathy
Muocal cyst of postmasticoytosis
Multiple rotaneous and uterine leiomyomatosis
Multiple endocrine neoplasia Type 1
Multiple endocrine neoplasia Type 2

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Preferred term

Neoplasm

Pre-defined MedDRA search

Myasthenic syndrome
Myeloblast present
Myeloblast present
Myelodysplastic syndrome
Myelodysplastic syndrome transformation
Myelodysplastic syndrome unclassifiable
Myelodysplastic syndrome unclassifiable
Myelofibrosis
Myeloid metaplasia
Myeloid metaplasia
Myeloproliferative neoplasm
Myoloproliferative neoplasm
Myoloproliferative neoplasm
Myoloproliferative neoplasm
Myopericytoma
NMP22 test abnormal
Nacyla benormal
Nacyla neoplasm
Nasal neoplasm
Nasal neoplasm
Nasal neoplasm
Nasal polyps
Nasopharyngeal polyp
Nasopharyngeal polyp
Nasopharyngeal tumour
Neck dissection
Nacylasm
Neoplasm

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | | Final Novo |
|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 176 of 229 |
| Pre-defined MedDRA search - list of preferred | preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | |

Neurolemental neoplasm surgery
Neuroectodermal neoplasm
Neurocachemal neoplasm
Neuroectodermal neoplasm
Neuroectodermal neoplasm
Neurofibroma
Neurogenic tumour
Neuroma
Neurogenic tumour
Neuroma
Nipple resection
Nipple resection
Nodular fasciitis
Non-serretory adenoma of pituitary
Numb chin syndrome
Ocular neoplasm
Ocular neoplasm
Ocular surface squamous neoplasia
Ocular surface squamous neoplasm
Ocsophageal polypectomy
Ocsophageal prosthesis insertion
Ocsophageal prosthesis insertion
Ocsophageal prosthesis insertion
Ocsophageal prosthesis
Ocsophageal prosthesis
Ocsophageal prosthesis
Ocsophageal prosthesis
Ocsophageal prosthesis
Ocsophageal prosthesis
Occoptoma
Omentectomy
Oncologic complication
Omentectomy
Oncologic complication
Occoptoma
Oral hairy leukoplasm
Oral hairy leukoplasm
Oral neoplasm
Oral papilloma
Oral papilloma
Oral papilloma
Oral papilloma
Oral papilloma
Oral papilloma

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 177 of 229 | |
| Pre-defined MedDRA search - list of preferrec | preferred terms | | | | | |

Preferred term Pre-defined MedDRA search

Neoplasm

Ovarian Sertoli-Leydig cell tumour
Ovarian adenoma
Ovarian cyst
Ovarian cyst ruptured
Ovarian cyst torsion
Ovarian dysplasia
Ovarian dysplasia
Ovarian germ cell teratoma benign
Ovarian germ cell tumour
Ovarian germ cell tumour
Ovarian neoplasm
Ovarian neoplasm
Ovarian heoplasm
Ovarian theca cell tumour
PHACES syndrome
PMI/RAR alpha expression
POEMS Syndrome Pancreaticosplenectomy
Papillary cystadenoma lymphomatosum
Papillary tumour of renal pelvis
Papilloma conjunctival Oropharyngeal dysplasia Oropharyngeal neoplasm Oropharyngeal neoplasm benign Pancoast's syndrome Pancreastatin abnormal Pancreastatin increased Pancreaticoduodenectomy Orbital exenteration Orchidectomy Orchidotomy Pancreatectomy Pancreatic neoplasm Pachydermodactyly Palliative care Palmar fasciitis Ostectomy Osteochondroma Osteofibroma Osteoma cutis Ota's naevus Osteoma

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | 0 Page: | 178 of 229 | |

Neoplasm

Pre-defined MedDRA search

Paraganglion neoplasm
Paraganglion neoplasm
Paraganglion neoplasm
Paranasal sinus benign neoplasm
Paranasal sinus benign neoplasm
Paranasal sinus benign neoplasm
Paranacoplastic dermatomyositis
Paraneoplastic dermatomyositis
Paraneoplastic dermatomyositis
Paraneoplastic dermatomyositis
Paraneoplastic myelopathy
Paraneoplastic myelopathy
Paraneoplastic nephrotic syndrome
Paraneoplastic nephrotic syndrome
Paraneoplastic nephrotic syndrome
Paraneoplastic pemphigus
Paraneoplastic retinopathy
Paraneoplastic retinopathy
Paraneoplastic syndrome
Paraneoplastic syndrome
Parathyroid cyst
Parathyroid tumour
Parathyroid cyst
Perile opoplasm
Penile warts excision
Penile warts excision
Penile warts excision
Penile warts excision
Pericardial cyst
Pericardial cyst

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 179 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ı İ |

Pericardial lipoma
Pericardial neoplasm
Pericardial neoplasm
Pericardial cyst
Perineal cyst
Perinential cyst
Peripheral nervous system neoplasm
Peritoneal pliomatosis
Peritonectomy
Peritonectomy
Peritonectomy
Peritonectomocytoma
Peritonecytoma
Peritonecytoma
Peritonecytoma
Peritonecytoma
Phaeochromocytoma crisis
Phaeochromocytoma crisis
Pharyngeal leukoplakia
Pharyngeal leukoplakia
Pharyngeal neoplasm
Photon radiation therapy to bloode
Photon radiation therapy to bone
Photon radiation therapy to brain
Photon radiation therapy to liver
Photon radiation therapy to pleura
Photon radiation therapy to pleura
Photon radiation therapy to soft tissue
Photon radiation therapy to soft tissue
Photon radiation therapy to soft tissue
Photon radiation therapy to shin
Photon radiation therapy to shin
Photon radiation therapy to short tissue
Photon radiation therapy to soft tissue
Photon radiation therapy to thorus
Photon radiation therapy to thorus
Photon radiation therapy to soft tissue
Photon radiation therapy to thorus
Photon radiation therapy to thorus
Photon radiation therapy to thorus
Photon radiation therapy to thorus
Photon radiation therapy to soft tissue
Photon radiation therapy to thorus

| NN9535 | Clinical Trial Report | Date: | 34 December 2020 St | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 Page | ige: | 180 of 229 | |
| Pre-defined MedDRA search - list of preferred | f preferred terms | | | | | |

Neoplasm

Pre-defined MedDRA search

Pineal gland cyst
Pineal neoplasm
Pineal neoplasm
Pineal meoplasm
Pineal meoplasm
Pineal meoplasm
Pituitary gland radiotherapy
Pituitary gland radiotherapy
Pituitary tumour benign
Pituitary tumour recurrent
Pituitary tumour recurrent
Placental chorioangioma
Placental neoplasm
Placental neoplasm
Placental neoplasm
Pleural cyst
Pleural cyst
Pleural cyst
Pleural cyst
Pleural proper proper property
Pleural neoplasm
Placental polyp
Pleural property
Polyp
Pleural property
Polyp
Post preast therapy pain syndrome
Post transplant lymphoproliferative disorder
Post transplant lymphoproliferative disorder
Post transplant lymphopedema syndrome
Post transplant lymphopedema syndrome
Post transplant lymphopedema syndrome
Precancerous condition
Precancerous skin lesion
Precancerous skin lesion
Precancerous skin lesion
Precancerous skin lesion
Precancerous skin lesion
Precancerous skin lesion
Precancerous receptor assay positive
Protectomy
Prostate clineralion
Prostate cryoablation
Prostate cryoablation
Prostate cryoablation
Prostatic cyst
Prostatic copst

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Final / | Novo Nordisk |
|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 Page: | 181 of 229 | |
| Dro_dofised ModDDs sees to list of reactived towns | 7 2 3 4 4 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 | | | | |

recognised MedDRA search - list of preferred terms

Preferred term

Neoplasm

Pre-defined MedDRA search

Prostatic dysplasia
Prostatic polyp
Prostatic polyp
Prostatic specific antigen abnormal
Prostatic specific antigen increased
Pseudomyxoma peritone;
Pyderma geritone;
Pyderma gangrenosum
Pyderma gangrenosum
Pydenic granuloma
Radical pysterectomy
Radical masterctomy
Radical masterctomy
Radical masterctomy
Radical masterctomy
Radical masterctomy
Radical masterctomy
Radical masterctomy
Radical prostatectomy
Radicherapy to adrenal gland
Radicherapy to bone
Radicherapy to bone
Radicherapy to bone
Radicherapy to breast
Radicherapy to breast
Radicherapy to ear
Radicherapy to ear
Radicherapy to ear
Radicherapy to breast
Radicherapy to wallbladder
Radicherapy to wallbladder
Radicherapy to wallbladder
Radicherapy to liver
Radicherapy to mediastinum
Radicherapy to mose

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 182 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | : preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ı |

Radiotherapy to oesophagus
Radiotherapy to oral cavity
Radiotherapy to oral cavity
Radiotherapy to pancreas
Radiotherapy to pancreas
Radiotherapy to percetate
Radiotherapy to prostate
Radiotherapy to prostate
Radiotherapy to spleen
Radiotherapy to spleen
Radiotherapy to spleen
Radiotherapy to spleen
Radiotherapy to thywoid
Radiotherapy to thywoid
Radiotherapy to thywoid
Radiotherapy to thywoid
Radiotherapy to turinary bladder
Radiotherapy to turinary bladder
Radiotherapy to turinary bladder
Radiotherapy to turinary bladder
Radiotherapy to vininary bladder
Radiotherapy to vininary bladder
Radiotherapy to vininary bladder
Radiotherapy to vininary bladder
Radiotherapy to vininary bladder
Radiotherapy to vyepenia with miltilineage dysplasia
Refractory anaemia with miltilineage dysplasia
Refractory cytopenia with unilineage dysplasia
Refractory cytopenia with unilineage dysplasia
Refractory cytopenia with unilineage dysplasia
Renal adenoma
Renal cost infection
Renal cost infection
Renal lamartoma
Renal haemangioma
Renal neoplasm
Renal neoplasm
Renal tumour excision
Respiratory papilloma
Respiratory tract neoplasm
Respiratory papilloma
Respiratory papilloma
Respiratory tract neoplasm
Retention cyst

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 183 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDBA search | Dreferred term | | | | | |

Retinal melanocytoma
Retinal neoplasm
Retinal tumour excision
Retro-orbital neoplasm
Retro-pubic prostatectomy
Retro-pubic prostatectomy
Retro-pubic prostatectomy
Retroperitoneal neoplasm
Rosai-Dorfman syndrome
Salivary gland adenoma
Salivary gland neoplasm
Salivary gland resection
Salivary gland resection
Salivary gland scan abnormal
Salpingo-cophorectomy
Scan adrenal gland abnormal
Scan adrenal gland abnormal
Scan adrenal gland abnormal
Scan adrenal gland abnormal
Scan with contrast abnormal
Scan with contrast abnormal
Schwannoma
Schoardown
Scarosing pneumocytoma
Schocous naevus
Sebaccous naevus
Seba
| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Vovo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 184 of 229 | |
| Pre-defined MedDRA search - list of preferre | f preferred terms | | | | | |

Neoplasm

Pre-defined MedDRA search

Skin cryotherapy
Skin neoplasm bleeding
Skin neoplasm bleeding
Skin neoplasm excision
Skin neoplasm excision
Skin neoplasm excision
Skall intestinal polypectomy
Small intestinal resection
Smooth muscle cell neoplasm
Sofitary epithelioid histiocytoma
Solitary fibrous tumour
Solitary fibrous tumour
Solitary fibrous tumour
Solitary fibrous tumour
Solitary fibrous tumour
Solitary fibrowal
Spermatocele
Spinal cord cyst
Spermatocele
Spinal cord lipoma
Spinal cord lipoma
Spinal cord lipoma
Spinal meningeal cyst
Spinal sonovial cyst
Spinal sonovial cyst
Spinal meningeal cyst
Spinal meningeal cyst
Spinal meningeal cyst
Spinal meningeal cyst
Spinal meningeal cyst
Spinal sonovial cyst
Spinal meningeal cyst
Spinal meningeal cyst
Spinal spinovial cyst
Spinal meningeal cyst
Spinal meningeal cyst
Stauffer: syndrome
Stauffer: syndrome
Stoma site polyp
Stoma si

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 185 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | l |

Neoplasm

Testicular neoplasm
Testicular papilloma
Testicular scan abnormal
Testicular teratoma benign
Thymic cyst
Thymic cyst
Thymodolossal cyst
Thyroid decoma
Thyroid decoma
Thyroid decoma
Thyroid alectron radiation therapy
Thyroid alectron radiation therapy
Thyroid alectron radiation therapy
Thyroid delectron radiation therapy
Thyroid delectron radiation therapy
Thyroid delectron radiation therapy
Thyroid delectron abnormal
Thyroid delectron abnormal
Thyroid delectron
Thyroid delectron
Thyroid delectron
Thyroid stimulating hormone-producing pituitary
Thyroid delectron
Thyroid delectron
Thyroid delectron
Thyroid delectron
Tongue neoplasm
Tongue neoplasm
Tonsillar neoplasm
Tonsillar neoplasm
Tonsillar cyst
Tonsillar neoplasm
Tonsillar neoplasm
Tracheal neoplasm
Tracheal papilloma
Tracheal papilloma
Tracheal papilloma
Tracheal papilloma
Tracheal resection
Transcatheter arterial chemoembolisation
Transcrehral prostatectomy
Transcrehral prostatectomy
Transcrehral brostatectomy
Trisomy 12
Twoour sclerosis complex
Tumour associated fever
Tumour cavitation
Tumour compression
Tumour excision
Tumour excision

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|
| NN9535-4506 | _ | Version: | 1.0 Page: | 186 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | l l |

Neoplasm

Tumour fistulisation
Tumour fistulisation
Tumour flate
Tumour haemorrhage
Tumour inflammation
Tumour inflammation
Tumour lysis syndrome
Tumour marker abnormal
Tumour marker decreased
Tumour marker increased
Tumour marker increased
Tumour perforation
Tumour perforation
Tumour perforation
Tumour perforation
Tumour pruritus
Tumour pruritus
Tumour pruritus
Tumour preding fields therapy
Tumour treating fields therapy
Tumour ulceration
Tumour accine therapy
Ulcerated haemangioma
Ultrasound scan vagina abnormal
Ultrasound scan vagina abnormal
Ultrasound scan vagina abnormal
Ultrasound scan vagina abnormal
Ultrasound scan abnormal
Ultrasound scan abnormal
Ultrasound scan abnormal
Ultrasound scan abnormal
Ultrasound scan abnormal
Ultrasound scan vagina ubnormal
Ultrasound scan vagina ubnormal
Ultrasound scan poplasm
Urethral popiloma
Urethral popiloma
Urethral popiloma
Urethral popiloma
Urethral popiloma
Urethral popiloma
Urethral popiloma
Urinary bladder adenoma
Urinary bladder polyp
Urinary tract poolyp
Urinary tract poolyp

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | 1.0 Page: | 187 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I I |

Neoplasm

Uterine leiomyoma
Uterine myoma expulsion
Uterine mosplasm
Uterine polyp
Uterine polyp
Uterine tumour excision
Uvulectomy
Vaccination site cyst
Vaginal cyst
Vaginal cyst
Vaginal polyp
Vaginal polyp
Vaginal polyp
Vascular neoplasm
Vaginectomy
Viral acanthoma
Viral acanthoma
Viral acanthoma
Viral accord leukoplakia
Vocal cord polyp
Vocal cord polyp
Vocal cord polyp
Volva cyst
Vocal cord polyp
Vulva cyst
Vulva colon
X-ray therapy to brant
X-ray therapy to colon
X-ray therapy to colon
X-ray therapy to colon
X-ray therapy to colon
X-ray therapy to colon
X-ray therapy to colon
X-ray therapy to colon
X-ray therapy to liver
X-ray therapy to liver
X-ray therapy to liver

| NN9535<br>NN9535-4506<br>Pre-defined MedDRA search - list | Clinical Trial Report<br> -<br>of preferred terms | Date:<br>Version: | 04 December 2020 Status:<br>1.0 Page: | Final Novo Nordisk |
|---|---|---|---|---|
| Pre-defined MedDRA search | Preferred term | | | 1 |
| Neoplasm | X-ray therapy to X-ray therapuloua | ay therapy to lung ay therapy to pancreas ay therapy to pleura ay therapy to prostate ay therapy to skin ay therapy to soft tissue ay therapy to thyroid ay therapy to uterus ay therapy to uterus ay treatment thogranuloma k sac tumour site unspecified | | |
| Pancreatitis | Alcoholic pancreatitis Alcoholic pancreatitis Autoimmune pancreatitis Haemorrhagic necrotic pancreat Immune-mediated pancreatitis Ischaemic pancreatitis Lupus pancreatitis Obstructive pancreatitis Obstructive pancreatitis Pancreatic necrosis Pancreatic phelogmon Pancreatic pseudocyst Pancreatic pseudocyst haemorrh Pancreatic pseudocyst rupture Pancreatitis seudocyst rupture Pancreatitis acute Pancreatitis acute Pancreatitis is acute Pancreatitis necrotising Chancreatitis haemorrhagic Pancreatitis is necrotising Chancreatitis shamorrhagic Pancreatitis shamorreatitis Cythomegalovirus pancreatitis Pancreatitis shamorreatitis Pancreatitis pancreatitis Pancreatitis pancreatitis Pancreatitis bacterial | ancreatitis cancreopathy pancreatitis concortic pancreatitis catific ancreatitis catifis catifis pancreatitis pancreatitis pancreatitis haemorrhage necrosis phelogmon pseudocyst haemorrhage pseudocyst haemorrhage pseudocyst rupture ts chronic ts haemorrhagic ts chronic ts haemorrhagic ts chronic | | |

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|
| NN9535-4506 | ı | Version: | 1.0 Page: | 189 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | |

Pancreatitis fungal
Pancreatitis helminthic
Pancreatitis mumps
Pancreatitis viral
Pancreatorenal syndrome

Rare events

Pancreatitis

Radiation pancreatitis
Traumatic pancreatitis
Traumatic pancreatitis
11-beta-hydroxylase deficiency
17,20-desmolase deficiency
17,20-desmolase deficiency
18 minus syndrome
20,22-desmolase deficiency
21-hydroxylase deficiency
3-hydroxyacetyl-coenzyme A dehydrogenase
deficiency
3-hydroxyacetyl-coenzyme A dehydrogenase
deficiency
3-hydroxyacetyl-coenzyme A dehydrogenase
deficiency
ADD Syndrome
5-alpha-reductase deficiency
ADC S-related dyskinesia
ADN Syndrome
ADO ASTAIL related dyskinesia
ADN Syndrome
ADN Syndrome
ADN Syndrome
ADO Syndrome
ADO Syndrome
ADO STAIL STAIL STAIL STAIL STAIL STAIL
ADD SYNDROM SACCESSORY KINDROM ACCESSORY KINDROM ACCESSORY MINDROM ACCESSORY MINDR

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 S | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 90 of 229 |
| Pre-defined MedDRA search - list of prefe | f preferred terms | | | | |

Novo Nordisk

Rare events

Pre-defined MedDRA search

Accessory spleen
Activated Thiers syndrome
Actured Thiers syndrome
Actured Thiers syndrome
Actured amegakaryocytic thrombocytopenia
Acquired dene mutation
Acquired mitochondrial DNA deletion
Acquired mitochondrial DNA mutation
Acquired mitochondrial DNA mutation
Acrocallosal syndrome
Acrocallosal syndrome
Acrocallosal syndrome
Acrocarmatitis enteropathica
Acrodermatitis enteropathica
Acrodermatitis enteropathica
Acrodermatitis enteropathica
Acroderosis verruciformis
Acroderosis verruciformis
Acromicric dysplasia
Activated P13 kinase delta syndrome
Activated P13 kinase delta syndrome
Activated P13 kinase delta syndrome
Activated P13 kinase delta syndrome
Activated P13 kinase delta syndrome
Activated P13 kinase delta syndrome
Activated P14 kinase deficiency
Adactyly
Adams-Oliver syndrome
Adenine phosphoribosyl transferase deficiency
Adenine phosphoribosyl transferase
Adenil polyglucosan body disease
Adardi's syndrome
Algiosile syndrome
Albinism
Albinism
Albinism
Alexander disease
Alexander disease
Alexander disease
Alexander disease
Alexander disease

Alpers disease
Alpha-1 antitrypsin deficiency
Alpha-mannosidosis
Alpha-to-1 antitrypsin deficit syndrome
Alpha-thalssaemia-intellectual deficit syndrome
Alport's syndrome

Allan-Herndon-Dudley syndrome

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 Page: | 191 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | |

Rare events

Pre-defined MedDRA search

Alstroem syndrome
Alternating hemiplegia of childhood
Alveolar capillary dysplasia
Alveolar capillary dysplasia
Alveolar lung disease
Alveolitis
Alveolitis necrotising
Alveolitis necrotising
Amblyopia congenital
Amegakaryocytic thrombocytopenia
Aminoaciduria
Aminoaciduria
Aminotic band syndrome
Amyotrophic lateral sclerosis gene carrier
Anal atresia
Angelman's syndrome
Angelman's syndrome
Angelman's syndrome
Angelman's syndrome
Angelman's syndrome
Angelman's syndrome
Angelman's syndrome
Angelman's congenital
Anitidia-cerebellar ataxia-mental deficiency
Anodontia
Anodontia
Anomaly of external ear congenital
Anomaly of external ear congenital
Anomaly of fiddle ear congenital
Anomaly of fiddle ear congenital
Anomaly of fiddle ear congenital
Anomaly of fiddle ear congenital
Anotic associated colitis
Anterior displaced anus
Antibiotic associated colitis

Rare events

Pre-defined MedDRA search

Aplasia Aplasia
Aplasia cutis congenita
Aplasia cutis congenita
Aplasia cutis congenita
Aplasia cutis anaemia
Apolipoprotein E e4 gene carrier
Apparent mineralocorticoid excess
Arachnodactyly
Argininosuccinate lyase deficiency
Argininosuccinate synthetase deficiency
Argininosuccinate synthetase deficiency
Argininosuccinate synthetase deficiency
Argininosuccinate synthemation
Aspartylglucosaminuria
Aspartylglucosaminuria
Aspartylglucosaminuria
Aspartylglucosaminuria
Aspartylglucosaminuria
Aspartylglucosaminuria
Aspartylglucosaminuria
Atxia telangiectasia
Atxia telangiectasia
Atxia telangiectasia
Atxia telangiectasia
Atxia telangiectasia
Autoimmune aplastic anaemia
Autoimmune aplastic anaemia
Autoimmune nephritis
Autoimmune nephritis
Autoimmune nephritis
Autoimmune nephritis
Autoimmune nephritis
Buttosomal recessive megaloblastic anaemia
Azygos lobe
B-lymphocyte count decreased
B-lymphocyte count decreased
B-lymphocyte count decreased
B-lymphocyte count decreased
B-lymphocyte count decreased
B-lymphocyte mutation
BRCA2 gene mutation
BRCA2 gene mutation
BRCA2 gene mutation
Baller-Gerold syndrome
Baller-Gerold syndrome
Baller-Gerold syndrome
Baller-Gerold syndrome
Baller-Gerold syndrome
Baller mycollonic epilepsy
Band neutrophil percentage decreased
Band neutrophil percentage decreased

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 Page: | 193 of 229 | |
| | 4 | | | | |

Preferred term Pre-defined MedDRA search - list of preferred terms Pre-defined MedDRA search

Rare events

```
Baraitser Rodeck Garner syndrome
Barakat syndrome
Barther Syndrome
Barther Syndrome
Barther Syndrome
Barther Syndrome
Basophil count decreased
Basophil percentage decreased
Beckwith-Wiedemann Syndrome
Benign familial neonatal convulsions
Benign familial pemphigus
Betaketothiolase deficiency
Bicketstaff's encephalitis
Bicketstaff's encephalitis
Bloch-Sulzberger syndrome
Bloch-Sulzberger syndrome
Bloch disorder
Blood disorder
Blood disorder
Blood disorder
Bone marrow failure
Bone marrow failure
Bone marrow failure
Bone marrow toxicity
Brachydactyly
Brachymetatarsia
```

| Final Novo Nordisk | 194 of 229 |
|-----------------------|-------------|
| Status: | Page: |
| 04 December 2020 | 1.0 |
| Clinical Trial Report | |
| NN9535 | NN9535-4506 |

Pre-defined MedDRA search - list of preferred terms

Preferred term

Rare events

Pre-defined MedDRA search

Brachyolmia

Brain malformation

Brain malformation

Branchial cleft sinus

Branchial cleft sinus

Branchial syndrome

Bronchial atreaia

C-kit gene mutation

C-kit gene mutation

C-kit gene wutation

C-kit gene wutation

C-kit gene wutation

C-kit gene wutation

C-kit gene mutation

C-kit gene mutation

C-kit gene mutation

C-kit gene mutation

C-kit gene mutation

C-kit gene wutation

C-kit gene wutatio

| NN9535<br>NN9535-4506 | Clinical Trial Report<br> - | Date: | 04 December 2020 Status: 1.0 Page: | 20 Status:<br>0 Page: | Final<br>195 of 229 | Final <b>Novo Nordisk</b><br>f 229 |
|---|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I |

Rare events

Carbonic anhydrase gene mutation
Cardiac malposition
Cardiac malposition
Cardiofaciocutaneous syndrome
Carnitine palmitoyltransferase deficiency
Carnitine palmitoyltransferase deficiency
Carnitine-acylcarnitine translocase deficiency
Carnitine-acylcarnitine translocase deficiency
Carnitine-acylcarnitine translocase deficiency
Carpenter syndrome
Carpenter syndrome
Cataract congenital
Catel Manzke syndrome
Cataract core disease
Careballar hypoplasia
Cereballar hypoplasia
Choral auricle
Cervical auricle
Chonal atresia
Choral auricle
Chonal atresia
Choral auricle
Choral auricle
Choral auricle
Choral auricle
Choral auricle
Choral auricle
Choral auricle
Choral Companion
Choral auricle
Correballar dysplasia
Correballar dysplasia
Correballar dysplasia
Correbal

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 196 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | : preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | ı |

Rare events

Cleft lip and palate
Cleft lip and palate
Cleft palate
Cleft towns
Cleidocranial dysostosis
Clinodactyly
Cloacal exstrophy
Cloactridian linfection
Clostridian bacteraemia
Clostridium difficile infection
Clostridium difficile colitis
Clostridium difficile infection
Cockayne's syndrome
Coffin-Lowry syndrome
Coffin-Lowry syndrome
Coffin-Lowry syndrome
Coffin-Lowry syndrome
Coffin-Lowry syndrome
Complement deficiency disease
Complement deficiency disease
Complement deficiency disease
Complement deficiency disease
Congenital Ebola virus infection
Congenital Bustachian tube anomaly
Congenital absence of bile ducts
Congenital absence of bile ducts
Congenital absence of cranial vault
Congenital absence of bile ducts
Congenital absence of bile ducts
Congenital absence of bile ducts
Congenital absence of vertebra
Congenital anaemia
Congenital anaemia
Congenital anaemia
Congenital anaemia
Congenital anaemia
Congenital anaemia
Congenital anaemia
Congenital anaemia
Congenital anoemial sof ear ossicles

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Final Novo N |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 197 of 229 | |
| Pre-defined MedDRA search - list of | of preferred terms | | | | | |

Nordisk

Rare events

Pre-defined MedDRA search

Congenital anomaly in offspring Congenital anomaly in offspring Congenital anomaly of inner ear Congenital anomaly of inner ear Congenital acrtic anomaly Congenital acrtic anomaly Congenital acrtic anomaly Congenital acrtic careaia Congenital acrtic stenosis Congenital acrtic valve stenosis Congenital acrtic valve stenosis Congenital acrterial malformation Congenital arterial malformation Congenital bladder anomaly Congenital bladder anomaly Congenital bladder anomaly Congenital bronchectasis Congenital bronchectasis Congenital bronchectasis Congenital bronchectasis Congenital calivosacular anomaly Congenital carticle dispetes inabjoidus Congenital carticle dispetes inabjoidus Congenital central hypoventilation syndrome Congenital central hypoventilation syndromic central central nervous system anomaly Congenital choroidal anomaly Congenital corneal anomaly Congenital concental carticle are agenesis Congenital congenital corneal anomaly Congenital corneal anomaly Congenital Corneal Acrtic Largenesis Congenital Corneal Acrtic Largenesis Congenital Corneal

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 198 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | f preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | I I |

Rare events

Congenital cystic lung
Congenital Cytomegalovirus infection
Congenital deformity of clavicle
Congenital dermal sinus
Congenital diaphragmatic anomaly
Congenital diaphragmatic eventration
Congenital diaphragmatic eventration
Congenital disorder of glycosylation
Congenital disorder of glycosylation
Congenital disorder of glycosylation
Congenital dyskeratosis
Congenital dyskeratosis
Congenital ectopic plander
Congenital ectopic plander
Congenital ectopic pancreas
Congenital ectopic pancreas
Congenital ectopic pancreas
Congenital elevation of scapula
Congenital elevation of scapula
Congenital epiblepharon
Congenital epiblepharon
Congenital facial nerve hypoplasia
Congenital facial nerve hypoplasia
Congenital facial nerve hypoplasia
Congenital facial nerve hypoplasia
Congenital facial nerve hypoplasic
Congenital facial nerve hypoplasic
Congenital facial nerve hypoplasic
Congenital facial nerve hypoplasic
Congenital gastrointectinal vessel anomaly
Congenital gastrointectinal disorder
Congenital genital malformation female
Congenital genital malformation male
Congenital genital malformation formental genital malformation male
Congenital genital malformation formental genital heart vessel anomaly
Congenital genital halformation
Congenital heart valve disorder
Congenital heart valve disorder
Congenital heart valve incompetence

| NN9535 | Clinical Trial Report | Date: 0 | 4 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 199 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |
| | | | | | | ı |

Rare events

Pre-defined MedDRA search

Congenital hepatici fibrosis
Congenital hepatitis B infection
Congenital hepatobiliary anomaly
Congenital hepatobiliary anomaly
Congenital hepatobiliary anomaly
Congenital hidra herpes simplex infection
Congenital hidra hermals
Congenital hydrocephalus
Congenital hydrocephalus
Congenital hydrocephalus
Congenital hypercoagulation
Congenital hyperextension of knee
Congenital hyperextension of spine
Congenital hyperextension of spine
Congenital hyperextension of spine
Congenital hyperextension of spine
Congenital hyperextension of spine
Congenital hyperthyroidism
Congenital hypotranadlobulinaemia
Congenital hypoparathyroidism
Congenital hypoparathyroidism
Congenital infection and formation
Congenital infection and formation
Congenital infectional malformation
Congenital intestinal malformation
Congenital intestinal malformation
Congenital intestinal obstruction
Congenital intestinal dostruction
Congenital intestinal dostruction
Congenital intestinal dostruction
Congenital here deformity
Congenital large intestinal atresia
Congenital lippishula
Congenital lippishula
Congenital lippishula
Congenital lippishula

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 200 of 229 | |
| Pre-defined MedDRA search - list of preferred | E preferred terms | | | | | |

Rare events

Pre-defined MedDRA search

Congenital mitochondrial cytopathy
Congenital mitral valve incompetence
Congenital mitral valve stenosis
Congenital multiplex arthrogryposis
Congenital muscle absence
Congenital muscle absence
Congenital mysthenic syndrome
Congenital mysthenic syndrome
Congenital myopathy
Congenital myopia
Congenital myopia
Congenital mitocher
Congenital mitocher
Congenital nasal septum deviation
Congenital nasal septum deviation
Congenital neshrogenic diabetes insipidus nephrotic syndrome neurological degeneration neurological disorder 1. pancreatic anomaly laterated nasal septum pharyngeal anomaly lipidentation disorder lipeumonia lipoikiloderma I nipple anomaly
I nipple inversion
I nose malformation
I nystagmus
Coulomotor apraxia
Cosophageal anomaly
Cosophageal stenosis
Cosophageal web Congenital optic nerve anomaly Congenital oral malformation Congenital osteodystrophy Congenital methaemoglobinaemia neuropathy night blindness Congenital ovarian anomaly midline defect malaria megacolon megaureter Congenital melanosis Congenital oxalosis Congenital n Congenital n Congenital n Congenital n Congenital n Congenital n Congenital p Congenital p Congenital p Congenital p Congenital p Congenital r Congenital r Congenital r Congenital o Congenital Congenital Congenital Congenital

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final Novo A | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 201 of 229 | |
| Pre-defined MedDRA search - list of preferred | preferred terms | | | | | |

Rare events

Pre-defined MedDRA search

Congenital pseudarthrosis
Congenital pulmonary artery anomaly
Congenital pulmonary valve atresia
Congenital pulmonary valve atresia
Congenital pulmonary valve atresia
Congenital rubella disorder
Congenital rubella syndrome
Congenital scleral disorder
Congenital scleral disorder
Congenital scleral hypertrophy
Congenital skin dimples
Congenital skin dimples
Congenital skin dimples
Congenital skin dimples
Congenital skin dimples
Congenital skin dimples
Congenital spinal fusion
Congenital spinal fusion
Congenital spinal stenosis
Congenital spondylolysis
Congenital spondylolysis
Congenital syphilitic encephalitis
Congenital syphilitic encephalitis
Congenital syphilitic osteochondritis
Congenital syphilitic osteochondritis
Congenital thrombocytopenia
Congenital thrombocytopenia
Congenital thrombocytopenia
Congenital tricuspid disorder
Congenital tricuspid valve atresia
Congenital tricuspid valve incompetence
Congenital tricuspid valve incompetence
Congenital uricuspid valve incompetence
Congenital uricuspid valve stenosis
Congenital ureteric anomaly
Congenital ureteric anomaly
Congenital ureterovesical junction anomaly

Preferred term Pre-defined MedDRA search - list of preferred terms Pre-defined MedDRA search

Rare events

Cutaneovisceral angiomatosis with thrombocytopenia Connective tissue dysplasia
Conradi-Huenermann syndrome
Constricted ear deformity
Cor biloculare
Cor triatriatum
Corneal dystrophy
Corneal opacity congenital
Cornelia de Lange syndrome
Corrected transposition of great vessels
Cortical dysplasia
Costello syndrome Cýclopia Cystathionine beta-synthase deficiency Cystic fibrosis Cystic fibrosis carrier Cystic fibrosis gastrointestinal disease Congenital urethral anomaly
Congenital uterine anomaly
Congenital uterine anomaly
Congenital varicella infection
Congenital varicocale
Congenital vas deferens absence
Congenital visual acuity reduced
Congenital visual acuity reduced
Congenital visual acuity reduced
Congenital white blood cell disorder Cryopyrin associated periodic syndrome Cryptophthalmos Conjunctivitis gonococcal neonatal Creatine deficiency syndrome Cri du Chat syndrome Crigler-Najjar syndrome Craniofacial deformity Craniofacial dysostosis Craniolacunia Craniorachischisis Craniosynostosis Cryptorchism Currarino syndrome Cyclic neutropenia Conjoined twins Craniotabes

| NN9535 | Clinical Trial Report | Date: 04 | December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| N9535-4506 | | Version: | 1.0 | Page: | 203 of 229 | |
| Pre-defined MedDRA search - list of prefe | preferred terms | | | | | |

Pre-defined MedDRA search

Rare events

Preferred term

Cystic fibrosis hepatic disease Cystic fibrosis lung Cystic fibrosis pancreatic Cystic fibrosis related diabetes

Cystinosis

Cystinuria

Cytogenetic abnormality Cytomegalovirus nephritis Cytopenia DNA mismatch repair protein gene mutation

Dacryocystocoele DOOR syndrome

Dacryostenosis congenital Dandy-Walker syndrome De Barsy syndrome Deaf mutism

Deafness congenital Deficiency of the interleukin-1 receptor antagonist

Deficiency of the interleukin-36 receptor antagonist
Delayed foetal renal development
Delta-beta thalassaemia
Demyelinating polyneuropathy

Dentatorubral-pallidoluysian atrophy Dentofacial anomaly Dermatofibrosis lenticularis disseminata Dent's disease

Developmental glaucoma Developmental hip dysplasia Desmin myopathy

Dermatoglyphic anomaly

Dextrocardia

Digeorge's syndrome Diabetic foetopathy Diaphragmatic aplasia

Diastrophic dysplasia
Diencephalic syndrome of infancy
Diethylstilboestrol syndrome
Differential white blood cell count abnormal
Diffuse alveolar damage
Dihydropyrimidine dehydrogenase deficiency

| NN9535 | Clinical Trial Report | Date: 04 De | 04 December 2020 Status: | | Final |
|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 204 of 229 |
| Pre-defined MedDBA search - list of prefe | f preferred terms | | | | |

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Pre-defined MedDRA search

Rare events

Dilatation intrahepatic duct congenital
Dissorder of sex development
Disseminated neonatal herpes simplex
Distichiasis
Districulitis Meckel's
Diverticulitis Meckel's
Diverticulum of pharynx, congenital
Dolichocolon
Donbue syndrome
Double heterozygous sickling disorders
Double heterozygous sickling disorders
Double outlet left ventricle
Double outlet left ventricle
Double outlet right ventricle
Double outlet right ventricle
Double outlet right ventricle
Double outlet fifty ventricle
Double outlet right ventricle
Double useter
Double useter
Double syndrome
Dubin-Johnson syndrome
Dubowitz syndrome
Dubowitz syndrome
Dubowitz syndrome
Dubowitz syndrome
Dubowitz syndrome
Dubowitz syndrome
Dubowitz syndrome
Dubonen muscular dystrophy
Duchone muscular dystrophy
Duchone muscular dystrophy
Duchone muscular dystrophy
Duchone muscular syndrome
Duboken algebedis
Ductus venosus agenesis
Ductus venosus agenesis
Duplication of inferior vena cava
Dyschondrosteosis
Dysgnathia
Dysmorphism
Dysmo

| NN9535 | Clinical Trial Report | Date: 04 Dece | 04 December 2020 Status: | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | 1.0 Page: | 205 of 229 |
| The state of the s | 4 | | | | |

Preferred term Pre-defined MedDRA search - list of preferred terms Pre-defined MedDRA search

Rare events

Encephalocele Encephalocutaneous angiomatosis Endothelial protein C receptor polymorphism Enteric duplication Ecsinophil count abnormal
Ecsinophil count decreased
Ecsinophil percentage decreased
Ecsinophilia myalgia syndrome
Ecsinophilic pneumonia acute
Ecsinophilic pneumonia acute
Ecsinophilic pneumonia chronic
Epidermal naevus
Epilepsy congenital
Epilepsy with myoclonic-atonic seizures
Epilepsy with myoclonic-atonic seizures
Erythroblastosis foetalis
Erythrokeratodermia variabilis
Essential fructosuria Eye anterior condenital anomaly Eyelid ptosis congenital Fabry's disease Faciodigitogenital dysplasia Facioscapulohumeral muscular dystrophy Factor I deficiency Ectopic kidney
Ectopic ovary
Ectopic ovsterior pituitary gland
Ectopic thyroid
Ectopic ureter Emanuel syndrome Emery-Dreifuss muscular dystrophy Exophthalmos congenital
External auditory canal atresia
Extrarenal pelvis Elbow synostosis Elliptocytosis hereditary Ellis-van Creveld syndrome Ectrodactyly
Ehlers-Danlos syndrome Entropion congenital Eosinopenia Exomphalos

Novo Nordisk

| Date: 04 December 2020 Status: Final Novo Nordisk Version: 1.0 Page: 206 of 229 | | + | _ | _ | _ | _ | _ | _ | _ | _ |
|---|---|---|---|---|---|---|---|---|---|---|
| N9535<br>N9535-4506 - Clinical Trial I | 20220+027 +0 +0 - 1 202000 VIII VON 7021+071 | ADDITION OF STREET | -defined Meduka search - list of breferred | -defined MedDKA search - list of preferred | -deiined MedDKA search - list of preferred | -deiined MedUKA search - list of preferred | -defined MedDKA search - list of preferred | -defined MedUKA search - list of preferred | -defined MedDKA search - list of preferred | -defined MedDKA search - list of preferred |

Rare events

Factor V Leiden mutation
Factor V Leiden mutation
Factor V Leiden mutation
Factor VII deficiency
Factor VIII deficiency
Factor XIII deficiency
Familial amyologosis
Familial amyologosis
Familial hypocalciuric hypercalcaemia
Familial hypocalciuric hypercalcaemia
Familial infantile bilateral striatal necrosis
Familial poriodic paralysis
Familial poriodic paralysis
Familial cond glycosuria
Familial renal glycosuria
Familial trenal glycosuria
Familial trenal glycosuria
Familial trenal
Familial trenal Femoral retroversion
Femoral retroversion
Femuratibula-ulna complex
Fibrillary glomerulonephritis
Fibrodysplasia ossificans progressiva
Fibrous dysplasia of bone Fatal familial insomnia
Fatty acid oxidation disorder
Febrile bone marrow aplasia
Febrile neutropenia Femoral anteversion Femoral facial syndrome Factor II mutation Factor III deficiency Factor IX deficiency Fanconi syndrome

Pre-defined MedDRA search

| NN9535 | Clinical Trial Report | Date: 04 D | December 2020 Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 Page: | 207 of 229 | |

Pre-defined MedDRA search - list of preferred terms

Preferred term

Rare events

Pre-defined MedDRA search

Gatad2b associated neurodevelopmental disorder Gaucher's disease Gaucher's disease type I Gaucher's disease type II Galactosaemia
Galactosialidosis
Gallbladder agenesis
Gallbladder anomaly congenital
Gap junction protein beta 2 gene mutation
Gastroenteritis clostridial
Gastrointestinal arteriovenous malformation
Gastrointestinal malformation Fraser syndrome Freeman-Sheldon syndrome Freenulum breve Friedreich's ataxia Fructose-1,6-bisphosphatase deficiency Floating-Harbor syndrome
Floating-Harbor syndrome
Foctal alcohol syndrome
Foctal anticonvulsant syndrome
Foctal chromosome abnormality
Foctal malformation
Foctal megacystis Fibrous dysplasia of jaw Fibula agenesis Filippi syndrome Fissure of tongue, congenital Foetal methotrexate syndrome Foetal retinoid syndrome Foetal warfarin syndrome Foramen magnum stenosis Fountain syndrome Fryns syndrome
Full blood count abnormal
Full blood count decreased
GMZ gangliosidosis
GNE myopathy
GRACILE syndrome Fragile X carrier Fragile X syndrome Gastroschisis

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 208 of 229 | |
| Pre-defined MedDRA search - list of preferred | f preferred terms | | | | | |

Rare events

Pre-defined MedDRA search

Gaucher's disease type III

Gelatinous transformation of the bone marrow
Gene mutations transformation of the bone marrow
Gene mutations transformation of the bone marrow
Genetic polymorphism
Genetic polymorphism
Gilbert's syndrome
Gilbert's syndrome
Gilbert's syndrome
Glomerulonephritis acute
Glomerulonephritis membranous
Glomerulonephritis membranous
Glomerulonephritis membranous
Glomerulonephritis minimal lesion
Glomerulonephritis minimal lesion
Glomerulonephritis rapidly progressive
Glomerulonephritis rapidly progressive
Glomerulonephritis rapidly progressive
Glowces transporter type I deficiency
Glucose transporter type I deficiency
Glucose fransporter type III
Glycogen storage disease type III
Glycogen storage disease type IV
Glycogen storage disease type VI
Glycogen storage disease type VI
Glycogen storage disease type VI
Glycogen storage disease type VII
Glycogen storage disease type VIII
Glycogen storage disease type VII
Glycogen storage disease type VII
Glycogen storage disease type VII
Glycogen storage disease type VII
Glycogen storage disease type VIII
Glycog

| NN9535 | Clinical Trial Report | Date: 0 | 04 December 2020 Status: | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: 209 | 209 of 229 |
| Pre-defined MedDRA search - list of prefe | : preferred terms | | | | |

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Rare events

H-ras gene mutation
HERZ gene amplification
HERZ gene amplification
HERZ gene mutation
HERG gene mutation
HIV associated nephropathy
Haematotoxicity
Haemochtomatosis trait
Haemoglobin C disease
Haemoglobin D disease
Haemoglobin E trait
Haemoglobin E trait
Haemoglobin E-thalassaemia disease
Haemoglobin E-thalassaemia disease
Haemoglobin E-thalassaemia disease
Haemoglobin E-thalassaemia disease
Haemoglobin E-thalassaemia disease
Haemopliia A without inhibitors
Haemophilia A without inhibitors
Haemophilia A without inhibitors
Haemophilia E-trait
Haemophilia A without inhibitors
Haemophilia Carrier
Haemophilia B with anti factor IX
Haemophilia Carrier
Haemophilia Carrier
Haemophilia Carrier
Haemophilia Carrier
Haemophilia Carrier
Haemophilia Savito
Hand-foot-genital syndrome
Hartup disease
Hartup disease
Herx disease congenital
Herx disease congenital
Herx disease congenital
Herx to virus-associated nephropathy
Hepatic arteriovenous malformation
Hepatici arteriovenous malformation
Hepatici arteriovenous malformation
Hepatici arteriovenous malformation
Hercditary ataxia
Hercditary ataxia
Hercditary disorder
Hercditary disorder
Hercditary disorder
Hercditary haemochromatosis
Hercditary haemochromatosis
Hercditary haemochromatosis
Hercditary haemochromatosis

Rare events

Pre-defined MedDRA search

Hereditary hypophosphataemic rickets
Hereditary motor and sensory neuropathy
Hereditary motor end sensory neuropathy
Hereditary metor between edisease
Hereditary neuropathic amyloidosis
Hereditary neuropathy with liability to pressure
palsies
Hereditary optic atrophy
Hereditary palmoplantar keratoderma
Hereditary reinal dystrophy
Hereditary sideroblastic anaemia
Hereditary sideroblastic anaemia
Hereditary sideroblastic anaemia
Hereditary stomatocytosis
Hollow visceral myopathy
Hollow visceral myopathy
Hollow visceral myopathy
Hollow visceral myopathy
Hollow visceral myopathy
Holt-oram syndrome
Homocystinnemia
Hodromephrosis
Hydronephrosis
Hydronephrosis
Hydronephrosis
Hydronephrosis
Hyper IgB syndrome
Hyper IgB syndrome
Hyper IgB syndrome
Hyper IgE syndrome
Hypermethioninaemia
Hypermethioninaemia
Hypermethioninaemia
Hypermethioninaemia
Hypermethioninaemia
Hypermethioninaemia
Hypermethioninaemia
Hypermethioninaemia

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final Novo A | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 211 of 229 | |
| Pre-defined MedDRA search - list of preferred | E preferred terms | | | | | |

Rare events

Pre-defined MedDRA search

Hyperpipecolic acidaemia Hyperpipecolic acidaemia Hyperpolinaemia Hypersplanism ongenital Hypersplanism or oxpit Hyperthermia malignant Hyperthermia malignant Hyperthermia malignant Hyperthermia malignant Hyperthermia malignant Hyperpolaxia malignant Hypodontia Hypoplastic left heart syndrome Hypoplastic right heart syndrome Hypoplastic right heart syndrome Hypoplastic right heart syndrome Hypoplastic right heart syndrome Hypoplastic right heart syndrome Hypotonia-cystinuria syndrome Hypotonia-cystinuria syndrome Hypotonia-cystinuria syndrome Idiopathic interstitial pneumonia Idiopathic pneumonia syndrome Infantate hymen Imporn error of amino acid metabolism Inborn error of bilirubin metabolism Inborn error of metabolism Inborn error of metabolism Infantile genetic agranulocytosis

| NN9535 | Clinical Trial Report | Date: 04 | December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 212 of 229 | |
| Pre-defined MedDRA search - list of preferre | f preferred terms | | | | | |

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Pre-defined MedDRA search

Rare events

Intercephaly
Interferon gamma receptor deficiency
Interferon gamma receptor deficiency
Interruption of aortic arch
Interruption of aortic arch
Interstinal lauresia
Intestinal malrotation
Intestinal malrotation
Intestinal malrotation
Intestinal malrotation
Intestinal malrotation
Intracranial arterial fenestration
Intracranial lipoma
Iris coloboma
Iris coloboma
Isovaleric acidaemia
Johanson-Blizzard syndrome
Johanson-Blizzard syndrome
Johanson-Blizzard syndrome
Johanson-Blizzard syndrome
Wearns-Sayre syndrome
Kaufman-McKusick syndrome
Kaufman-McKusick syndrome
Kearns-Sayre syndrome
Kearns-Sayre syndrome
Keartitis-ichthyosis-deafness syndrome
Keartitis-ichthyosis-deafness syndrome
Keartitis-ichthyosis-deafness syndrome
Keratolysis exfoliativa congenital
Kidney malformation
Kidney malformation
Kidney malformation
Kidney malformation
Kidney malformation
Kineflete's syndrome
Klippel-Feil syndrome
Klibpel-Feil syndrome
Libband syndrome
Libband syndrome
Libband syndrome

| Novo Nordisk | |
|-----------------------|-------------|
| Final N | 213 of 229 |
| Status: | Page: |
| 04 December 2020 | 1.0 |
| Clinical Trial Report | <u>.</u> |
| NN9535 | NN9535-4506 |

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Rare events

Lacrimal punctum agenesis
Laevocardia
Laevocardia
Laerora 'S mycolonic epilepsy
Lamin A'C gene mutation
Lampar-Giedion syndrome
Laryngeal web
Laryngeal cleft
Laryngocale
Laryngocale
Laryngocole
Lecithin-cholesterol acyltransferase deficiency
Left ventricular false tendon
Left ventricular false tendon
Left ventricular false tendon
Left ventricular syndrome
Limb hypoplasia congenital
Lipid proteinosis
Lipid proteinosis
Lipid proteinosis
Lipid proteinosis
Lipid syndrome
Lipid syndrome
Lipid syndrome
Long-chain acyl-coenzyme A dehydrogenase
Geficiency
Lowy-wood syndrome
Lumparisation
Lumpus nephritis
Lymphangiectasia intestinal congenital

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: 2 | 214 of 229 |
| Pre-defined MedDRA search - list of prefe | preferred terms | | | | |

Novo Nordisk

Rare events

Pre-defined MedDRA search

Lymphocyte count abnormal
Lymphocyte count decreased
Lymphocyte percentage abnormal
Lymphocyte percentage abnormal
Lymphocyte percentage abnormal
Lymphocyte percentage decreased
Lymphocytopenia neonatal
Lymphocytopenia neonatal
Lymphocytopenia
Lymphocytopenia
Lymphocytopenia
Macka syndrome
MTASA syndrome
MTASA syndrome
MTASA syndrome
MTASA syndrome
MTASA syndrome
MTASA syndrome
Macrocophaly
Macrocophaly
Macrocophaly
Macrocophaly
Macrocophaly
Macrocophaly
Macrocophaly
Macrocophaly
Macrocophaly
Macrocophal

Final Novo Nordisk 215 of 229 04 December 2020 Status: 1.0 Page: Version: Date: | Clinical Trial Report NN9535-4506 NN9535

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term

Rare events

Mesangioproliferative glomerulonephritis
Metabolic myopathy
Metabolic myopathy
Metachromatic leukodystrophy
Metarpulocyte count decreased
Metaphyseal dysplasia
Metatarsus primus varus
Metatrasus primus varus
Metatropic dysplasia
Methylenetetrahydrofolate reductase gene mutation
Methylenetetrahydrofolate reductase gene mutation
Methylenetetrahydrofolate reductase polymorphism
Methylenetetrahydrofolate reductase polymorphism
Methylenetetrahydrofolate reductase gene mutation
Methylenetetrahydrofolate reductase polymorphism
Methylenetetrahydrofolate
Methylenetetrahydrofolate
Microcophaly
Microcophaly
Microconea
Microconea
Microgonia
Microphthalmos
Microphthalmos
Microphthalmos
Microphthalmos
Microphthalmos
Microphthalmos
Microphthalmos
Microcophial
Microcophial
Microcondrial
Microcondrial
Microcondrial
Microcondrial
Microcondrial
Microcondrial myopathy
Mitchondrial hepatopathy
Mitchondrial myopathy
Mitchondrial
Mitc

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Final | Final Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 216 of 229 | |
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | | |

Rare events

Pre-defined MedDRA search

Monoblast count decreased
Monocyte count decreased
Monocyte count decreased
Monocyte count decreased
Monocytopenia
Monolid eyes
Monolid eyes
Monopodia
Moragani-Stewart-Morel syndrome
Moraning glory syndrome
Moraning glory syndrome
Moralipidosis type II
Mucolipidosis type II
Mucolipidosis type II
Mucolipidosis type II
Mucolipidosis type III
Mucolipidosis type III
Mucolipidosis type III
Mucopolysaccharidosis II
Mucopolysaccharidosis III
Mucopolysaccharidosis III
Mucopolysaccharidosis III
Mucopolysaccharidosis III
Mucopolysaccharidosis III
Mucopolysaccharidosis VI
Mucopolysaccharidosis VI
Mucopolysaccharidosis VI
Multiple cardiac defects
Multiple cardiac defects
Multiple gastrointestinal atresias
Multiple gastrointestinal atresias
Multiple gastrointestinal atresias
Multiple gastrointestinal atresias
Multiple gastrointestinal atresias
Multiple lentigines syndrome
Muscolar dystrophy
Mutagenic effect
Myelocyte count decreased
Myelocyte count decreased
Myelocyte count decreased
Myelocyte percentage decreased
Myelocyte percentage decreased
Myelocyte percentage decreased
Myelocyte percentage decreased
Myelocyte count decreased
Myelocyte percentage decreased
Myelocyte percentage decreased
Myelocyte percentage decreased
Myelocyte count decreased
Myelocyte count decreased
Myelocyte count decreased
Myelocyte gencentage decreased
Myelocyte percentage deficiency
Myelocyte gencentage decreased
Myelocyte gencentage decreased
Myelocyte gencentage decreased
Myelocyte gencentage decreased
Myelocyte gencentage decreased
Myelocyte gencentage decreased

| NN9535 | Clinical Trial Report | Date: 04 Decem | December 2020 | Status: | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: 2 | 17 of 229 |
| Pre-defined MedDRA search - list of prefe | f preferred terms | | | | |

Novo Nordisk

Rare events

Pre-defined MedDRA search

Myoclonic epilepsy and ragged-red fibres
Myotonia congenita
Myotonia congenita
Myotonia congenita
Narotolia dystrophy
N-acstylglutamate synthase deficiency
N-ras gene mutation
NATI polymorphism
NATI polymorphism
NATY polymorphism
NATY polymorphism
NATY polymorphism
NATY polymorphism
NATY polymorphism
NATY polymorphism
NATY polymorphism
NATY polymorphism
NATY polymorphism
Naturation
Naturation
Nail aplasia
Nacious pider congenital
Nail aplasia
Nail-patella syndrome
Nasopharyngeal atreals
Nacortising bronchiclitis
Neonatal lupus erythematosus
Nephritis
Neonatal lupus erythematosus
Nephritis radiation
Neurodegeneration with brain iron accumulation
disorder
Neurodegeneration with brain iron disorder
Neurodegeneration disorder
Neuropenia neonatal
Neuropenia neonatal
Neuropenia neonatal
Neuropenia neonatal
Neuropenia cont decreased
Neurophil count decreased
Neurophil count decreased
Newborn persistent pulmonary hypertension
Niemann-Pick disease

| NN9535 | Clinical Trial Report | Date: 0 | 4 December 2020 | Status: | Final / | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 218 of 229 | |
| Pre-defined MedDRA search - list of pref | f preferred terms | | | | | |

Rare events

Pre-defined MedDRA search

Nievergelt-Pearlman syndrome
Nijmegen breakage syndrome
Non-compaction cardiomyopathy
Non-compaction cardiomyopathy
Non-compaction cardiomyopathy
Non-compaction cardiomyopathy
Non-compaction syndrome
Obliterative bronchiolitis
Ocular albinism
Oculocarborrenal syndrome
Oculocarborrenal syndrome
Oculocarborrenal syndrome
Oculocarborrenal syndrome
Oculocarborrenal syndrome
Oculocarborrenal syndrome
Oculocarborrenal syndrome
Offactory nerve agenesis
Olfactory nerve agenesis
Olfactory nerve agenesis
Olfactory nerve agenesis
Olfactory nerve hypoplasia
Optic claial-digital syndrome
Optic also pit
Optic disc pit
Optic disc pit
Oral-facial-digital syndrome
Optic disc pit
Oral-facial-digital syndrome
Optic disc pit
Oral-facial-digital syndrome
Optic disc pit
Oral-facial-digital syndrome
Optic disc pit
Oral-facial-digital syndrome
Optic computation
Osteogenesis imperfecta
Osteogenesis imperfecta
Osteogenesis
Osteogenesis
Osteogenesis
Ovarian hypoplasia

| Novo Nordisk | | ı |
|---|---|---|
| Final | 219 of 229 | |
| Status: | Page: | |
| 04 December 2020 | 1.0 | |
| Clinical Trial Report | 1 | f preferred terms |
| NN9535 | NN9535-4506 | Pre-defined MedDRA search - list of preferred |

Rare events

Pre-defined MedDRA search

Pachyonychia congenita
Pallister-Killian syndrome
Panlister-Killian syndrome
Pancreas divisum
Pancreas divisum
Pancreas divisum
Pancreas divisum
Pancreas divisum
Parachute mitral valve
Paranasal sinus aplasia
Paranasal sinus hypoplasia
Paranasal sinus hypoplasia
Paranasal sinus hypoplasia
Paranasal sinus hypoplasia
Paranasal sinus syndrome
Paroxyamal extreme pain disorder
Pareson's syndrome
Pectus excavatum
Pelizaeus-Merzbacher disease
Pelizeus-Merzbacher disease
Pelizeus-Gestruction
Pelizeus-Gestruction
Pelizeus-Merzbacher disease
Pelizeus-Merzbacher disease
Pelizeus-Merzbacher disease
Persion Felizeus
Penic fibrosis
Pelizeus-Merzbacher disease
Persistent fordome
Persistent dusion
Persistent doedal circulation
Persistent left superior vena cava
Persistent urogenital sinus
Persistent urogenital sinus
Pelifer syndrome
Phalangeal agenesis
Phalangeal hypoplasia
Phimosis
Phimosis
Phimosis
Phimosis
Phytosterolaemia
Plionidal cyst congenital

Final Novo Nordisk 220 of 229 04 December 2020 Status: 1.0 Page: Version: Date: | Clinical Trial Report NN9535-4506 NN9535

Pre-defined MedDRA search - list of preferred terms

Preferred term

Rare events

Pre-defined MedDRA search

Plasma cell disorder
Plasma cells absent
Plasmablast count decreased
Plasminogen activator inhibitor polymorphism
Plasminogen activator inhibitor type 1 deficiency Platelet count decreased
Platelet glycoprotein gene mutation
Platelet maturation arrest
Platelet production decreased
Platelet toxicity
Platelet toxicity
Platelet-derived growth factor receptor gene Portal venous system anomaly
Post infection glomerulonephritis
Post streptococcal glomerulonephritis
Postauricular fistula
Posterior segment of eye anomaly congenital Platelet-derived growth factor receptor Potter's syndrome
Prader-Willi syndrome
Preduricular cyst
Preduodenal portal vein
Preternatural anus
Primary cerebellar degeneration
Primary ciliary dyskinesia Porphyria Porphyria acute Porphyria non-acute Porphyrin metabolism disorder Popliteal pterygium syndrome Poland's syndrome Polycystic liver disease Polydactyly Polymicrogyria overexpression Platonychia Platýspondylia Polyorchidism Porokeratosis Porphyrinuria Porencephaly Pneumonitis Platybasia mutation

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 | Status: | Ē |
|---|---|---|---|---|---|
| NN9535-4506 | | Version: | 1.0 | Page: | 221 of: |
| Pre-defined MedDRA search - list of | of preferred terms | | | | |

Rare events

Pre-defined MedDRA search

Progesterone receptor gene overexpression Progressive cerebellar degeneration Progressive external ophthalmoplegia Progressive manilial intrahepatic cholestasis Progressive massive fibrosis Prominent epicanthal folds Prominent epicanthal folds Promes C deficiency Primary coenzyme Q10 deficiency
Primary familial hypomagnesaemia
Primary hypercholesterolaemia
Primary hyperoxaluria
Primary immunodeficiency syndrome
Primary insulin like growth factor-1 deficiency
Pro-opiomelanocortin deficiency Pulmonary aplasia
Pulmonary arteriovenous fistula
Pulmonary artery atresia
Pulmonary artery stenosis congenital
Pulmonary fibrosis
Pulmonary hypoplasia
Pulmonary lymphangiectasia Proximal focal femoral deficiency Pseudocholinesterase deficiency Pseudohermaphroditism Pseudohermaphroditism female Pulmonary necrosis Pulmonary radiation injury Pulmonary renal syndrome Pulmonary sequestration Pulmonary toxicity Pseudohermaphroditism male Pseudohypoparathyroidism Pseudomembranous colitis Pseudotruncus arteriosus Pseudoxanthoma elasticum Pseudohypoaldosteronism Pulmonary malformation Proteus syndrome Protuberant ear Pterygium colli Progeria

Final Novo Nordisk

Final Novo Nordisk 222 of 229 04 December 2020 Status: 1.0 Page: Version: Date: | Clinical Trial Report NN9535-4506 NN9535

Pre-defined MedDRA search - list of preferred terms

Preferred term

Rare events

Pre-defined MedDRA search

Progenic sterile arthritis pyoderma gangrenosum Pyruvate carboxylase deficiency
Pyruvate dehydrogenase complex deficiency
Pyruvate kinase deficiency anaemia
RET gene mutation
RPE65 gene mutation Renal dysplasia
Renal fusion anomaly
Renal hypoplasia
Renal malposition
Renal vessel congenital anomaly
Reproductive tract hypoplasia, male
Respiratory tract malformation Rhesus haemolytic disease of newborn Rib hypoplasia Rib synostosia Riba yanostosia Right aortic arch Right ventricular false tendon Pulmonary valve stenosis congenital Pure white cell aplasia Pycnodysostosis Retinal anomaly congenital
Retinal arteriovenous malformation
Retinal coloboma
Retinitis pigmentosa
Retinopathy congenital
Retinoschisis congenital Rapid-onset dystonia-parkinsonism Rathke's cleft cyst Rectal atresia
Red blood cell enzymes abnormal
Refsum's disease
Renal aplasia
Renal arteriovenous malformation Radiation alveolitis
Radiation fibrosis - lung
Radiation leukopenia
Radiation pneumonitis and acne syndrome Pyloric stenosis Retroperitonitis

04 December 2020 Status: 1.0 Page: Version: Date: Clinical Trial Report NN9535-4506 NN9535

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Rare events

Septo-optic dysplasia
Septo-optic dysplasia
Septum pellucidum agenesis
Serotonin syndrome
Sertoli-cell-only syndrome
Severe myoclonic epilepsy of infancy
deficiency
Sex chromosome abnormality Shone complex Short stature homeobox gene mutation Short-chain acyl-coenzyme A dehydrogenase deficiency Scaphocephaly Schimke immunoosseous dysplasia Schinzel-Giedion syndrome Schizencephaly
Schmid Fraccaro syndrome
Schwartz Jampel syndrome
Scimitar syndrome
Sclerctylosis
Sensory neuropathy hereditary
Septate hymen Shprintzen-Goldberg syndrome Shwachman-Diamond syndrome Sickle cell anaemia Sickle cell disease Sickle cell disease Sickle cell trait Silver-Russell syndrome Single atrium Right-to-left cardiac shunt Riley-Day syndrome Ring chromosome Rippling muscle disease Rotor's syndrome Rubinstein-Taybi syndrome SADDAN syndrome SATB2-associated syndrome Sacral hypoplasia Sacralisation Saposin C deficiency Sarcoglycanopathy Shawl scrotum Sarcosinaemia

Final Novo Nordisk


| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | | Final |
|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: 22 | 24 of 229 |
| Pre-defined MedDRA search - list of prefe | E preferred terms | | | | |

Novo Nordisk

Rare events

Pre-defined MedDRA search

Single umbilical artery

Preferred term

Spondylopphyseal dysplasia Stahl's ear Stanl's ear Standson Stargardt's disease Stickler's syndrome Stickler's syndrome Strabismus congenital Stradding tricuspid valve Sturge-Weber syndrome Subacute inflammatory demyelinating polyneuropathy Sucrase-isomaltase deficiency Supernumerary vertebra siringre unbilited aftery
Sirenomelia
Sjogren-Larsson syndrome
Skeletal dysplasia
Skin hypoplasia
Skin malformation
Skull malformation
Small airways disease
Smith-Lemli-Opitz syndrome
Smith-Magenis syndrome
Special senses congenital anomaly
Spherophabitida
Spina bifida cystica
Spina bifida cystica
Spina bifida coculta
Spina muscular atrophy
Spine malformation
Spine malformation Synostosis Syringomyelia Syringomyelia Systemic right ventricle T-lymphocyte count abnormal T-lymphocyte count decreased TORCH infection TRPV4 gene mutation Talipes Tangier disease Telangiectasia congenital Teratogenicity Syndactyly

| Final <b>Novo Nordisk</b><br>f 229 | |
|---|---|
| Final 225 of 229 | |
| 120 Status:<br>1.0 Page: | |
| 04 December 2020 Status: | |
| Date:<br>Version: | |
| Clinical Trial Report | of preferred terms |
| NN9535<br>NN9535-4506 | Pre-defined MedDRA search - list of preferred |

Rare events

Pre-defined MedDRA search

Testicular dysplasia
Testotoxicosis
Testotoxicosis
Tetrahydrobiopterin deficiency
Thalassaemia alpha
Thalassaemia alpha
Thalassaemia beta
Thalassaemia minor
Thalassaemia minor
Thalassaemia sickle cell
Thalidomide embryopathy
Thanatophoric dwarfism
Thopurine methyltransferase polymorphism
Thrombocytopenia
Thrombocytopenia
Thrombocytopenia
Thrombocytopenia
Thronglossal fistula
Thyroid hemiagenesis
Thyroid hemiagenesis
Thyroid malformation
Tibial agenesis
Tibial dorsion
Tibial torsion
Tibial torsion
Tibial torsion
Tibial sacolouration congenital
Tooth hypoplasia
Tooth malformation hereditary
Tourette's disorder
Tracheal atresia
Tracheal web
Tracheal web
Tracheal web
Tracheal web
Tracheal web
Transcobalamin deficiency
Transgenerational epigenetic inheritance
Transgenerational epigenetic inheritance
Transgenerational vertebrae
Transgenerational vertebrae
Transmembrane receptor tyrosine kinase
overexpression
Transpension of the great vessels
Trinchninophalangeal syndrome
Triple A syndrome
Trisomy 13
Trisomy 13
Trisomy 13

| NN9535 | Clinical Trial Report | Date: 04 | December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 226 of 229 | |
| Pre-defined MedDBA search - list of | - list of preferred terms | | | | | |

Rare events

Pre-defined MedDRA search

Trisomy 15
Trisomy 16
Trisomy 17
Trisomy 17
Trisomy 21
Trisomy 21
Trisomy 21
Trisomy 22
Trisomy 8
Trisomy 8
Trisomy 8
Trisomy 9
Trisomy 10
Trisomy 9
Trisomy 10
Trisomy 1

| NN9535 | Clinical Trial Report | Date: 0 | 4 December 2020 | Status: | Final | Novo Nordisk |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | Page: | 227 of 229 | |
| Pre-defined MedDRA search - list of preferred | f nraferrad terms | | | | | |

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Pre-defined MedDRA search

Rare events

Urinary tract malformation
Urinary tract malformation
Usher's syndrome
Usher's syndrome
Uterine aplasia
Uterine cervix hypoplasia
Uterine cervix hypoplasia
Uterine hypoplasia
Uterine hypoplasia
Uterine hypoplasia
Uterine hypoplasia
VACTERL syndrome
VRORCI gene polymorphism
Vaginal atresia
Vaginal atresia
Vaginal septum
Vascular malformation
Vascular malformation
Vascular malformation
Vascular malformation
Velo-carding-facial syndrome
Ventricular hypoplasia
Vertebral artery hypoplasia
Vertebral artery hypoplasia
Vertebral artery hypoplasia
Vertebral atrestinal duct remnant
Verticular hypoplasia
Vertebral actery disease
Verticular septal defect
Vertebral actery hypoplasia
Verticular septal defect
Vertebral actery hypoplasia
Verticular septal defect
Vertebral actery hypoplasia
V

| NN9535 | Clinical Trial Report | Date: | 04 December 2020 Status: | Status: | Final | Novo |
|---|---|---|---|---|---|---|
| NN9535-4506 | 1 | Version: | 1.0 | 1.0 Page: | 228 of 229 | |
| Pre-defined MedDRA search - list of preferred | of preferred terms | | | | | |
| Pre-defined MedDRA search | Preferred term | | | | | 1 1 |

Wolfram syndrome
Woodhouse-Sakati syndrome
Woodhouse-Sakati syndrome
Wyburn Mason's syndrome
X-linked chromosomal disability, Siderius type
XXX syndrome
XXXY syndrome
XXYY syndrome
XXYY syndrome
XXYY syndrome Young's syndrome
Zhu-Tokita-Takenouchi-Kim syndrome
Zika virus associated Guillain Barre syndrome
Zika virus associated birth defect
Zika virus associated microencephaly
Zika virus associated coular birth defect Y-linked chromosomal disorder Wolf-Hirschhorn syndrome Xeroderma pigmentosum Suspected transmission of an infectious agent Rare events

Infection transmission via personal contact
Infection via vaccine
Infectious disease carrier
Nosocomial infection Faecal-oral transmission of infection Fungal disease carrier HIV carrier HHIV-1 carrier Human immunodeficiency virus transmission Primary transmission SARS-CoV-2 carrier Secondary transmission Sexual transmission of infection Sexually transmitted disease Sexually transmitted disease Air-borne transmission
Arthropod-borne disease
Bacterial disease carrier
Community acquired infection
Diphtheria carrier
Direct infection transmission Indirect infection transmission **latrogenic** infection

| NN9535<br>NN9535-4506 | Clinical Trial Report<br>- | Date:<br>Version: | 04 December 2020 Status:<br>1.0 Page: | Final 229 of 229 | Final <b>Novo Nordisk</b><br>f 229 |
|---|---|---|---|---|---|
| Pre-defined MedDRA search - list of preferred terms | preferred terms | | | | |
| Pre-defined MedDRA search | Preferred term | | | | |
| Suspected transmission of an infectious agent | | Suspected transmission of an infectious agent via product Transmission of an infectious agent via product Transmission of an infectious agent via transplant Vaccine bacteria shedding Vaccine virus shedding Vaccine virus shedding Vector-borne transmission of infection Viral disease carrier Viral hepatitis carrier | us agent via<br>ia product<br>ia transplant<br>n | | |

MeDRA version 23.0

nn9535/nn9535-4506/ctr 20201204 er 04DEC20201214:40:12 - lmeddrapt.sas/lmeddrapt.txt